# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN

for

**DMID Protocol: 17-0078** 

A Phase II Study to Assess the Safety, Reactogenicity and Immunogenicity of Different Prime-Boost Vaccination Schedules of 2013 and 2017 A/H7N9 Inactivated Influenza Vaccines Administered Intramuscularly with or without AS03 Adjuvant in Healthy Adults

19-50 Years of Age

17-0078: NCT03589807

Version 1.0

**DATE: 18 March 2021** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

#### **STUDY TITLE**

| Protocol Number Code: | DMID Protocol: 17-0078 |
|---|---|
| <b>Development Phase:</b> | Phase II |
| Products: | Sanofi 2013 and 2017 A/H7N9 Inactivated Influenza Vaccines<br>GSK AS03 Adjuvant<br>Patheon Manufacturing Services (PBS) diluent |
| Form/Route: | IM |
| Indication Studied: | Influenza A/H7N9 |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | August 21, 2018 |
| Clinical Trial Completion Date: | March 12, 2020 |
| Date of the Analysis Plan: | March 18, 2021 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY ' | TITLE | 2 |
|---|---|---|
| LIST OF | ABBREVIATIONS | 6 |
| 1. | PREFACE | 8 |
| 2. | INTRODUCTION | 9 |
| 2.1. | Purpose of the Analyses. | 9 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 10 |
| 3.1. | Study Objectives | 10 |
| 3.1.1. | Primary | 10 |
| 3.1.2. | Secondary | 10 |
| 3.1.3. | Exploratory | 10 |
| 3.2. | Endpoints | 11 |
| 3.2.1. | Primary | 11 |
| 3.2.2. | Secondary | 11 |
| 3.2.3. | Exploratory | 12 |
| 3.3. | Study Definitions and Derived Variables | 13 |
| 4. | INVESTIGATIONAL PLAN | 14 |
| 4.1. | Overall Study Design and Plan | 14 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 14 |
| 4.3. | Selection of Study Population | 15 |
| 4.4. | Treatments | 15 |
| 4.4.1. | Treatments Administered | 15 |
| 4.4.2. | Identity of Investigational Product(s) | 15 |
| 4.4.3. | Method of Assigning Subjects to Study Groups (Randomization) | 15 |
| 4.4.4. | Selection of Doses in the Study | 15 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 15 |
| 4.4.6. | Blinding | 16 |
| 4.4.7. | Prior and Concomitant Therapy | 16 |
| 4.4.8. | Treatment Compliance | 16 |
| 4.5. | Immunogenicity and Safety Variables | 16 |
| 4.5.1. | Safety Variables | 16 |
| 4.5.2. | Immunogenicity Variables | 17 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 19 |

| Table of Contents (continued) | | |
|---|---|---|
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 20 |
| 6.1. | General Principles | 20 |
| 6.2. | Timing of Analyses. | 20 |
| 6.2.1. | CSR | 20 |
| 6.3. | Analysis Populations | 21 |
| 6.3.1. | Safety Population | 21 |
| 6.3.2. | Modified Intent-to-Treat (mITT) Population | 21 |
| 6.3.3. | Per Protocol Population | 21 |
| 6.4. | Covariates and Subgroups | 23 |
| 6.5. | Missing Data | 23 |
| 6.6. | Interim Analyses and Data Monitoring | 23 |
| 6.6.1. | Interim Safety Review | 23 |
| 6.6.2. | Interim Immunogenicity Review | 24 |
| 6.7. | Multicenter Studies | 24 |
| 6.8. | Multiple Comparisons/Multiplicity | 24 |
| 7. | STUDY SUBJECTS | 25 |
| 7.1. | Disposition of Subjects | 25 |
| 7.2. | Protocol Deviations | 25 |
| 8. | IMMUNOGENICITY EVALUATION | 26 |
| 8.1. | Primary Immunogenicity Analysis | 26 |
| 8.2. | Secondary Immunogenicity Analyses | 26 |
| 8.3. | Exploratory Immunogenicity Analyses | 26 |
| 8.3.1. | HAI and Neut Covariate Analysis | 27 |
| 8.3.2. | HAI and Neut Regression Modeling | 27 |
| 8.3.3. | Antibody Secreting Cells (Plasmablasts) | 28 |
| 8.3.4. | Other Assays | 28 |
| 9. | SAFETY EVALUATION | 29 |
| 9.1. | Demographic and Other Baseline Characteristics | 29 |
| 9.1.1. | Prior and Concurrent Medical Conditions | 29 |
| 9.1.2. | Prior and Concomitant Medications | 29 |
| 9.2. | Measurements of Treatment Compliance | 29 |
| 9.3. | Adverse Events | 30 |

| Table of | Contents (continued) | |
|---|---|---|
| 9.3.1. | Solicited Events and Symptoms | 30 |
| 9.3.2. | Unsolicited Adverse Events | 31 |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 31 |
| 9.5. | Pregnancies | 32 |
| 9.6. | Clinical Laboratory Evaluations | 32 |
| 9.7. | Vital Signs and Physical Evaluations | 32 |
| 9.8. | Concomitant Medications | 33 |
| 10. | REPORTING CONVENTIONS | 34 |
| 11. | TECHNICAL DETAILS | 35 |
| 12. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 36 |
| 13. | REFERENCES | 37 |
| 14. | APPENDICES | 38 |
| APPENI | DIX 1. TABLE MOCK-UPS | 39 |
| APPENI | DIX 2. FIGURE MOCK-UPS | 160 |
| APPENI | DIX 3 LISTINGS MOCK-UPS | 178 |

# LIST OF ABBREVIATIONS

| 2013 A/H7N9 | Influenza A Virus A/Shanghai/2/2013 |
|-------------|--------------------------------------------------|
| 2017 A/H7N9 | Influenza A Virus A/Hong Kong/125/2017 |
| A/H7N9 | Influenza A Virus of the H7N9 Subtype |
| AE | Adverse Event/ Adverse Experience |
| AESIs | Adverse Events of Special Interest |
| ALT | Alanine Aminotransferase |
| ASC | Antibody-Secreting Cells |
| AS03 | Adjuvant System (03) |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| С | Celsius |
| CI | Confidence Interval |
| Cr | Creatinine |
| CRF | Case Report Form |
| °C | Degrees Celsius |
| CSR | Clinical Study Report |
| DC | Dendritic Cells |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-Linked Immunosorbent Assay |
| ELLA | Enzyme-Linked Lectin Assay |
| ESR | Erythrocyte Sedimentation Rate |
| °F | Degrees Fahrenheit |
| FDA | U.S. Food and Drug Administration |
| GMT | Geometric Mean Titer |
| GSK | GlaxoSmithKline Biologicals |
| HAI | Hemagglutination Inhibition Antibody |
| Hgb | Hemoglobin |
| DHHS | Department of Health and Human Services |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IgA | Immunoglobulin A |

# **List of Abbreviations** (continued)

| IgG | Immunoglobulin G |
|---------|-----------------------------------------------|
| IgM | Immunoglobulin M |
| IIV | Inactivated Influenza Vaccine |
| IM | Intramuscularly |
| IRB | Institutional Review Board |
| L | Liter |
| MAAE | Medically Attended Adverse Event |
| mcg | Microgram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mITT | Modified Intent-to-Treat |
| N, n | Number of Subjects |
| NA | Neuraminidase |
| NAI | Neuraminidase Inhibition |
| Neut | Neutralizing Antibody |
| NIH | National Institutes of Health |
| NK | Natural Killer |
| NOCMC | New Onset Chronic Medical Condition |
| PBS | Phosphate Buffered Saline |
| PIMMC | Potentially Immune Mediated Medical Condition |
| PP | Per Protocol |
| PLT | Platelets |
| PT | Preferred Term |
| RCD | Reverse Cumulative Distribution |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| SP | Sanofi Pasteur |
| T. Bili | Total Bilirubin |
| VTEU | Vaccine and Treatment Evaluation Unit |
| WBC | White Blood Cell |
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) DMID Protocol 17-0078, "A Phase II Study to Assess the Safety, Reactogenicity and Immunogenicity of Different Prime-Boost Vaccination Schedules of 2013 and 2017 A/H7N9 Inactivated Influenza Vaccines Administered Intramuscularly with or without AS03 Adjuvant in Healthy Adults 19-50 Years of Age" describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures (TFLs) planned for (1) final analyses included in the topline set, and (2) analyses included in the Clinical Study Report (CSR). Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity and safety outcomes, and (4) a list of proposed TFLs. Following any protocol amendment, this SAP will be reviewed and revised (if needed) to address any changes in the protocol impacting analysis. Any deviation from the final SAP will be described and justified in the CSR. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

Since March of 2013 [1], avian influenza A/H7N9 viruses have continued to circulate in China causing discrete outbreaks (or waves) in humans with high mortality over the past 5 years. By late 2016, a fifth wave of outbreaks was identified in China and as of May 18, 2017, a total of 1,463 laboratory-confirmed human infections with avian influenza A/H7N9 virus have been reported by the World Health Organization [2, 3]. Since the onset of the fifth wave of H7N9 outbreaks in October 2016, more human cases of H7N9 infection have been reported in China than any prior H7N9 epidemic wave [3]. The U.S. Department of Health and Human Services (DHHS) recently assessed H7N9 influenza virus as having a significant potential to cause a pandemic, and the greatest risk of causing severe disease. As a result, DHHS has supported the production of fifth wave A/H7N9 inactivated influenza vaccines (IIVs) for the U.S. stockpile and for an assessment of their safety and immunogenicity in clinical trials.

The goal of this trial is to assess in healthy adults the safety, reactogenicity, and immunogenicity of one or two vaccinations of 2013 and 2017 A/H7N9 (influenza A viruses A/Shanghai/2/2013 and A/Hong Kong/125/2017, respectively) IIVs administered intramuscularly at different dosages (3.75 or 15 mcg of hemagglutinin (HA) per dose), given with or without AS03 adjuvant, using different heterologous and homologous prime-boost vaccination schedules to evaluate the study vaccine dosage, dose-sparing potential of the adjuvant, optimal prime-boost interval for immunogenicity (two doses administered 21 days vs. 4 months apart), and priming effects of different A/H7N9 IIVs. In addition to assessing antigen-sparing strategies, another goal of this study is to assess in at least a subset of samples, if serum immunoglobulin elicited by the 2013 and 2017 A/H7N9 IIVs recognize antigenically drifted variants of influenza A/H7 viruses.

# 2.1. Purpose of the Analyses

These analyses will assess the immunogenicity and safety of two vaccinations of 2013 and 2017 A/H7N9 IIVs administered IM either approximately 21 days or approximately 4 months apart with or without AS03 adjuvant and will be included in the topline set of tables and/or clinical study report.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

#### **3.1.1. Primary**

#### Safety:

• To assess the safety and reactogenicity of 2013 and 2017 A/H7N9 IIVs given with or without AS03 adjuvant following receipt of each study vaccine.

#### Immunogenicity:

• To assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of the second study vaccine.

#### 3.1.2. Secondary

#### Safety:

- To assess unsolicited non-serious adverse events (AEs) following receipt of each study vaccine.
- To assess medically attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs), following receipt of each study vaccine.

#### Immunogenicity:

• To assess the kinetics and durability of serum HAI and Neut antibody responses following receipt of each study vaccine.

# 3.1.3. Exploratory

#### Immunogenicity:

- To assess the effects of age, sex, body mass index (BMI), and prior receipt of seasonal or non-study pandemic influenza vaccine(s) on serum HAI and Neut antibody responses following receipt of the second study vaccine.
- To assess the neuraminidase (NA) content of the 2013 and 2017 A/H7N9 IIVs and determine, in at least a subset of samples, the serum antibody responses to N9 NA.
- To assess, in at least a subset of samples, HA stem-specific antibody responses.
- To assess, in at least a subset of samples, the cross-reactivity of serum HAI and Neut antibody responses to antigenically drifted variants of influenza A/H7 viruses.
- To assess, in at least a subset of samples, the frequency of influenza-specific (A/H7N9 antigens) IgA, IgG and IgM memory B cells (MBCs).
- To assess, in at least a subset of samples, the frequency of influenza-specific (A/H7N9 antigens) IgA, IgG and IgM plasmablasts (antibody-secreting cells [ASCs]).
- To assess, in at least a subset of samples, the multifunctional cytokine/chemokine profile of influenza A/H7N9-specific CD4 and CD8 T cells.

- To assess, in at least a subset of samples, the characterization of circulating T follicular helper (cT<sub>FH</sub>) cells.
- To assess, in at least a subset of samples, the study vaccine-induced changes in populations and/or activation status of innate immune cells (monocytes, dendritic cells [DCs] and natural killer [NK] cells).
- To assess, in at least a subset of samples, the study vaccine-induced activation status of B cells.
- To assess, in at least a subset of samples, the B cell receptor repertoire and degree of somatic hypermutation generated in response to study vaccination.

# 3.2. Endpoints

#### **3.2.1. Primary**

#### Safety:

- Occurrence of all serious adverse events (SAEs) from the time of the first study vaccination through approximately 12 months after the last study vaccination.
- Occurrence of solicited injection site and systemic reactogenicity events from the time of each study vaccination through 7 days after each study vaccination.
- Occurrence of clinical safety laboratory AEs from the time of each study vaccination through approximately 7 days after each study vaccination.

#### Immunogenicity:

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion against the influenza A/H7N9 study vaccine viruses (defined as either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and a minimum four-fold rise in post-vaccination antibody titer) approximately 21 days after the second study vaccination.
- For HAI and Neut antibodies, percentage of subjects achieving titer ≥1:40 against the influenza A/H7N9 study vaccine viruses approximately 21 days after the second study vaccination.
- Geometric mean titers (GMTs) of serum HAI and Neut antibodies against the influenza A/H7N9 study vaccine viruses approximately 21 days after the second study vaccination.

#### 3.2.2. Secondary

#### Safety:

- Occurrence of all unsolicited non-serious AEs from the time of each study vaccination through approximately 21 days after each study vaccination.
- Occurrence of all MAAEs, including NOCMCs and PIMMCs, from the time of the first study vaccination through approximately 12 months after the last study vaccination.

#### <u>Immunogenicity:</u>

• For HAI and Neut antibodies, percentage of subjects achieving seroconversion against the influenza A/H7N9 study vaccine viruses approximately 21 days after the first study vaccination as well as immediately prior to and approximately 180 days after the second study vaccination.

- For HAI and Neut antibodies, percentage of subjects achieving titer ≥1:40 against the influenza A/H7N9 study vaccine viruses immediately prior to each study vaccination, approximately 21 days after the first study vaccination and approximately 180 days after the second study vaccination.
- GMTs of serum HAI and Neut antibodies against the influenza A/H7N9 study vaccine viruses immediately prior to each study vaccination, approximately 21 days after the first study vaccination and approximately 180 days after the second study vaccination.

#### 3.2.3. Exploratory

#### Immunogenicity:

- For HAI and Neut antibodies, GMTs and percentage of subjects achieving seroconversion against the influenza A/H7N9 study vaccine viruses approximately 21 days after the second study vaccination, by age, sex, BMI, and prior receipt of seasonal or non-study pandemic influenza vaccine(s).
- GMTs and percentage of subjects achieving seroconversion (defined as four-fold change from baseline) of serum anti-NA (by enzyme-linked immunosorbent assay [ELISA]) or antineuraminidase inhibition (NAI) (by enzyme-linked lectin assay [ELLA]) antibodies immediately prior to and approximately 21 days after each study vaccination as well as approximately 180 days after the second study vaccination.
- Correlate the HA and/or NA content of 2013 and 2017 A/H7N9 IIVs with the elicited HA or N9
  NA-specific antibody titer approximately 21 days after each study vaccination as well as
  immediately prior to and approximately 180 days after the second study vaccination.
- GMTs of HA stem-specific antibody immediately prior to and approximately 21 days after each study vaccination as well as approximately 180 days after the second study vaccination.
- For HAI and Neut antibodies, GMTs and percentage of subjects achieving seroconversion against antigenically drifted variants of influenza A/H7 viruses approximately 21 days after the second study vaccination.
- Percentage of influenza-specific (A/H7N9 antigens) IgA, IgG and IgM MBCs at baseline and approximately 90 and 180 days after the second study vaccination.
- Frequency of influenza-specific (A/H7N9 antigens) IgA, IgG and IgM plasmablasts (ASCs) present in circulation approximately 7 days after each study vaccination.
- Percentage of influenza A/H7N9-specific CD4 and CD8 T cells producing cytokines/chemokines immediately prior to and approximately 7 days after each study vaccination as well as approximately 90 days after the second study vaccination.
- Percentage of cT<sub>FH</sub> cells producing cytokines/chemokines immediately prior to and approximately 3, 7 and 14 days after each study vaccination.
- Percentage and activation status of innate immune cells (monocytes, DCs and NK cells) immediately prior to and approximately 1, 3, 7 and 14 days after each study vaccination.
- Percentage of activated B cells immediately prior to and approximately 1, 3, 7 and 14 days after each study vaccination.

- Evaluation of B cell receptor repertoire and degree of somatic hypermutation of anti-HA (H7) and anti-NA (N9) antibodies at baseline and approximately 180 days after the second study vaccination.
- Correlation of the above exploratory immunologic parameters with HAI and Neut antibodies.

# 3.3. Study Definitions and Derived Variables

For individual subjects, fold rise will be calculated as the ratio of:  $\frac{post-vaccination\ titer}{pre-vaccination\ titer}$ , where pre-vaccination value is always the result obtained at Day 1, prior to the priming vaccination.

HAI Seroconversion is defined as either a pre-vaccination HAI titer <10 and a post-vaccination HAI titer  $\ge40$  or a pre-vaccination HAI titer  $\ge10$  and a minimum four-fold rise in post-vaccination HAI titer [5].

Neut Seroconversion is defined as either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer  $\ge 1:40$  or a pre-vaccination Neut titer  $\ge 1:10$  and a minimum four-fold rise in post-vaccination Neut antibody titer.

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

DMID Protocol 17-0078 follows a Phase II randomized, partially-blinded study design enrolling males and non-pregnant females aged 19 to 50 years of age, inclusive, who are in good health as determined by medical history and physical examination, and meet all eligibility criteria, including erythrocyte sedimentation rate (ESR), hematology, and biochemistry parameter within acceptable range, and negative urine or serum pregnancy test (for females). This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of one or two vaccinations of monovalent inactivated split influenza 2013 and 2017 A/H7N9 virus vaccines (2013 and 2017 A/H7N9 IIVs) manufactured by Sanofi Pasteur (SP), administered intramuscularly at different dosages (3.75 or 15 mcg of HA per dose), given with or without AS03 adjuvant manufactured by GlaxoSmithKline Biologicals (GSK), using different heterologous and homologous prime-boost vaccination schedules.

Subjects will be randomly assigned to 1 of 6 study groups with equal allocation 1:1:1:1:1:1 (see Table 1). Subjects assigned to Groups 1, 2, and 3 will receive an adjuvanted 2013 A/H7N9 IIV on Day 1 while those in Groups 4, 5, and 6 receive an adjuvanted 2017 A/H7N9 IIV on Day 1. Subjects assigned to Groups 1 and 4 will return approximately 21 days after their first vaccination to receive an adjuvanted 2017 A/H7N9 IIV. Subjects assigned to Groups 2,3,5, and 6 will return approximately after 120 days to receive their second vaccination of 2017 A/H7N9 IIV with or without AS03.

Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions from the time of each study vaccination through 7 days after each study vaccination. Unsolicited non-serious AEs will be collected from the time of each study vaccination through approximately 21 days after each study vaccination. SAEs and MAAEs, including NOCMCs and PIMMCs, will be collected from the time of the first study vaccination through approximately 12 months after the last study vaccination. Clinical laboratory evaluations for safety will be performed on venous blood collected prior to each study vaccination and approximately 7 days after each study vaccination.

Immunogenicity testing will include performing HAI and Neut antibody assays against the influenza A/H7N9 study vaccine viruses on serum samples collected immediately on Day 1, Day 22 post vaccination 1, Day 121 post vaccination 1 for study groups 2,3,5,6, and on approximately Day 181 post vaccination 2.

Novel methods for identifying and assessing alternative correlates of protection against influenza infection are needed. To assess the NA specific antibody response to vaccination, it is first necessary to determine the NA content of inactivated influenza vaccine; this assay is under development. If successful, the NA content in a dosage specific manner can be correlated to the N9 NA-specific antibody responses elicited by the 2013 and 2017 H7N9 IIVs. The analyses for this exploratory endpoint will be described in an addendum to this SAP, if the assay becomes available.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

This study uses a dose comparison concurrent control design. Study subjects received either 2013 A/H7N9 IIV or 2017 A/H7N9 IIV with differing dosages with or without adjuvants and on differing administration schedules.

# 4.3. Selection of Study Population

The study population for this clinical trial is 180 males and non-pregnant females, 19 to 50 years of age, inclusive, who are in good health and meet all eligibility criteria. The subjects will be recruited from the general population at the participating Vaccine Trial and Evaluation Unit (VTEU) sites that have substantial experience conducting large influenza vaccine studies.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

2013 and 2017 A/H7N9 Inactivated Influenza Vaccines and AS03 Adjuvant will be administered.

## 4.4.2. Identity of Investigational Product(s)

See the study protocol for details of study product formulation.

#### 4.4.3. Method of Assigning Subjects to Study Groups (Randomization)

Enrollment/randomization will be performed through the enrollment module in the electronic data capture system, maintained by the SDCC.

Eligible subjects will be stratified by clinical site and prior receipt of seasonal influenza vaccine and randomly assigned with equal allocation (1:1:1:1:1) to 1 of 6 study groups indicated in Table 1. The treatment sequence was generated using permuted block randomization to provide an approximately balanced allocation to the study groups during the study.

#### 4.4.4. Selection of Doses in the Study

Subjects in Groups 1, 2, and 3 are to receive a first vaccination of AS03 adjuvanted 2013 A/H7N9 IIV at HA dose of 3.75mcg, and a second vaccination of either AS03 adjuvanted 2017 A/H7N9 IIV at HA dose of 3.75mcg (Groups 1 and 2) or unadjuvanted 2017 A/H7N9 IIV at HA dose of 15mcg (Group 3). Subjects in Groups 4, 5 are to receive two AS03 adjuvanted 2017 A/H7N9 vaccinations at HA dose of 3.75. Subjects in Group 6 are to receive a first vaccination of AS03 adjuvanted 2017 A/H7N9 IIV at HA dose of 3.75mcg, and a second vaccination of unadjuvanted 2017 A/H7N9 IIV at HA dose of 15mcg.

The 3.75 mcg with AS03 dose was selected to evaluate safety and immunogenicity of antigen sparing dose strategies compared to that of using a higher dose of 15 mcg without adjuvant. Using the 2013 and 2017 A/H7N9 IIVs allows the evaluation of priming effects of different A/H7N9 IIVs.

#### 4.4.5. Selection and Timing of Dose for Each Subject

Each subject is to be randomly assigned to a study group which will define the number and timing of 2013 and/or 2017 A/H7N9 vaccinations. The first vaccination for all subjects takes place on the day of randomization and will include vaccination with AS03 adjuvanted 2013 A/H7N9 IIV (Groups 1,2,3) or AS03 adjuvanted 2017 A/H7N9 IIV (Groups 4,5,6). The second vaccination of 2017 A/H7N9 IIV takes place approximately 21 days after the first vaccination for Groups 1 and 4 (protocol defined window of 21-28 days post first vaccination), and approximately 120 days after the first vaccination for Groups 2, 3, 5, and 6 (protocol defined window of 113-134 days post first vaccination).

#### 4.4.6. Blinding

This is a partially blinded clinical trial. Subjects, site investigators, and study personnel performing any study-related assessments following study vaccine administration to the subject are partially blinded (blinded to vaccine antigen and dosage and unblinded to vaccine administration interval). Laboratory personnel performing HAI and Neut antibody assays will receive serum specimens blinded to subject ID number and specimen visit number.

The randomization scheme will be generated by the SDCC and provided to unblinded study personnel (i.e., research pharmacists performing study vaccination preparations and unblinded study vaccine administrators) at the participating VTEU sites.

The unblinded study vaccine administrator is a study personnel member credentialed to administer vaccines and may also participate in dose preparation but will not be involved in study-related assessments or have subject contact for data collection following study vaccine administration to the subject.

The Data and Safety Monitoring Board (DSMB) may receive data in aggregate and presented by study groups. The DSMB may also be provided with expected and observed rates of the expected AEs in an unblinded fashion and may request the treatment assignment be unblinded for an individual subject if required for safety assessment. The DSMB will review grouped and unblinded data in the closed session only.

#### 4.4.7. Prior and Concomitant Therapy

Administration of any medications, therapies, or vaccines (including prescription and over-the-counter drugs as well as herbals, vitamins, and supplements) from 60 days prior to study vaccination through 21 days post final vaccination will be solicited from the participant during screening, enrollment, and follow-up. Any reported prior therapies from up to 30 days prior to vaccination through 21 days post final vaccination will be recorded in the appropriate data collection form.

Use of concomitant medications is allowed prior to and during the trial with the exception of medications and therapies that might interfere with the evaluation of the investigational product. Medications in this category include the prohibited medication per the Subject Exclusion Criteria (protocol Section 5.1.2). In addition, the site principal investigator or appropriate sub-investigator may identify other medications that should not be used due to a risk to subject safety or assessment of reactogenicity and immunogenicity.

#### 4.4.8. Treatment Compliance

All subjects are to receive two vaccinations of study product administered in the clinic based on study group assignment.

# 4.5. Immunogenicity and Safety Variables

See Table 2, Table 3, Table 4, and Table 5 for schedules of study procedures by study groups.

#### 4.5.1. Safety Variables

Safety will be assessed by the frequency and severity of:

- 1. SAEs occurring from the time of the first study vaccination through approximately 12 months after the last study vaccination.
- 2. Solicited AEs reactogenicity events occurring from the time of each study vaccination through 7 days after each study vaccination:

- Injection site reactions including pruritus, ecchymosis, erythema, induration (hardness)/edema (swelling), pain, and tenderness.
- Systemic reactions including fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea.
- 3. Clinical safety laboratory AEs occurring from the time of each study vaccination through approximately 7 days after each study vaccination. Parameters to be evaluated include white blood cells (WBC), hemoglobin (Hgb), platelets (PLT), alanine aminotransferase (ALT), total bilirubin (T. Bili), and creatinine (Cr).
- 4. Unsolicited AEs non-serious AEs occurring from the time of each study vaccination through approximately 21 days after each study vaccination.
- 5. MAAEs, including NOCMCs, and PIMMCs occurring from the time of the first study vaccination through approximately 12 months after the last study vaccination.

Grading scales for injection site and systemic solicited reactions, vital signs, and clinical laboratory parameters are provided in Table 10, Table 11, Table 12, and Table 13.

For each unsolicited AE experienced, the subject will be asked if he/she had received medical attention, defined as hospitalization, an emergency room visit or an otherwise unscheduled visit to or from medical personnel for any reason. AEs characterized by such unscheduled medical care will be designated as MAAEs.

NOCMCs are defined as any new ICD-10 diagnosis (10th revision of the International Statistical Classification of Diseases and Related Health Problems) that is applied to the subject during the course of the study, after receipt of the study agent, that is expected to continue for at least 3 months and requires continued health care intervention.

PIMMCs constitute a group of AEs that includes diseases which are clearly autoimmune in etiology and other inflammatory and/or neurologic disorders which may or may not have autoimmune etiologies. For a list of PIMMCs currently if effect, refer to protocol Appendix B.

#### 4.5.2. Immunogenicity Variables

Individual HAI and Neut results will be reported by the central immunology laboratory for the homologous 2013 A/H7N9 vaccine strain and 2017 A/H7N9 vaccine strain. Assay results are reported as a reciprocal titer with values of  $10*2^k$ , where k=0, 1, 2, etc. The lower limit of detection (LLOD) for the HAI and Neut assays is 1:10; values below the limit of detection are imputed for analysis as one-half the limit of detection (10/2 = 5). For analysis, the geometric mean (calculated on natural log scale) of repeated results for each sample will be computed and used as the response for all subsequent calculations. The variation arising from multiple measurements for an individual at a single time point is not used in subsequent calculations. See Section 3.3 for definitions of derived variables for the analysis of HAI and Neut data. HAI and Neut data will be uploaded into the SDCC's electronic data capture system.

Frequency of strain-specific (2013 and 2017 A/H7N9) plasmablasts (IgA, IgG and IgM ASCs) will be characterized by the local laboratory using freshly collected PBMCs. A single frequency value will be reported, with a LLOD of 6 and an ULOD of 8000. Values below the LOD will be reported as one-half the LLOD (6/2 = 3). Values above the ULOD will be assessed for accuracy.

A plan for receipt of exploratory data will be determined with the assaying laboratories and documented in the SAP addendum.

The assay to determine the influenza virus N9 Neuraminidase (NA) antibody response to vaccination is under development. An addendum to the SAP will be generated to outline the planned analyses when assay development is complete and after receiving confirmation of this plan from DMID.

#### 5. SAMPLE SIZE CONSIDERATIONS

This study is planned to enroll up to 180 subjects. This study is not designed to test a formal null hypothesis. Rather, it is intended to obtain sufficient data to obtain meaningful estimates of the immune response and to uncover any safety issues that occur at a sufficiently high rate that they might be observed in a study of this size. As such, the type I error rate, alpha = 0.05, is not adjusted for multiple comparisons. While this study is not designed to test any specific null hypothesis, the following tables illustrate the precision and power that is available for select estimates and comparisons of interest.

Table 6 indicates the probability of observing one or more safety events, such as solicited injection site or systemic reactogenicity events or an unsolicited non-serious AE of a particular type for a single study group (N = 30), or in the trial as a whole (N=180).

Binomial confidence intervals (CI) are widest (have the least precision) when the response rate is 50%. Table 7 is presented to indicate the worst-case scenario for precision of observed exact (Clopper-Pearson) binomial confidence intervals.

Table 8 illustrates the minimum detectable differences in the proportion of subjects responding (e.g. attaining seroconversion or a titer  $\ge 1:40$ ) between any two study groups (N=30) using a two-sided Likelihood Ratio Test and alpha = 0.05. It is assumed that up to 10% of subjects (N=3) will be excluded from the per protocol analysis. Seroconversion rates of 10% to 50% are considered.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

Unless otherwise specified, continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean and/or geometric mean (as appropriate), standard deviation, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by study vaccination and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each study group in the following order:

- Group 1: 2013 3.75 + AS03 / 2017 3.75 + AS03 (D1-D22)
- Group 2: 2013 3.75 + AS03 / 2017 3.75 + AS03 (D1-D121)
- Group 3: 2013 3.75 + AS03 / 2017 15 (D1-D121)
- Group 4: 2017 3.75 + AS03 / 2013 3.75 + AS03 (D1-D22)
- Group 5: 2017 3.75 + AS03 / 2017 3.75 + AS03 (D1-D121)
- Group 6: 2017 3.75 + AS03 / 2017 15 (D1-D121)

All tables will be annotated with the total population size relevant to that table/treatment, including any missing observations.

# **6.2.** Timing of Analyses

#### 6.2.1. CSR

Clinical, safety and reactogenicity data through approximately 180 days after the last study vaccination will represent the primary clinical database for this trial. Once the last subject completes the visit that occurs approximately 180 days after the last study vaccination and all HAI and Neut results are received and clinical data lock has occurred, a "topline" subset of the immunogenicity and safety tables will be provided to DMID on an expedited timeline. These analyses may be made available to the sponsor for planning subsequent trials and to the lead PI for publication. These analyses will not be used to make any decisions concerning the conduct of this trial. As it is anticipated that subjects may remain in long-term safety and immunogenicity follow-up at the time of these analyses, blinded site investigators and DMID Medical Monitors not involved in the analysis, publication or clinical study report (CSR) preparation will be responsible for assessing SAEs and MAAEs, including NOCMCs and PIMMCs, until all subjects have completed the final follow-up visit. All analyses of data included in the topline tables for early release will be considered the final analysis of these data, and also included in the final CSR.

Tables and figures to be included in the topline set are indicated with the symbol \* in the title.

Analysis of exploratory immunogenicity endpoints, including cellular immunology and additional serological assays, may be performed and released as the data are available from the research laboratories. Any such analyses would be considered the final analysis for the endpoint and included in the CSR.

The final CSR will be completed after the last subject's last visit is completed, and the final clinical database, including all long-term safety follow-up data, is cleaned, monitored and locked. Additional exploratory

immunogenicity endpoint data not available at the time of CSR preparation may be included in an addendum to the CSR.

# 6.3. Analysis Populations

#### **6.3.1.** Safety Population

The Safety Analysis population includes all subjects who received at least one study vaccination.

#### 6.3.2. Modified Intent-to-Treat (mITT) Population

The modified Intent-to-treat (mITT) population includes all subjects who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for immunogenicity testing (HAI or Neut antibody assays) for which valid results were reported. For analyses using the mITT population, subjects will be grouped based on randomized study group. Subject inclusion in mITT analyses will be considered individually for each assay.

#### **6.3.3.** Per Protocol Population

The per protocol (PP) population includes all subjects in the mITT subset with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent to major protocol deviations, such as:
  - Second study vaccination not received,
  - Second study vaccination received out of window,
  - Receipt of non-study licensed, live vaccine within 30 days before or after each study vaccination,
  - Receipt of non-study licensed, inactivated vaccine within 14 days before or after each study vaccination,
  - Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days before or after each study vaccination.
- Data from any visit that occurs out of window by more than one day. However, use exact window for visits that occur either 1 day or 3 days post study vaccinations:
  - Visit 2 data collected before 1 day or after 2 days post first study vaccination.
  - Visit 3 data collected before 3 days or after 4 days post first study vaccination.
  - Visit 4 data collected before 5 days or after 10 days post first study vaccination.
  - Visit 5 data collected before 12 days or after 16 days post first study vaccination.
  - Visit 6 data collected before 20 days or after 29 days post first study vaccination.
  - Visit 7 data collected before 1 day or after 2 days post second study vaccination for study groups 1 and 4.

#### - Visit 8

- ➤ Data collected before 3 days or after 4 days post second study vaccination for study groups 1 and 4.
- ➤ Data collected before 112 days or after 135 days post first study vaccination for study groups 2, 3, 5, and 6.

#### Visit 9

- ➤ Data collected before 5 days or after 10 days post second study vaccination for study groups 1 and 4.
- ➤ Data collected before 1 day or after 2 days post second study vaccination for study groups 2, 3, 5, and 6.

#### Visit 10

- ➤ Data collected before 12 days or after 16 days post second study vaccination for study groups 1 and 4.
- ➤ Data collected before 3 days or after 4 days post second study vaccination for study groups 2, 3, 5, and 6.

#### - Visit 11

- ➤ Data collected before 20 days or after 29 days post second study vaccination for study groups 1 and 4.
- ➤ Data collected before 5 days or after 10 days post second study vaccination for study groups 2, 3, 5, and 6.

#### Visit 12

- ➤ Data collected before 53 days or after 67 days post second study vaccination for study groups 1 and 4.
- ➤ Data collected before 12 days or after 16 days post second study vaccination for study groups 2, 3, 5, and 6.

#### - Visit 13

- ➤ Data collected before 75 days or after 105 days post second study vaccination for study groups 1 and 4.
- ➤ Data collected before 20 days or after 29 days post second study vaccination for study groups 2, 3, 5, and 6.

#### - Visit 15

- ➤ Data collected before 165 days or after 195 days post second study vaccination for study groups 1 and 4.
- ➤ Data collected before 75 days or after 105 days post second study vaccination for study groups 2, 3, 5, and 6.

 Visit 17 data collected before 165 days or after 195 days post second study vaccination for study groups 2, 3, 5, and 6.

For analyses using the PP population, subjects will be grouped based on study vaccinations received. Analyses will be conducted using the PP population only if 10% or more of subjects are excluded from a primary or secondary analysis timepoint.

## 6.4. Covariates and Subgroups

As a protocol defined exploratory analysis, HAI antibody response following the second vaccination will be summarized stratified by the following covariates: age (categorical: 19-34, 35-50), sex (male, female), body mass index (<30, ≥30), and prior receipt of seasonal influenza vaccine(s). Prior receipt of influenza vaccines, including any reported prior receipt of A/H5 vaccinations, or reported seasonal vaccination receipt will also be included as covariates. Summaries of prior seasonal vaccination will include breakdowns of receipt of the two seasonal vaccinations prior to study initiation (did not receive 2016-2017 or 2018-2019; received 2016-2017 and/or 2018-2019) as well as independently assessing subject receipt of 2018-2019 seasonal vaccine (did not receive/received) prior to the second dose of study vaccine. These covariates will be considered in statistical modeling as described in Section 8.3. As these analyses are exploratory, the study was not powered for any subgroup analyses.

# 6.5. Missing Data

All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If data points are identified as outliers, sensitivity analyses will be performed to examine the impact of including or excluding the outliers. Any substantive differences in these analyses will be reported.

# 6.6. Interim Analyses and Data Monitoring

Interim analyses will only be used to terminate this trial in the event that unanticipated safety events deemed to be of sufficient concern require such action by the sponsor. These assessments will not be made on the basis of testing a formal statistical hypothesis; therefore, p-value adjustment will not be made to any analyses. A DSMB will be convened by DMID to review study progress and participant, clinical, safety, and reactogenicity and immunogenicity data.

Emergent public health needs may dictate additional interim safety, reactogenicity, and/or immunogenicity analyses be performed on available information at any time during the trial. If this occurs, immunogenicity data will be analyzed as results are available from the central immunogenicity laboratory.

#### **6.6.1.** Interim Safety Review

An interim safety review may include enrollment and demographic information, medical history, concomitant medications, physical assessments, clinical laboratory values, dosing compliance, and solicited and unsolicited AE/SAEs. Additional data may be requested by the DSMB, and interim statistical reports may be generated as deemed necessary and appropriate by DMID. The DSMB may receive data in aggregate and presented by study group. The DSMB may also be provided with expected and observed rates of the expected AEs in an unblinded fashion and may request the treatment assignment be unblinded for an individual subject if required for safety assessment. The DSMB will review grouped and unblinded data in the closed session

only. The DSMB will meet and review this data at trial-specific time frames or ad hoc as needed during this trial as defined in the DSMB charter. As an outcome of each review/meeting, the DSMB will make a recommendation as to the advisability of proceeding with study vaccinations, as applicable, and to continue, modify or terminate this trial.

The interim safety reports generated for the DSMB are not intended to be published; they will be used only for informing emergency preparedness.

Additionally, this trial will be monitored to determine if any of the halting rules described in Protocol Section 9.5 are met.

### 6.6.2. Interim Immunogenicity Review

No interim immunogenicity analysis is planned. Should emergent public health needs dictate interim immunogenicity review, immune responses will be summarized in terms of strain-specific 2013 and 2017 A/H7N9 HAI and Neut antibody titers and the relationship to study vaccine dosage, adjuvant use and study vaccination schedule. It is anticipated that all analyses will be carried out in parallel for both assays, but reports may be prepared separately for HAIs and Neuts if results are available on different timelines. Interim analyses will focus on rates of titers ≥1:40, seroconversion (see definition in Section 3.3) and GMTs, along with corresponding 95% CIs. No formal hypothesis testing will be included in the interim analysis, and interim results will not have impact on conduct of this trial. All interim analyses will use the mITT population.

Any immunogenicity reports would be provided by the SDCC to the DMID Scientific Lead, DMID Clinical Project Manager and DSMB. Reports will include data summarized by unblinded study group, but the presentation will be in a format that prevents inadvertent unblinding of any individual subject.

There is no plan to halt this trial prior to full enrollment and completion of all follow-up visits based on any interim immunogenicity results.

#### 6.7. Multicenter Studies

Randomization was stratified by site, but data will be pooled across all clinical sites for all analyses. Center effects are not anticipated because the sites use standardized procedures for vaccination and assessment of solicited and unsolicited AEs, and the study relies on a central laboratory for immunogenicity assessments.

# 6.8. Multiple Comparisons/Multiplicity

This study was designed to obtain preliminary estimates of safety and immune response to the 2013 and 2017 A/H7N9 vaccinations in healthy adults. The study was not designed to test any specific null hypothesis, and as such no adjustment for multiple comparisons will be performed.

#### 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

Table 14 will present a summary of the reasons that subjects were screened but not enrolled.

The number and percentage of enrolled subjects excluded from each analysis population by study group are presented in Table 15. A listing of subjects excluded from each analysis population will be presented in Listing 5.

The disposition of subjects in the study will be tabulated by study group (Table 16). The table will show the total number of subjects screened, randomized, receiving the first vaccination, receiving the second vaccination, completing the blood draw for the primary immunogenicity endpoints, and completing the last visit.

A flowchart showing the disposition of study subjects, adapted from the CONSORT Statement [4] will be included and will present the number of subjects screened, randomized, lost to follow up, and analyzed, by study group (Figure 1).

A listing of subjects who were discontinued from treatment or terminated from study follow-up and the reason will be included in Listing 2.

#### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the deviation category and deviation type, and study group for all enrolled subjects (Table 9). Major deviations that will be reviewed for possible exclusion of immunogenicity results from the PP population include deviations related to eligibility/enrollment, treatment administration schedule, follow-up visit schedule, and receipt of exclusionary vaccines or medications. All subject-specific protocol deviations and non-subject-specific protocol deviations will be included in Listing 3 and Listing 4.

#### 8. IMMUNOGENICITY EVALUATION

Immunogenicity data summaries and analysis for primary and secondary endpoints will be presented for the mITT population, which is the primary population for analysis. The Per Protocol population displays will be generated only if >10% of subjects are found to have data excluded from a primary or secondary timepoint. Immune responses in terms of strain-specific 2013 and 2017 A/H7N9 HAI and Neut antibody titers will be summarized by study group at each time point. Descriptive summary statistics will be provided for all assays and time points including number of subjects with non-missing results, percentage of subjects with titers ≥1:40, percentage of subjects achieving seroconversion, and GMTs along with corresponding 95% CI. Exact confidence intervals will be presented for proportional endpoints. Summaries of primary and secondary immunogenicity endpoints are presented for the 2013 A/H7N9 strain in Table 24, Table 25, Table 26, and Table 27 and for the 2017 A/H7N9 strain in Table 28, Table 29, Table 30, and Table 31.

Reverse cumulative distribution (RCD) curves will be presented for post-vaccination HAI and Neut antibody titers. Plots for each assay will be generated with 3 columns (Day 22 post vaccination 1, Day 22 post vaccination 2, and Day 181 post vaccination 2) and 2 rows (2013 A/H7N9, 2017 A/H7N9), and separate curves within each panel for each study group, as shown in Figure 2, Figure 3, Figure 4, and Figure 5.

Figure 8, and Figure 9 for both 2013 and 2017 A/H7N9 strains.

The spearman correlation between HAI and Neut antibody titers will be calculated at each time point over all groups. The correlation will be depicted in scatter plots as Figure 10 and Figure 11 for both the 2013 and 2017A/H7N9 strain.

Individual HAI and Neut assay results will be provided in Listing 9.

# 8.1. Primary Immunogenicity Analysis

The primary immunogenicity endpoints HAI and Neut seroconversion, percentage of subjects with titer ≥1:40, and GMTs against the 2013 and 2017A/H7N9 vaccine strains 21 days after the second vaccination will be summarized as described above. The primary analysis population will be mITT, with results from the PP population providing a comparison of the sensitivity of immunogenicity results to subject adherence to protocol-defined conditions. Regression modelling of seroconversion and log titers is planned as described in Section 8.3.2.

# 8.2. Secondary Immunogenicity Analyses

The secondary immunogenicity endpoints HAI and Neut seroconversion, percentage of subjects with titer ≥40, and GMTs against the 2013 and 2017 A/H7N9 vaccine viruses prior to each study vaccination, 21 days after the first vaccination and 180 days after the second vaccination will be summarized as described above. No formal hypothesis testing is planned.

# 8.3. Exploratory Immunogenicity Analyses

Exploratory immunogenicity data summaries and analysis for exploratory endpoints will be presented for the PP population if >10% of subjects are found to have data excluded from a primary or secondary timepoint. Otherwise, exploratory displays will be presented for the modified intent to treat population.

#### 8.3.1. HAI and Neut Covariate Analysis

As an exploratory analysis, seroconversion and GMT of serum antibody for both HAI and Neut against the homologous 2013 A/H7N9 strain at 21 and 180 days after the second study vaccination will be summarized by study group stratified by age (categorized as those subjects ages 19-34, 35-50 years) (Table 32, Table 33, Table 34, and Table 35), by sex (Table 40, Table 41, Table 42, and Table 43), by BMI (Table 48, Table 49, Table 50, and Table 51), and by prior receipt of the 2016-2017 and/or 2017-2018 and /or 2018-2019 seasonal influenza vaccines (Table 56, Table 57, Table 58, and Table 59). These analyses will be repeated for HAI and Neut titer results against the 2017 A/H7N9 strain at 21 and 180 days post receipt of the second study vaccination by age category (Table 36, Table 37, Table 38, and Table 39) by sex (Table 44, Table 45, Table 46, and Table 47), by BMI (Table 52, Table 53, Table 54, and Table 55) by prior receipt of seasonal influenza vaccine (Table 60, Table 61, Table 62, and Table 63).

The stratified summaries will be presented for the PP population. It is anticipated that subjects will have little to no pre-existing antibody at baseline, so seroconversion and titer  $\geq$ 40 endpoints will be similar.

#### 8.3.2. HAI and Neut Regression Modeling

Regression modeling will be utilized to test for the effect of treatment variables i.e. prime boost combination (PrimeBoost), Boost dose (BoostDose), and interval between vaccinations (Interval), on immune response. Logistic regression will be fit for the seroconversion outcome. If the available titer data meet the required assumptions of normality after log transformation, multiple linear regression will be fit to log-transformed titers. Separate models will be fit for each assay (HAI, Neut), each strain (2013 A/H7N9, 2017 A/H7N9) and each time point (Day 22 post vaccination 1, Day 22 post vaccination 2, Day 181 post vaccination 2). All models will be fit with a similar structure for *PrimeBoost*, *BoostDose*, *Interval*, and covariates, for the PP population. The treatment variables will be defined as *PrimeBoost* (homologous, heterologous), *BoostDose* (3.75 mcg+AS03, 15 mcg), and *Interval* (21 days, 120 days). All models will be fit with and without adjustment for the following covariates (Z): age in years, sex (female, male), BMI ( $<30, \ge 30$ ), and prior receipt of seasonal influenza vaccine in the current season (did not receive 2018-2019 seasonal influenza vaccine, received 2018-2019 seasonal influenza vaccine) (did not receive 2016-2017 or 2017-2018 seasonal influenza vaccines, received 2016-2017 and/or 2017-2018 seasonal influenza vaccine). The models as shown below assume a linear relationship between age in years and both probability of seroconversion and GMT. The validity of this assumption will be assessed prior to analysis and, if the relationship between age and response is found to be non-linear, adjustments will be made to model parameters to satisfy regression assumptions. Modeling assumptions will be checked using standard diagnostic methods (e.g., using the INFLUENCE option in PROC LOGISTIC or PROC GLM). Parameter estimates and odds ratio estimates for the logistic models will be presented for the 2013 and 2017 A/H7N9 strains without covariate adjustment in Table 64, Table 65, Table 66, Table 67, and with covariate adjustment in Table 68, Table 69, Table 70, Table 71. Parameter estimates for the multiple linear regression models will be presented for the 2013 and 2017 A/H7N9s strain without covariate adjustment in Table 72, Table 73, Table 74, Table 75, and with covariate adjustment in Table 76, Table 77, Table 78, Table 79.

Model 1A: Logistic Regression (without covariate adjustment):

```
\begin{split} logit[P(seroconversion)] &= \beta_0 + \beta_1 \times PrimeBoost + \beta_2 \times BoostDose + \beta_3 \times Interval \\ &+ \beta_4 \times (PrimeBoost * BoostDose) + \beta_5 \times (PrimeBoost * Interval) + \varepsilon \end{split}
```

Model 1B: Logistic Regression (with covariate adjustment):

logit[P(seroconversion)]

$$= \beta_0 + \beta_1 \times PrimeBoost + \beta_2 \times BoostDose + \beta_3 \times Interval \\ + \beta_4 \times (PrimeBoost * BoostDose) + \beta_5 \times (PrimeBoost * Interval) + \beta_6 \times Z + \varepsilon$$

Model 2A: Multiple Linear Regression (without covariate adjustment):

$$log(titer) = \beta_0 + \beta_1 \times PrimeBoost + \beta_2 \times BoostDose + \beta_3 \times Interval + \beta_4 \times (PrimeBoost * BoostDose) + \beta_5 \times (PrimeBoost * Interval) + \varepsilon$$

Model 2B: Multiple Linear Regression (with covariate adjustment):

$$log(titer) = \beta_0 + \beta_1 \times PrimeBoost + \beta_2 \times BoostDose + \beta_3 \times Interval + \beta_4 \times (PrimeBoost * BoostDose) + \beta_5 \times (PrimeBoost * Interval) + \beta_6 \times Z + \varepsilon$$

Where Z is the matrix of covariates age, sex, BMI, and prior receipt of seasonal influenza vaccine as defined in Section 6.4. Subjects missing data for one or more covariates will be excluded from Models 1B and 2B.

#### 8.3.3. Antibody Secreting Cells (Plasmablasts)

Due to the requirement for freshly isolated PBMCs, the plasmablast (antibody secreting cell [ASC]) assay will be performed only on specimens collected from subjects enrolled at Emory Children's Center and the Hope Clinic of Emory Vaccine Center. Values below the lower limit of detection will be handled as described in Section 4.5.2. The frequency of strain-specific 2013 and 2017 A/H7N9 IgA, and IgG ASCs will be summarized for the mITT and PP populations by study group at 8 days post each study vaccination. Descriptive summary statistics will be provided for both time points including the number of subjects with non-missing results, mean, standard deviation and corresponding 95% CI as well as median, minimum and maximum values. Geometric mean and 95% CI may also be assessed depending on the observed distribution of the data. Summaries are presented for the 2013 A/H7N9 strain in Table 80 and for the 2017 A/H7N9 strain in Table 81.

Box and whisker plots will summarize the distribution of ASC results for each immunoglobulin type, strain, and study day (Figure 12, Figure 13, Figure 14, Figure 15, Figure 16, Figure 17). Scatterplot matrices depicting the relationship and correlation between immunoglobulin types for the strain-specific ASCs at the same day, as well as between the same immunoglobulin types post each study vaccination, will be shown in Figure 18, Figure 19, Figure 20, Figure 21, Figure 22, Figure 23, Figure 24 and Figure 25. Strain-specific ASC frequency at 8 days post vaccination will also be correlated with HAI and Neut titer at 21 days post vaccination as shown in Figure 22, Figure 23, Figure 24, and Figure 25. The statistician will determine if the Pearson or the Spearman Rank-Order correlation is appropriate at the time of analysis.

#### 8.3.4. Other Assays

Descriptions of the NA assays and all other exploratory assays and the associated planned analyses will be described in an addendum to this SAP.

#### 9. SAFETY EVALUATION

All summaries and analysis of safety data will be presented for the Safety Analysis Population. Safety summaries will be presented overall and grouped by study group.

Continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. All categorical measures will be summarized by the frequency and percentages of observed levels will be reported for all categorical measures. The denominator for the percentages may be based on the number of non-missing observations for an assessment or based on the number of subjects in a population. This will be described for each table.

## 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, race, BMI, and prior receipt of seasonal influenza vaccine will be presented by site (Table 19, Table 20) and by study group (Table 21, Table 22). Age will be summarized as a continuous variable. Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the electronic case report form (eCRF) as "No" to each racial option. BMI will be summarized as a continuous as well as categorical variable, categorized as (<30, ≥30). Self-reported history of prior receipt of influenza vaccines will be broken down by the following categories: receipt of seasonal vaccines for prior seasons (2016-2017, 2017-2018), receipt of seasonal vaccine for the current season (2018-2019; considered up to receipt of study dose 2), and receipt of any A/H5 vaccines prior to enrollment. Demographic information for individual subjects will be provided in Listing 6. Subjects' prior influenza vaccination history (seasonal and non-seasonal) will be provided in Listing 8.

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past or pre-existing medical conditions will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 20.0 or higher.

Summaries of subjects' prior and concurrent medical conditions will be presented by study group (Table 23). Individual subject listings will be presented for all reported medical history including prior and concurrent medical conditions (Listing 7).

#### 9.1.2. Prior and Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of concomitant medications during the study will be summarized by ATC1 and ATC2 code and study group for the Safety population (Table 132). A listing of concomitant medications will be presented (Listing 18).

# **9.2.** Measurements of Treatment Compliance

All subjects are to receive 2 study vaccinations administered in the clinic. The number of study vaccinations administered to subjects will be presented by study group in Table 17 and Table 18 and as part of the subject disposition tables (Table 16). Listing 1 presents subjects who received investigational product with study group and study product received for each vaccination.

#### 9.3. Adverse Events

A summary of all adverse events is provided in Table 82. A summary of those events that occurred in  $\geq$ 5% of subjects in any study group is provided in Table 83.

#### 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-vaccination, and systemic and local solicited adverse events were collected at-least 20 minutes post-vaccination and then daily for 7 days after each vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea. The grading scale for systemic events, including quantitative grading for fever, is included in Table 11. Local events include pruritus, ecchymosis, erythema, induration/swelling, pain, and tenderness. Ecchymosis, erythema, and induration are measured by both functional and measurement grading scales as defined in Table 10.

When calculating the incidence of solicited events, each subject will be counted once at the highest severity following the applicable vaccination, and any repetitions will be ignored. For summaries presented separately for each vaccination, the denominator for percentages will be the number of subjects who received the respective vaccination with non-missing data for the event summarized. For summaries over all vaccinations the denominator will be the number of subjects who received at least one vaccination with non-missing data for the event summarized.

The number and percentage of subjects reporting at least one solicited adverse event of each severity will be summarized for each solicited symptom, any systemic symptom, any local symptom, and any symptoms. For each event the denominator is the number of subjects who received the applicable vaccination with non-missing data for the specific event. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (Table 84, Table 85, Table 86). Logistic regression models will be fit to estimate the effect of prime-boost combination (*PrimeBoost*), Boost dose (*BoostDose*), and interval between vaccinations (*Interval*) on the probability of reporting any local event or reporting any systemic event after either vaccination (Table 87, Table 88). If statistically significant effects are observed in the model for local events or systemic events, then additional models will be fit for each individual event of that type.

```
logit[P(Event)] = \beta_0 + \beta_1 \times PrimeBoost + \beta_2 \times BoostDose + \beta_3 \times Interval + \beta_4 \times (PrimeBoost * BoostDose) + \beta_5 \times (PrimeBoost * Interval) + \varepsilon,
```

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the Safety population. The number and percentage of subjects reporting each event will be summarized by the maximum severity and study group, separately for each vaccination and over both vaccinations. For each event the denominator is the number of subjects who received the applicable vaccination with non-missing data for the specific event. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (Table 89, Table 90, Table 91).

The number of subjects reporting a solicited adverse event will be summarized for each day post vaccination for each vaccination and for both vaccinations combined both in a summary table (Table 92, Table 93, Table 94) and graphically in a bar chart (Figure 26 and Figure 27). A comparison of the event rate for each study group between study vaccinations will be presented, including p-values from McNemar's test performed (Table 95, Table 96).

Systemic and Local solicited events reported by subject will be presented in Listing 11 and Listing 12, sorted by subject ID, vaccination number, parameter, and study day.

#### 9.3.2. Unsolicited Adverse Events

When calculating the incidence of unsolicited AEs (i.e., on a per subject basis), each subject will only be counted once at the highest severity and/or relationship, and any repetitions of AEs within a subject will be ignored; the denominator will be the total number of subjects in the safety population. All AEs reported will be included in the summaries and analyses.

The number and percentage of subjects reporting at least one unsolicited AE will be summarized by MedDRA system organ class and preferred term. A 95% CI will be presented for the percentage of subjects reporting any unsolicited AE (serious or non-serious) for each MedDRA system organ class and preferred term over all study vaccinations (Table 97).

The following summaries for unsolicited AEs will be presented by MedDRA system organ class, preferred term, and study group:

- Incidence of AEs by severity and relationship to study product (Table 98, Table 99);
- Incidence of non-serious, related AEs by severity (Table 100, Table 101);
- Incidence of AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 102);
- Incidence of non-serious, related AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 103) note this table presents results for secondary safety endpoint, "Occurrence of study vaccine-related unsolicited non-serious AEs from the time of each study vaccination through approximately 21 days after each study vaccination";
- Total frequency of AEs over time (Days 1-8, Day 9 through approximately Day22 post each study vaccination) (Table 104, Table 105);
- Subject listing of non-serious AEs of moderate or greater severity (Table 110);
- Bar chart displaying total frequency of AEs by severity and MedDRA system organ class and study group (Figure 28, Figure 29);
- Bar chart displaying incidence of AEs by severity and MedDRA system organ class, and study group (Figure 30, Figure 31);
- Bar chart displaying total frequency and incidence of AEs by relationship to study product, MedDRA system organ class, and study group (Figure 32, Figure 33, Figure 34, Figure 35).

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Age (years) AE Description, AE Onset Date/End Date, Last Vaccination Received/Days Post Vaccination, Reason Reported as an SAE, Relationship to Study Vaccination, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 106);
- Medically Attended Adverse Events (Table 107);
- Potentially Immune Mediated Medical Conditions (Table 108);

New Onset Chronic Medical Conditions (Table 109).

A listing of all reported AEs by subject will be presented in Listing 13, sorted by Study Group, Subject ID, and AE Number.

## 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery.

Listing 19, Listing 20, Listing 21, Listing 22, and Listing 23 will present any study pregnancies and their outcomes.

# 9.6. Clinical Laboratory Evaluations

Clinical safety laboratory parameters (WBC, Hgb, PLT, ALT, T. Bili, Cr) will be collected from each subject prior to each study vaccination and approximately 7 days after each study vaccination. These evaluations will be performed by the central clinical laboratory. The grading scale for clinical laboratory evaluations is presented in Table 13. Clinical laboratory evaluations assessed on Day 1 prior to the first study vaccination will be considered as baseline. Safety laboratory parameters are allowed to be repeated at the central clinical laboratory one time per protocol for AE follow-up, after which follow-up is required to be done at the site's local laboratory, if needed. Results from safety laboratories run locally are not included in any exhibits but rather are used to inform subject safety and may be included in unsolicited adverse event comments, if applicable.

The distribution of laboratory results by severity, study day and study group will be presented in Table 111, Table 112, Table 113, Table 114, Table 118, Table 119, Table 120, and Table 121. Descriptive statistics including mean, standard deviation, median, minimum and maximum values and change from baseline by study day will be summarized for each parameter in Table 115, Table 116, Table 117, Table 122, Table 123, and Table 124. Box plots illustrating the change from baseline for each laboratory parameter will be presented in Figure 36, Figure 37, Figure 38, Figure 39, Figure 40, and Figure 41. Subject visits with abnormal laboratory results, Grade 1 severity or higher, will be presented in Table 125 and Table 126 for Chemistry and Hematology parameters, respectively.

A complete listing of individual clinical laboratory results will be presented in Listing 14 and Listing 15 for chemistry and hematology, respectively, sorted by subject ID, parameter, and visit number.

# 9.7. Vital Signs and Physical Evaluations

Vital signs oral temperature, systolic blood pressure, diastolic blood pressure, and pulse will be assessed prior to study vaccination on Days 1 and 22 for study groups 1 and 4 and on Days 1 and 121 for study groups 2, 3, 5, and 6. The grading scale for vital sign evaluations is presented in Table 12. Summaries of vital signs by maximum severity will be tabulated by visit, and study group (Table 127, Table 128, Table 129, Table 130, Table 131). A listing of vital signs will be presented (Listing 16).

Targeted physical examinations will be performed, if indicated, based a subject's medical history. A listing of physical exam findings will be presented (Listing 17).

# 9.8. Concomitant Medications

Concomitant medications will be collected for the 30 days prior to the first study vaccination through 21 days after the second study vaccination. Concomitant medications will be coded to the Anatomical Therapeutic Classification (ATC) using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented (Listing 18). The use of concomitant medications during the study will be summarized by ATC1, ATC2 code, study group for the Safety population (Table 132).

## 10. REPORTING CONVENTIONS

P-values ≥0.001 and ≤0.999 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001"; p-values greater than 0.999 will be reported as "> 0.999". The mean, standard deviation, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles, such as median, or minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as two decimal places; values <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; non-zero values < 1% will be presented as "<1%"; values greater than 99% but less than 100% will be presented as ">99%". Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

# 11. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

# 12. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

This SAP does not include any changes from the analyses described in the protocol.
#### 13. REFERENCES

- 1. Gao, R., et al., Human infection with a novel avian-origin influenza A (H7N9) virus. N Engl J Med, 2013. 368(20): p. 1888-97.
- 2. Analysis of recent scientific information on avian influenza A(H7N9) virus. WHO Influenza Update, 2017.
- 3. Human infection with avian influenza A(H7N9) virus China: 18 May 2017. WHO Emergencies preparedness, response, 2017.
- 4. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.
- 5. FDA Guidance for Industry: Clinical Data Needed to Support the Licensure of Seasonal Inactivated Influenza Vaccines (US DHHS, FDA, CBER, May 2007).

# 14. APPENDICES

Table, figure, and listing shells are presented in Appendices 1, 2, and 3. Tables included in the topline set are indicated by \*.

# APPENDIX 1. TABLE MOCK-UPS

# LIST OF TABLES

| Table 1: | Study Design |
|---|---|
| Table 2: | Schedule of Study Procedures – Vaccination Period for Study Groups 1 and 449 |
| Table 3: | Schedule of Study Procedures – Follow-Up Period for Study Groups 1 and 4 (Including early termination and unscheduled visits) |
| Table 4: | Schedule of Study Procedures – Vaccination Period for Study Groups 2, 3, 5, and 656 |
| Table 5: | Schedule of Study Procedures – Follow-Up Period for Study Groups 2, 3, 5, and 6 (Including early termination and unscheduled visits) |
| Table 6: | Power (%) to Detect Safety Events |
| Table 7: | Precisions of Binomial Confidence Intervals |
| Table 8: | Minimum Detectable Difference in Proportion Responders |
| Table 9: | Distribution of Protocol Deviations by Category, Type, and Study Group65 |
| Table 10: | Solicited Adverse Event Grading Scale – Local |
| Table 11: | Solicited Adverse Event Grading Scale - Systemic |
| Table 12: | Vital Signs Adverse Event Grading Scale |
| Table 13: | Laboratory Adverse Event Grading Scale |
| Table 14: | Ineligibility Summary of Screen Failures |
| Table 15: | Analysis Populations by Study Group – All Enrolled Subjects |
| Table 16: | Subject Disposition by Study Group, All Enrolled Subjects |
| Table 17: | Dates of First Study Vaccination by Site and Study Group |
| Table 18: | Dates of Second Study Vaccination by Site and Study Group |
| Table 19: | Summary of Categorical Demographic and Baseline Characteristics by Site, All Enrolled Subjects |
| Table 20: | Summary of Continuous Demographic and Baseline Characteristics by Site, All Enrolled Subjects |
| Table 21: | Summary of Categorical Demographic and Baseline Characteristics by Study Group, All Enrolled Subjects |
| Table 22: | Summary of Continuous Baseline Characteristics by Study Group, All Enrolled Subjects |
| Table 23: | Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA® System Organ Class and Study Group, Safety Population |
| Table 24: | Summaries of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population*87 |
| Table 25: | Summaries of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Per Protocol Population* |

| Table 26: | Summaries of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population*89 |
|---|---|
| Table 27: | Summaries of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Per Protocol Population* |
| Table 28: | Summaries of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population*89 |
| Table 29: | Summaries of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Per Protocol Population* |
| Table 30: | Summaries of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population* |
| Table 31: | Summaries of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Per Protocol Population* |
| Table 32: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population |
| Table 33: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 34: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population91 |
| Table 35: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 36: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population |
| Table 37: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 38: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population91 |
| Table 39: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 40: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population |

| Table 41: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 180 Days Post Second Vaccination, Per Protocol Population |
|---|---|
| Table 42: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population93 |
| Table 43: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 180 Days Post Second Vaccination, Per Protocol Population93 |
| Table 44: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population |
| Table 45: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 46: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population93 |
| Table 47: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 180 Days Second Vaccination, Per Protocol Population93 |
| Table 48: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population |
| Table 49: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 50: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population95 |
| Table 51: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 180 Days Post Second Vaccination, Per Protocol Population95 |
| Table 52: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population |
| Table 53: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 54: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population95 |
| Table 55: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 180 Days Second Vaccination, Per Protocol Population95 |

| Table 56: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Seasonal Influenza Vaccination Status at 21 Days Post Second Vaccination, Per Protocol Population |
|---|---|
| Table 57: | Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 58: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study<br>Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per<br>Protocol Population |
| Table 59: | Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 60: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per Protocol Population |
| Table 61: | Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per Protocol Population |
| Table 62: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per Protocol Population |
| Table 63: | Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Second Vaccination, Per Protocol Population |
| Table 64: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Per Protocol Population |
| Table 65: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Per Protocol Population |
| Table 66: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Per Protocol Population |
| Table 67: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Per Protocol Population |
| Table 68: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population (N=X)100 |

| Table 69: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population101 |
|---|---|
| Table 70: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population |
| Table 71: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population101 |
| Table 72: | Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Per Protocol Population (N=X) |
| Table 73: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 180 Days Post Second<br>Study Vaccination, Per Protocol Population |
| Table 74: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 21 Days Post Second<br>Study Vaccination, Per Protocol Population |
| Table 75: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 180 Days Post<br>Second Study Vaccination, Per Protocol Population |
| Table 76: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 21 Days Post Second<br>Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population103 |
| Table 77: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 180 Days Post Second<br>Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population104 |
| Table 78: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 21 Days Post Second<br>Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population104 |
| Table 79: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 180 Days Post<br>Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population<br> |
| Table 80: | Summary of A/Shanghai/2/2013 (A/H7N9)–Specific Antibody Secreting Cells by Immunoglobulin Type, Study Group, and Study Day, Per Protocol Population105 |
| Table 81: | Summary of A/Hong Kong/125/2017 (A/H7N9)–Specific Antibody Secreting Cells by Immunoglobulin Type, Study Group, and Study Day, Per Protocol Population106 |
| Table 82: | Overall Summary of Adverse Events, Safety Population*107 |

| Table 83: | Number of Adverse Events Occurring in 5% of Subjects in Any Study Group by MedDRA® System Organ Class and Preferred Term, and Study Group, Safety Population |
|---|---|
| Table 84: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Study Group (Safety Population) – Post Any Study Vaccination |
| Table 85: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Study Group (Safety Population) – Post Study Vaccination 1 |
| Table 86: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Study Group (Safety Population) – Post Study Vaccination 2 |
| Table 87: | Logistic Regression Model to Evaluate the Relationship of Study Vaccination with Reporting Any Local Event Post Second Study Vaccination, Safety Population113 |
| Table 88: | Logistic Regression Model to Evaluate the Relationship of Study Vaccination with Reporting Any Systemic Event Post Second Study Vaccination, Safety Population113 |
| Table 89: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Study Group (Safety Population) – Post Any Study Vaccination |
| Table 90: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Maximum Severity and Study Group (Safety Population) – Post Study Vaccination 1119 |
| Table 91: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Maximum Severity and Study Group (Safety Population) – Post Study Vaccination 2119 |
| Table 92: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, and Study Group (Safety Population) – Post Any Study Vaccination |
| Table 93: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Severity, Day Post Study Vaccination, and Study Group (Safety Population) – Post Study<br>Vaccination 1 |
| Table 94: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Severity, Day Post Study Vaccination, and Study Group (Safety Population) – Post Study<br>Vaccination 2 |
| Table 95: | Number and Percentage of Subjects Experiencing Solicited Systemic Events for Study Vaccination 1 Compared with Study Vaccination 2 by Study Group—Safety Population |
| Table 96: | Number and Percentage of Subjects Experiencing Solicited Local Events for Study Vaccination 1 Compared with Study Vaccination 2 by Study Group, Safety Population |

| Table 97: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Study Group, Safety Population* |
|---|---|
| Table 98: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship, and Study Group, Safety Population |
| Table 99: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events within 21 Days of Study Vaccination by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship, and Study Group, Safety Population |
| Table 100 | Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Study Group, Safety Population |
| Table 101: | Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Study Group, Safety Population133 |
| Table 102: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA® System Organ Class and Preferred Term, Day Post Study Vaccination, and Study Group, Safety Population |
| Table 103: | Number and Percentage of Subjects Experiencing Non-Serious, Related Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA® System Organ Class and Preferred Term, Vaccination and Study Group, Safety Population135 |
| Table 104: | Number of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Day Post Study Vaccination, and Study Group, Safety Population136 |
| Table 105: | Number of Non-Serious, Related, Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Day Post Study Vaccination, and Study Group, Safety Population |
| Table 106: | Listing of Serious Adverse Events – Safety Population * |
| Table 107: | Listing of Medically Attended Adverse Events – Safety Population138 |
| Table 108: | Listing of Potentially Immune Mediated Medical Conditions |
| Table 109: | Listing of New Onset Chronic Medical Conditions |
| Table 110: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events138 |
| Table 111: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – All Chemistry Parameters– Safety Population140 |
| Table 112: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – Alanine aminotransferase (ALT)142 |
| Table 113: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – Total Bilirubin |
| Table 114: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) Creatining |

| Table 115: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Alanine Aminotransferase (ALT)143 |
|---|---|
| Table 116: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Total Bilirubin |
| Table 117: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Creatinine |
| Table 118: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – All Hematology Parameters |
| Table 119: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – Hemoglobin |
| Table 120: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – White Blood Cells |
| Table 121: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – Platelets |
| Table 122: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Hemoglobin |
| Table 123: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – White Blood Cells |
| Table 124: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Platelets |
| Table 125: | Listing of Abnormal Laboratory Results - Chemistry |
| Table 126: | Listing of Abnormal Laboratory Results - Hematology |
| Table 127: | Vital Signs by Assessment, Maximum Severity, Study Day, Study Group (Safety Population) – Any Assessment |
| Table 128: | Vital Signs by Assessment, Maximum Severity, Study Day, Study Group (Safety Population) – Oral Temperature |
| Table 129: | Vital Signs by Assessment, Maximum Severity, Study Day, and Study Group (Safety Population) – Systolic Blood Pressure |
| Table 130: | Vital Signs by Assessment, Maximum Severity, Study Day, and Study Group (Safety Population) – Diastolic Blood Pressure |
| Table 131: | Vital Signs by Assessment, Maximum Severity, Study Day, and Study Group (Safety Population) – Pulse |
| Table 132: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Study Group |

# 9.1 Overall Study Design and Plan Description

Table 1: Study Design

| Influenza A/H7<br>Vaccine/Infection Naïve<br>Subjects (Total N=180) | | Study<br>Group/N | 1st Study Vaccination Day 1 | 2 <sup>nd</sup> Study<br>Vaccination<br>~ Day 22 post<br>Vaccination 1 | 2 <sup>nd</sup> Study Vaccination<br>~ Day 121 post<br>Vaccination 1 |
|---|---|---|---|---|---|
| | | 1/30 | 2013 A/H7N9 IIV 3.75<br>mcg + AS03 | 2017 A/H7N9 IIV<br>3.75 mcg + AS03 | |
| | Heterologous<br>Prime-Boost | 2/30 | 2013 A/H7N9 IIV 3.75<br>mcg + AS03 | | 2017 A/H7N9 IIV 3.75<br>mcg + AS03 |
| Study<br>Vaccination | | 3/30 | 2013 A/H7N9 IIV 3.75<br>mcg + AS03 | | 2017 A/H7N9 IIV<br>15 mcg |
| Schedule | | 4/30 | 2017 A/H7N9 IIV 3.75<br>mcg + AS03 | 2017 A/H7N9 IIV<br>3.75 mcg + AS03 | |
| | Homologous<br>Prime-Boost | 5/30 | 2017 A/H7N9 IIV 3.75<br>mcg + AS03 | | 2017 A/H7N9 IIV 3.75<br>mcg + AS03 |
| | | 6/30 | 2017 A/H7N9 IIV 3.75<br>mcg + AS03 | | 2017 A/H7N9 IIV<br>15 mcg |

### 9.5.1 Immunogenicity and Safety Measurements Assessed and Flow Chart

Table 2: Schedule of Study Procedures – Vaccination Period for Study Groups 1 and 4

| Study Visit Number | 000 | V01 | V02 | V03 | V04 | V05 | 901 | V07 | V08 | 601 | V10 | V111 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D23 | D25 | D29 | D36 | D43 |
| Study Day post second study vaccination | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |
| | Study Pr | ocedure/Eval | uation | | • | | | | | l . | | l. |
| Informed $Consent^{\infty}$ | X | X <sup>†</sup> ¬ | | | | | | | | | | |
| Demographic Information | X | $X^{\dagger^*}$ | | | | | | | | | | |
| Eligibility Criteria | X | $X^{\dagger - 1}$ | | | | | $X^{\dagger 1}$ | | | | | |
| Medical History@ | X | X <sup>†</sup> ¬ | X | X | X | X | $X^{\dagger}$ | X | X | X | X | X |
| Concomitant Medications <sup>c</sup> | X | X <sup>†</sup> ¬ | X | X | X | X | $X^{\dagger}$ | X | X | X | X | X |
| Vital Signs (Oral Temperature%, Pulse and BP) | X | X <sup>†\$</sup> | | | | | $X^{\dagger 2}$ | | | | | |
| Height and Weight | X | $X^{\dagger^*}$ | | | | | | | | | | |
| Physical Examination | $X^3$ | X <sup>†3*{}</sup> | {X} | {X} | {X} | {X} | $\{X\}^{\dagger}$ | {X} | {X} | {X} | {X} | {X} |
| Urine or Serum Pregnancy Test | X^ | $X^{\dagger ^{\wedge}}$ | | | | | $X^{\dagger^{\wedge}}$ | | | | | |
| Venous Blood Collection for ESR | $X^{\neq}$ | $X^{\neq *}$ | | | | | | | | | | |
| Enrollment in AdvantageEDCSM and Randomization | | $X^{\dagger}$ | | | | | | | | | | |

| Study Visit Number | 000 | V01 | V02 | V03 | V04 | V05 | 90Λ | V07 | 80A | V09 | V10 | V11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D23 | D25 | D29 | D36 | D43 |
| Study Day post second study vaccination | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |
| | Study Pr | ocedure/Eval | uation | • | | | | • | | | | |
| Venous Blood Collection for Clinical Safety Laboratory<br>Evaluations~ | | X <sup>†#</sup> | | | X | | $X^{\dagger}$ | | | X | | |
| Venous Blood Collection for Serological Assays | | $X^{\dagger}$ | | | | | $X^{\dagger\Psi}$ | | | | | X |
| Venous Blood Collection for Cellular Immunology<br>Assays | | Χ <sup>†</sup> | X | X | X | X | $X^{\dagger}$ | X | X | X | X | |
| Venous Blood Collection for Future Research | | $X^{\dagger}$ | X | X | X | X | $X^{\dagger}$ | X | X | X | X | X |
| Pre-Administration Reactogenicity Assessments | | $X^{\dagger}$ | | | | | $X^{\dagger}$ | | | | | |
| Study Vaccination | | X | | | | | X | | | | | |
| 20-minute Evaluation After Study Vaccination | | X | | | | | X | | | | | |
| Examine Study Vaccination Site | | X | X | X | X | | X | X | X | X | | |
| Post-Administration Reactogenicity Assessments | | X | | | | | X | | | | | |
| Distribute Memory Aid and Study-Related Materials | | X | | | | | X | | | | | |
| Review Memory Aid | | | X | X | X | | | X | X | X | | |
| AE/SAE Assessment | | X <sup>&amp;</sup> | X& | X& | X& | X | X&4 | X&4 | X&4 | X&4 | $X^4$ | $X^4$ |
| ∞ Prior to study procedures. | | | | | | | | | | | | |

| Study Visit Number | V00 | V01 | V02 | V03 | V04 | V05 | 901 | V07 | 801 | 601 | V10 | V11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D23 | D25 | D29 | D36 | D43 |
| Study Day post second study vaccination | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |

- Review/confirm information or activity in subjects previously consented and screened.
- † Prior to study vaccination.
- \* Not required if done at the optional screening visit.
- Review results of ESR or clinical safety laboratory evaluations.
- @ Complete medical history will be obtained by interview of subjects at the screening visit (optional) or on Day 1 prior to the first study vaccination, and interim medical history will be obtained by interview of subjects at follow-up visits after the first study vaccination.
- Receipt of any non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.
- \$ Vital signs assessed on Day 1 prior to the first study vaccination will be considered as baseline.
- % Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.
- Vital signs are not required for subjects who are discontinued from receipt of the second study vaccination and being followed for safety.
- At the screening visit (optional) or on Day 1 prior to the first study vaccination, a physical examination will be performed on all subjects to include the following organs and organ systems: skin, head and neck, lungs, heart, liver, spleen, extremities, lymph nodes, and nervous system, and as an assessment for signs suggestive of PIMMCs.
- Targeted physical examination if indicated based on review of interim medical history.
- Performed locally by the site at the screening visit (optional) or within 24 hours prior to each study vaccination for all women of childbearing potential. Results must be negative and known prior to randomization on Day 1 and administration of each study vaccination.
- Performed locally by the site at the screening visit (optional) or on Day 1 prior to the first study vaccination. The ESR value must be confirmed as less than 30 mm per hour prior to randomization on Day 1 and administration of the first study vaccination.
- ~ Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.
- # Clinical safety laboratory evaluations assessed on Day 1 prior to the first study vaccination will be considered as baseline.

| Study Visit Number | 000 | V01 | V02 | V03 | V04 | V05 | 901 | V07 | 801 | 601 | V10 | V11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D23 | D25 | D29 | D36 | D43 |
| Study Day post second study vaccination | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |

- Ψ Subjects who receive only one dose of study vaccine will be encouraged to remain in this trial for follow-up safety assessments (may be conducted by phone call rather than in person) continuing through approximately 12 months after their last study vaccination. These subjects will also be encouraged to provide a venous blood sample for serological assays approximately 21 and 180 days after their last study vaccination.
- & Inclusive of reactogenicity assessments performed on the day of each study vaccination through 7 days after each study vaccination.
- <sup>4</sup> AEs limited to SAEs and MAAEs, including NOCMCs and PIMMCs, for subjects who are discontinued from receipt of the second study vaccination and being followed for safety.

Table 3: Schedule of Study Procedures – Follow-Up Period for Study Groups 1 and 4 (Including early termination and unscheduled visits)

| Study Visit Number | V12** | V13 | V14** | V15 | V16** | Early Termination<br>(if needed) | Unscheduled<br>(if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | D82 | D112 | D142 | D202 | D387 | | |
| Study Day post second study vaccination | D61±7d | D91±14d | D121±14d | D181±14d | D366±14d | | |
| Study Pr | ocedur | ·e/Eval | uation | | | | |
| Medical History <sup>@</sup> | | X | | X | | X | X (if indicated) |
| Concomitant Medications <sup>c</sup> | X | X | X | X | | X (if prior to 21 days<br>after last study<br>vaccination and<br>receipt of any non-<br>study influenza<br>vaccines if within 180<br>days after last study<br>vaccination) | X (if prior to 21 days<br>after last study<br>vaccination and receipt<br>of any non-study<br>influenza vaccines if<br>within 180 days after<br>last study vaccination) |
| Vital Signs (Oral Temperature%, Pulse and BP) | | | | | | X (may be obtained if indicated) | X (may be obtained if indicated) |
| Physical Examination | | {X} | | {X} | | {X} | {X} |
| Venous Blood Collection for Clinical Safety Laboratory Evaluations~ | | | | | | X (if within 7 days<br>after last study<br>vaccination) | X (if indicated) |

| Study Visit Number | V12** | V13 | V14** | V15 | V16** | Early Termination (if needed) | Unscheduled (if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | D82 | D112 | D142 | D202 | D387 | | |
| Study Day post second study vaccination | D61±7d | D91±14d | D121±14d | D181±14d | D366±14d | | |
| Study Pr | ocedui | e/Eval | uation | | | | |
| Venous Blood Collection for Serological Assays | | | | $X^{\Psi}$ | | X (if within 21 days<br>after last study<br>vaccination) | X (if within 21 days<br>after last study<br>vaccination) |
| Venous Blood Collection for Cellular Immunology Assays | | X | | X | | X (if within 21 days<br>after last study<br>vaccination) | X (if within 21 days<br>after last study<br>vaccination) |
| Venous Blood Collection for Future Research | | X | | X | | X (if within 21 days<br>after last study<br>vaccination) | X (if within 21 days<br>after last study<br>vaccination) |
| Examine Study Vaccination Site | | | | | | X (if within 7 days<br>after last study<br>vaccination) | X (if within 7 days<br>after last study<br>vaccination) |
| Post-Administration Reactogenicity Assessments | | | | | | X (if within 7 days<br>after last study<br>vaccination) | X (if within 7 days<br>after last study<br>vaccination) |
| Review Memory Aid | | | | | | X (if within 7 days<br>after last study<br>vaccination) | X (if within 7 days<br>after last study<br>vaccination) |

| Study Visit Number | V12** | V13 | V14** | V15 | V16** | Early Termination<br>(if needed) | Unscheduled<br>(if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | D82 | D112 | D142 | D202 | D387 | | |
| Study Day post second study vaccination | D61±7d | D91±14d | D121±14d | D181±14d | D366±14d | | |
| Study Pr | ocedur | e/Eval | uation | | | | |
| AE/SAE Assessment! | X | X | X | X | X | X (if after 21 days<br>after last study<br>vaccination) | X (if after 21 days after last study vaccination) |

<sup>\*\*</sup> Phone call assessment.

- @ Complete medical history will be obtained by interview of subjects at the screening visit (optional) or on Day 1 prior to the first study vaccination, and interim medical history will be obtained by interview of subjects at follow-up visits after the first study vaccination.
- Receipt of any non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.
- % Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.
- {} Targeted physical examination if indicated based on review of interim medical history.
- ~ Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.
- Ψ Subjects who receive only one dose of study vaccine will be encouraged to remain in this trial for follow-up safety assessments (may be conducted by phone call rather than in person) continuing through approximately 12 months after their last study vaccination. These subjects will also be encouraged to provide a venous blood sample for serological assays approximately 21 and 180 days after their last study vaccination.
- ! AEs limited to SAEs and MAAEs, including NOCMCs and PIMMCs, that have occurred since the previous clinic visit or phone call.

Table 4: Schedule of Study Procedures – Vaccination Period for Study Groups 2, 3, 5, and 6

| Study Visit Number | 000 | V01 | V02 | V03 | V04 | V05 | 90Λ | V07** | V08 | 60Λ | V10 | V111 | V12 | V13 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D61±7d | D121-7/+14d | D122 | D124 | D128 | D135 | D142 |
| Study Day post second study vaccination | | | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |
| | | Study Pro | ocedur | e/Eval | uation | | | | | | | | | |
| Informed Consent∞ | X | X <sup>†</sup> ¬ | | | | | | | | | | | | |
| Demographic Information | X | $X^{\dagger^*}$ | | | | | | | | | | | | |
| Eligibility Criteria | X | $X^{\dagger \lnot l}$ | | | | | | | $X^{\dagger 1}$ | | | | | |
| Medical History@ | X | Χ <sup>†¬</sup> | X | X | X | X | X | $\mathbf{X}^{\varsigma}$ | Χ <sup>†</sup> | X | X | X | X | X |
| Concomitant Medications <sup>c</sup> | X | X <sup>†</sup> ¬ | X | X | X | X | X | X | $X^{\dagger}$ | X | X | X | X | X |
| <sup>\$</sup> Vital Signs (Oral Temperature <sup>%</sup> , Pulse and BP) | X | X <sup>†\$</sup> | | | | | | | $X^{\dagger 2}$ | | | | | |
| Height and Weight | X | $X^{\dagger *}$ | | | | | | | | | | | | |
| Physical Examination | $X^3$ | $X^{\dagger 3*\{\}}$ | {X} | {X} | {X} | {X} | {X} | | $\{X\}^{\dagger}$ | {X} | {X} | {X} | {X} | {X} |
| Urine or Serum Pregnancy Test | X^ | $X^{\dagger^{\wedge}}$ | | | | | | | $X^{\dagger^{\wedge}}$ | | | | | |
| Venous Blood Collection for ESR | $X^{\neq}$ | $X^{\neq *}$ | | | | | | | | | | | | |
| Enrollment in AdvantageEDC <sup>SM</sup> and Randomization | | Χ <sup>†</sup> | | | | | | | | | | | | |

| Study Visit Number | 000 | V01 | V02 | V03 | V04 | V05 | 90Λ | **TOV | 80A | V09 | V10 | V111 | V12 | V13 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D61±7d | D121-7/+14d | D122 | D124 | D128 | D135 | D142 |
| Study Day post second study vaccination | | | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |
| | | Study Pro | ocedur | e/Eval | uation | | | | | | | | | |
| Venous Blood Collection for Clinical Safety<br>Laboratory Evaluations~ | | $X^{\dagger^{\#}}$ | | | X | | | | $X^{\dagger}$ | | | X | | |
| Venous Blood Collection for Serological<br>Assays | | $X^{\dagger}$ | | | | | X | | $X^{\dagger\Psi}$ | | | | | X |
| Venous Blood Collection for Cellular<br>Immunology Assays | | $X^{\dagger}$ | X | X | X | X | | | $X^{\dagger}$ | X | X | X | X | |
| Venous Blood Collection for Future<br>Research | | Χ <sup>†</sup> | X | X | X | X | X | | $X^{\dagger}$ | X | X | X | X | X |
| Pre-Administration Reactogenicity Assessments | | $X^{\dagger}$ | | | | | | | $X^{\dagger}$ | | | | | |
| Study Vaccination | | X | | | | | | | X | | | | | |
| 20-minute Evaluation After Study<br>Vaccination | | X | | | | | | | X | | | | | |
| Examine Study Vaccination Site | | X | X | X | X | | | | X | X | X | X | | |
| Post-Administration Reactogenicity Assessments | | X | | | | | | | X | | | | | |

| Study Visit Number | 000 | V01 | V02 | V03 | V04 | V05 | 90Λ | V07** | V08 | V09 | V10 | V11 | V12 | V13 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D61±7d | D121-7/+14d | D122 | D124 | D128 | D135 | D142 |
| Study Day post second study vaccination | | | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |
| | | Study Pro | ocedur | e/Eval | uation | | | | | | | | | |
| Distribute Memory Aid and Study-Related<br>Materials | | X | | | | | | | X | | | | | |
| Review Memory Aid | | | X | X | X | | | | | X | X | X | | |
| AE/SAE Assessment | | X <sup>&amp;</sup> | X& | X& | X <sup>&amp;</sup> | X | X | X! | X& | X&4 | X&4 | X <sup>&amp;4</sup> | $X^4$ | $X^4$ |

- \*\* Phone call assessment.
- $\infty$  Prior to study procedures.
- Review/confirm information or activity in subjects previously consented and screened.
- † Prior to study vaccination.
- \* Not required if done at the optional screening visit.
- <sup>1</sup> Review results of ESR or clinical safety laboratory evaluations.
- @ Complete medical history will be obtained by interview of subjects at the screening visit (optional) or on Day 1 prior to the first study vaccination, and interim medical history will be obtained by interview of subjects at follow-up visits after the first study vaccination.
- Receipt of any non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination and reported in the eCRF.
- \$ Vital signs assessed on Day 1 prior to the first study vaccination will be considered as baseline.
- % Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.
- Vital signs are not required for subjects who are discontinued from receipt of the second study vaccination and being followed for safety.

| Study Visit Number | 000 | V01 | V02 | V03 | V04 | V05 | 90Λ | V07** | V08 | 60A | V10 | V11 | V12 | V13 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d | D61±7d | D121-7/+14d | D122 | D124 | D128 | D135 | D142 |
| Study Day post second study vaccination | | | | | | | | | Dose 2<br>D1 | D2+1d | D4+1d | D8-1/+2d | D15±1d | D22+7d |

- At the screening visit (optional) or on Day 1 prior to the first study vaccination, a physical examination will be performed on all subjects to include the following organs and organ systems: skin, head and neck, lungs, heart, liver, spleen, extremities, lymph nodes, and nervous system, and as an assessment for signs suggestive of PIMMCs.
- {} Targeted physical examination if indicated based on review of interim medical history.
- ^ Performed locally by the site at the screening visit (optional) or within 24 hours prior to each study vaccination for all women of childbearing potential. Results must be negative and known prior to randomization on Day 1 and administration of each study vaccination.
- Performed locally by the site at the screening visit (optional) or on Day 1 prior to the first study vaccination. The ESR value must be confirmed as less than 30 mm per hour prior to randomization on Day 1 and administration of the first study vaccination.
- ~ Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.
- # Clinical safety laboratory evaluations assessed on Day 1 prior to the first study vaccination will be considered as baseline.
- Ψ Subjects who receive only one dose of study vaccine will be encouraged to remain in this trial for follow-up safety assessments (may be conducted by phone call rather than in person) continuing through approximately 12 months after their last study vaccination. These subjects will also be encouraged to provide a venous blood sample for serological assays approximately 21 and 180 days after their last study vaccination.
- & Inclusive of reactogenicity assessments performed on the day of each study vaccination through 7 days after each study vaccination.
- ! AEs limited to SAEs and MAAEs, including NOCMCs and PIMMCs, that have occurred since the previous clinic visit or phone call.
- <sup>4</sup> AEs limited to SAEs and MAAEs, including NOCMCs and PIMMCs, for subjects who are discontinued from receipt of the second study vaccination and being followed for safety.

Table 5: Schedule of Study Procedures – Follow-Up Period for Study Groups 2, 3, 5, and 6 (Including early termination and unscheduled visits)

| Study Visit Number | V14** | V15 | V16** | V17 | V18** | Early Termination (if needed) | Unscheduled<br>(if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | D181 | D2111 | D241 | D301 | D486 | | |
| Study Day post second study vaccination | D61±7d | D91±14d | D121±14d | D181±14d | D366±14d | | |
| Study I | Proced | ure/Ev | aluati | on | | | |
| Medical History <sup>@</sup> | | X | | X | | X | X (if indicated) |
| Concomitant Medications <sup>c</sup> | X | X | X | X | | X (if prior to 21 days<br>after last study<br>vaccination and receipt of<br>any non-study influenza<br>vaccines if within 180<br>days after last study<br>vaccination) | X (if prior to 21 days<br>after last study<br>vaccination and<br>receipt of any non-<br>study influenza<br>vaccines if within 180<br>days after last study<br>vaccination) |
| Vital Signs (Oral Temperature%, Pulse and BP) | | | | | | X (may be obtained if indicated) | X (may be obtained if indicated) |
| Physical Examination | | {X} | | {X} | | {X} | {X} |
| Venous Blood Collection for Clinical Safety Laboratory Evaluations~ | | | | | | X (if within 7 days after last study vaccination) | X (if indicated) |
| Venous Blood Collection for Serological Assays | | | | XΨ | | X (if within 21 days after last study vaccination) | X (if within 21 days<br>after last study<br>vaccination) |

| Study Visit Number | V14** | V15 | V16** | V17 | V18** | Early Termination<br>(if needed) | Unscheduled<br>(if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | D181 | D211 | D241 | D301 | D486 | | |
| Study Day post second study vaccination | D61±7d | D91±14d | D121±14d | D181±14d | D366±14d | | |
| Study P | roced | ure/Ev | aluatio | on | | | |
| Venous Blood Collection for Cellular Immunology Assays | | X | | X | | X (if within 21 days after last study vaccination) | X (if within 21 days<br>after last study<br>vaccination) |
| Venous Blood Collection for Future Research | | X | | X | | X (if within 21 days after last study vaccination) | X (if within 21 days<br>after last study<br>vaccination) |
| Examine Study Vaccination Site | | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days<br>after last study<br>vaccination) |
| Post-Administration Reactogenicity Assessments | | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days<br>after last study<br>vaccination) |
| Review Memory Aid | | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days<br>after last study<br>vaccination) |
| AE/SAE Assessment! | X | X | X | X | X | X (if after 21 days after last study vaccination) | X (if after 21 days<br>after last study<br>vaccination) |
| ** Phone call assessment. | | | | | | last study vaccination) | |

| Study Visit Number | V14** | V15 | V16** | V17 | V18** | Early Termination<br>(if needed) | Unscheduled<br>(if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post first study vaccination | DI8I | D2111 | D241 | D301 | D486 | | |
| Study Day post second study vaccination | D61±7d | D91±14d | D121±14d | D181±14d | D366±14d | | |

- @ Complete medical history will be obtained by interview of subjects at the screening visit (optional) or on Day 1 prior to the first study vaccination, and interim medical history will be obtained by interview of subjects at follow-up visits after the first study vaccination.
- Receipt of any non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.
- % Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.
- {} Targeted physical examination if indicated based on review of interim medical history.
- ~ Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.
- Ψ Subjects who receive only one dose of study vaccine will be encouraged to remain in this trial for follow-up safety assessments (may be conducted by phone call rather than in person) continuing through approximately 12 months after their last study vaccination. These subjects will also be encouraged to provide a venous blood sample for serological assays approximately 21 and 180 days after their last study vaccination.
- ! AEs limited to SAEs and MAAEs, including NOCMCs and PIMMCs, that have occurred since the previous clinic visit or phone call.

### 9.7.1 Sample Size

**Table 6:** Power (%) to Detect Safety Events

| <b>Event Frequency</b> | N=30 | N=180 |
|------------------------|------|-------|
| ≥10%<br>Very Common | 95 | >99 |
| ≥1%<br>Common | 26 | 83 |
| ≥0.1%<br>Uncommon | 2 | 16 |
| ≥0.01%<br>Rare | <1 | 1 |

**Table 7: Precisions of Binomial Confidence Intervals** 

| N | 95% CI |
|-----|--------|
| 30 | 31-69 |
| 180 | 42-58 |

**Table 8:** Minimum Detectable Difference in Proportion Responders

| N per Group | <b>Proportion Responders</b> | 80% Power | |
|---|---|---|---|
| | in Comparator Group A | Minimal Detectable<br>Difference | Proportion Responders in<br>Comparator Group B |
| N=27 | 0.10 | 0.32 | 0.42 |
| | 0.20 | 0.35 | 0.55 |
| | 0.30 | 0.38 | 0.68 |
| | 0.40 | 0.37 | 0.77 |
| | 0.50 | 0.34 | 0.84 |

### 10.2 Protocol Deviations

Table 9: Distribution of Protocol Deviations by Category, Type, and Study Group

| Category | Deviation Type | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 1<br>013<br>-AS03/<br>017<br>-AS03<br>-D22)<br>=X) | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 2<br>013<br>AS03/<br>017<br>-AS03<br>D121)<br>=X) | Grou<br>201<br>3.75+A<br>2017<br>(D1-I<br>(N= | 13<br>AS03/<br>115<br>D121) | 3.75-<br>2<br>3.75-<br>(D1 | oup 4<br>017<br>+AS03/<br>017<br>+AS03<br>-D22) | 3.75-<br>2:<br>3.75-<br>(D1- | oup 5<br>017<br>-AS03/<br>017<br>+AS03<br>-D121) | Grou<br>201<br>3.75+A<br>2017<br>(D1-D<br>(N=2 | 7<br>AS03/<br>15<br>0121) | | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Eligibility/<br>enrollment | Any type | | | | | | | | | | | | | | |
| | Did not meet inclusion criterion | х | х | х | Х | Х | х | х | х | х | X | х | Х | х | х |
| | Met exclusion criterion | | | | | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | | | |
| | Missed treatment administration | | | | | | | | | | | | | | |
| | Delayed treatment administration | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |

| Category | Deviation Type | 20<br>3.75+<br>20<br>3.75+<br>(D1 | oup 1<br>013<br>-AS03/<br>017<br>-AS03<br>-D22)<br>=X)<br># of | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 2<br>013<br>-AS03/<br>017<br>-AS03<br>D121)<br>=X)<br># of | Grou<br>201<br>3.75+4<br>2017<br>(D1-I<br>(N= | 13<br>AS03/<br>15<br>D121) | 3.75-<br>2<br>3.75-<br>(D1 | oup 4<br>017<br>+AS03/<br>017<br>+AS03<br>-D22)<br>=X)<br># of | 3.75+<br>20<br>3.75-<br>(D1- | oup 5<br>017<br>-AS03/<br>017<br>+AS03<br>-D121)<br>=X)<br># of | Grou<br>201<br>3.75+A<br>2017<br>(D1-D<br>(N=) | 7<br>.S03/<br>15<br>121) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Subj. | Dev. | Subj. | Dev. | Subj. | Dev. | Subj. | Dev. | Subj. | Dev. | Subj. | Dev. | Subj. | Dev. |
| Follow-up visit schedule | Any type | | | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Protocol<br>procedure/<br>assessment | Any type | | | | | | | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | | | | | | | |
| | Blood not collected | | | | | | | | | | | | | | |
| | Urine not collected | | | | | | | | | | | | | | |
| | Other specimen not collected | | | | | | | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | | | | | | | |
| | Specimen result not obtained | | | | | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | | | |

| Category | Deviation Type | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 1<br>013<br>-AS03/<br>017<br>-AS03<br>-D22)<br>=X) | 20<br>3.75+<br>20<br>3.75+<br>(D1-1 | up 2<br>113<br>AS03/<br>117<br>-AS03<br>D121)<br>=X) | Grou<br>201<br>3.75+4<br>2017<br>(D1-I<br>(N= | 13<br>AS03/<br>115<br>D121) | 3.75+<br>20<br>3.75-<br>(D1 | oup 4<br>017<br>-AS03/<br>017<br>+AS03<br>-D22)<br>=X) | 3.75-<br>2<br>3.75-<br>(D1- | oup 5<br>017<br>+AS03/<br>017<br>+AS03<br>-D121)<br>(=X) | Grou<br>201<br>3.75+A<br>2017<br>(D1-D<br>(N=) | 7<br>\$803/<br>15<br>(121) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| | Study product temperature excursion | | | | | | | | | | | | | | |
| | Specimen temperature excursion | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Treatment administration | Any type | | | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Blinding policy/<br>procedure | Any type | | | | | | | | | | | | | | |
| | Treatment unblinded | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |

N = Number of subjects enrolled.

Implementation Note: Shell has placeholders for all types of deviations possible. The final table will be limited to deviations actually reported in the study.

### 12.2.2 Displays of Adverse Events

 Table 10:
 Solicited Adverse Event Grading Scale – Local

| | Local (Injection Site) Reactogenicity Grading | | |
|---|---|---|---|
| Local (Injection Site)<br>Reaction | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Pain – experienced<br>without touching the<br>injection site<br>(spontaneous discomfort) | Subject is aware of pain,<br>but it does not interfere<br>with daily activity, <b>and</b> no<br>pain medication is taken | Subject is aware of pain;<br>there is interference with<br>daily activity, <b>or</b> it<br>requires repeated use of a<br>non-narcotic pain reliever<br>for >24 hours | Subject is aware of pain, and it prevents daily activity or requires any use of a narcotic pain reliever |
| Tenderness – hurts only<br>when injection site is<br>touched, or the arm is<br>moved | The area immediately surrounding the injection site hurts only when touched or with arm motion, and it does not interfere with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, and it interferes with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, <b>and</b> it prevents daily activity |
| Pruritus (Itching) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Ecchymosis (Bruising)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Erythema (Redness)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Induration (Hardness)/Swelling* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| | Local (Injection Site) Re | actogenicity Measurements | |
| Local (Injection Site)<br>Reaction | Small (Grade 1) | Medium (Grade 2) | Large (Grade 3) |
| Ecchymosis (Bruising)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Erythema (Redness)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Induration (Hardness)/Swelling* | <20 mm | 20 mm – 50 mm | >50 mm |

**Table 11:** Solicited Adverse Event Grading Scale - Systemic

| | Subjective Systemic Reactogenicity Grading | | |
|---|---|---|---|
| Systemic (Subjective) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Feverishness (Chills/Shivering/Sweating) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Fatigue (Tiredness) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Malaise (General Unwell<br>Feeling) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Myalgia (Body Aches/Muscular<br>Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Arthralgia (Joint Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Headache | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Nausea | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| | Quantitative Systemic | Reactogenicity Grading | |
| Systemic (Quantitative) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Fever# - oral† | 38.0°C – 38.4°C | 38.5°C – 38.9°C | >38.9°C |
| | 100.4°F – 101.1°F | 101.2°F – 102.0°F | >102.0°F |

<sup>\*</sup> Not at injection site.

<sup>&</sup>lt;sup>#</sup> Oral temperature assessed on Day 1 prior to the first study vaccination will be considered as baseline. A fever can be considered not related to the study product if an alternative etiology can be documented.

**Table 12:** Vital Signs Adverse Event Grading Scale

| Physiologic Parameter | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Bradycardia - beats per minute | 45 - 46 | 40 – 44 | <40 |
| Tachycardia - beats per minute | 101 – 130 | 131 – 155 | >155 |
| Hypotension (systolic) mmHg | 80 - 84 | 75 – 79 | <75 |
| Hypotension (diastolic) mmHg | 50 – 54 | 45 – 49 | <45 |
| Hypertension (systolic) mmHg | 151 – 155 | 156 – 160 | >160 |
| Hypertension (diastolic) mmHg | 96 – 100 | 101 – 105 | >105 |

<sup>&</sup>lt;sup>#</sup> Pulse and blood pressure assessed on Day 1 prior to the first study vaccination will be considered as baseline.

### 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

**Table 13:** Laboratory Adverse Event Grading Scale

| Hematology | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| WBC 10 <sup>3</sup> /μL (Decrease) | 2.5 – 3.9 | 1.5 – 2.4 | <1.5 |
| WBC 10 <sup>3</sup> /μL (Increase) | 10.6 – 15.0 | 15.1 – 20.0 | >20.0 |
| Hgb g/dL (Decrease) (Female) | 10.1 – 11.4 | 8.5 – 10 | <8.5 |
| Hgb g/dL (Decrease) (Male) | 11.0 – 12.4 | 9.5 – 10.9 | <9.5 |
| Platelets 10 <sup>3</sup> /μL (Decrease) | 125 – 139 | 100 – 124 | <100 |
| Platelets 10 <sup>3</sup> /μL (Increase) | 416 – 550 | 551-750 | >750 |
| Chemistry | Mild | Moderate | Severe |
| | (Grade 1) | (Grade 2) | (Grade 3) |
| ALT IU/L (Increase) (Female) | 44 - 100 | 101 – 200 | >200 |
| ALT IU/L (Increase) (Male) | 61 - 138 | 139 – 275 | >275 |
| Total Bilirubin mg/dL (Increase) – when accompanied by any increase in ALT | 1.30 – 1.59 | 1.60 – 1.80 | >1.80 |
| Total Bilirubin mg/dL (Increase) – when ALT is normal | 1.30 – 1.89 | 1.90 – 2.40 | >2.40 |
| Creatinine mg/dL (Increase) (Female) | 1.1 – 1.7 | 1.8 - 2.0 | >2.0 |
| Creatinine mg/dL (Increase) (Male) | 1.4 - 1.7 | 1.8 - 2.0 | >2.0 |

### 14.1 Description of Study Subjects

#### 14.1.1 Disposition of Subjects

**Table 14:** Ineligibility Summary of Screen Failures

| Category | Criterion | n <sup>a</sup> | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | x | X |
| Inclusion | Any inclusion criterion | x | X |
| | [inclusion criterion 1] | x | X |
| | [inclusion criterion 2] | x | X |
| | [inclusion criterion 3] | x | X |
| Exclusion | Any exclusion criterion | х | X |
| | [exclusion criterion 1] | X | X |
| | [exclusion criterion 2] | X | X |
| | [exclusion criterion 3] | x | X |
| Eligible but Not Enrolled | Any reason | X | X |
| | [reason 1] | x | X |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup> Denominator for percentages is the total number of screen failures.
**Table 15:** Analysis Populations by Study Group – All Enrolled Subjects

[Implementation Note: Only include reasons actually reported, omit lines for any reasons that were not observed in the trial.]

| Analysis Populations | Reason Subjects Excluded | 20<br>3.75+<br>20173.7<br>(D1 | oup 1<br>013<br>AS03/<br>75+AS03<br>-D22)<br>=X) | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 2<br>013<br>AS03/<br>017<br>-AS03<br>D121)<br>=X) | 20<br>3.75+<br>201<br>(D1- | oup 3<br>013<br>AS03/<br>7 15<br>D121)<br>=X) | 3.75<br>3.75<br>(D | roup 4<br>2017<br>+AS03/<br>2017<br>5+AS03<br>1-D22)<br>N=X) | 20<br>3.75+<br>20<br>3.75-<br>(D1- | oup 5<br>017<br>-AS03/<br>017<br>+AS03<br>-D121)<br>=X) | 20<br>3.75+<br>201<br>(D1- | up 6<br>17<br>AS03/<br>7 15<br>D121)<br>=X) | Subj | ll<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Safety Population | Any Reason | X | xx | X | XX | X | XX | x | xx | X | XX | X | XX | X | XX |
| | Study Vaccination 1 Not Received | X | xx | X | XX | X | XX | X | XX | X | XX | x | XX | X | xx |
| Modified Intent-to-Treat | Any Reason | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Study Vaccination 1 Not Received | Х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | Х | XX |
| | No Baseline Results Available | Х | XX | Х | XX | х | XX | X | XX | х | XX | х | XX | Х | XX |
| | No Post-Vaccination Results<br>Available | Х | XX | Х | xx | х | XX | X | XX | Х | XX | х | xx | х | XX |
| Per Protocol, Day 22 post<br>Vac 1 | Any Reason | Х | XX | Х | xx | х | xx | X | XX | х | XX | х | XX | х | xx |
| | Study Vaccination 1 Not Received | Х | XX | х | XX | х | XX | X | XX | х | XX | х | XX | Х | XX |
| | No Baseline Results Available | Х | XX | х | XX | х | XX | X | XX | х | XX | х | XX | Х | XX |
| | No Day 22 post Vac 1 Result<br>Reported by Lab | х | XX | Х | xx | х | xx | X | XX | х | XX | х | XX | х | xx |
| | Lost to Follow-up Before Day 22 post Vac 1 | X | XX | Х | XX | Х | xx | Х | XX | X | XX | X | xx | х | xx |
| | Receipt of Non-Study Vaccination | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Receipt of Immunosuppressive medication | Х | XX | Х | xx | Х | xx | X | XX | X | XX | X | XX | х | xx |

| Analysis Populations | Reason Subjects Excluded | 20<br>3.75+<br>20173.7<br>(D1 | oup 1<br>013<br>AS03/<br>75+AS03<br>-D22)<br>=X) | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 2<br>013<br>AS03/<br>017<br>-AS03<br>D121)<br>=X) | 20<br>3.75+<br>201<br>(D1- | oup 3<br>013<br>AS03/<br>7 15<br>D121)<br>=X) | 3.75<br>3.75<br>(D | roup 4<br>2017<br>i+AS03/<br>2017<br>5+AS03<br>1-D22)<br>N=X) | 3.75+<br>20<br>3.75-<br>(D1- | Dup 5<br>D17<br>-AS03/<br>D17<br>+AS03<br>-D121) | 20<br>3.75+<br>201<br>(D1- | oup 6<br>017<br>AS03/<br>7 15<br>D121)<br>=X) | A<br>Subj<br>(N= | jects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Day 22 post Vac 1 Visit Out of<br>Window | х | XX | Х | xx | х | xx | Х | XX | X | xx | Х | XX | х | xx |
| Per Protocol, Day 121 post<br>Vac 1 | Any Reason | NA | NA | Х | xx | х | xx | NA | NA | х | xx | х | xx | х | xx |
| | Study Vaccination 1 Not Received | NA | NA | Х | XX | х | XX | NA | NA | х | xx | х | xx | X | xx |
| | Study Vaccination 2 Not Received | NA | NA | X | XX | х | XX | NA | NA | х | xx | х | xx | Х | xx |
| | Study Vaccination 2 Out of Window | NA | NA | Х | xx | х | xx | NA | NA | X | xx | Х | XX | х | xx |
| | No Baseline Results Available | NA | NA | Х | XX | х | XX | NA | NA | Х | XX | Х | XX | X | XX |
| | No Day 121 post Vac 1 Result<br>Reported by Lab | NA | NA | х | xx | х | xx | NA | NA | х | xx | х | xx | Х | XX |
| | Lost to Follow-up Before Day 121 post Vac 1 | NA | NA | х | xx | х | xx | NA | NA | Х | xx | Х | xx | х | xx |
| | Receipt of Non-Study Vaccination | NA | NA | Х | XX | х | XX | NA | NA | Х | XX | Х | XX | X | XX |
| | Receipt of Immunosuppressive medication | NA | NA | х | xx | х | xx | NA | NA | Х | xx | Х | XX | х | XX |
| | Day 121 post Vac 1 Visit Out of<br>Window | NA | NA | х | xx | х | XX | NA | NA | Х | xx | Х | xx | х | xx |
| Per Protocol, Day 22 post<br>Vac 2 | Any Reason | х | xx | х | xx | X | XX | х | XX | X | xx | X | XX | х | xx |
| | Study Vaccination 1 Not Received | Х | XX | X | XX | х | XX | X | XX | х | XX | х | XX | Х | XX |
| | Study Vaccination 2 Not Received | Х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |

| Analysis Populations | Reason Subjects Excluded | 20<br>3.75+<br>20173.7<br>(D1 | oup 1<br>013<br>-AS03/<br>75+AS03<br>-D22)<br>=X) | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 2<br>013<br>-AS03/<br>017<br>-AS03<br>D121)<br>=X) | 20<br>3.75+<br>201<br>(D1- | oup 3<br>013<br>AS03/<br>7 15<br>D121)<br>=X) | 3.75<br>3.75<br>(D | roup 4<br>2017<br>5+AS03/<br>2017<br>5+AS03<br>1-D22)<br>N=X) | 20<br>3.75+<br>20<br>3.75-<br>(D1- | oup 5<br>017<br>+AS03/<br>017<br>+AS03<br>-D121) | 20<br>3.75+<br>201<br>(D1- | oup 6<br>017<br>AS03/<br>7 15<br>D121)<br>=X) | Sub | ill<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Study Vaccination 2 Out of Window | Х | XX | Х | XX | X | xx | х | XX | Х | xx | Х | XX | х | xx |
| | No Baseline Results Available | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX | X | xx |
| | No Day 22 post Vac 2 Result<br>Reported by Lab | Х | XX | Х | XX | х | XX | х | XX | х | xx | х | xx | х | xx |
| | Lost to Follow-up Before Day 22 post Vac 2 | Х | XX | Х | XX | х | xx | х | xx | Х | xx | х | XX | х | xx |
| | Receipt of Non-Study Vaccination | х | xx | Х | XX | х | XX | х | xx | х | XX | х | XX | X | xx |
| | Receipt of Immunosuppressive medication | х | XX | X | XX | х | xx | Х | xx | Х | xx | х | XX | X | xx |
| | Day 22 post Vac 2 Visit Out of Window | Х | XX | Х | XX | х | xx | х | xx | Х | xx | х | XX | х | xx |
| Per Protocol, Day 181 post<br>Vac 2 | Any Reason | х | XX | х | XX | Х | xx | х | XX | Х | xx | X | XX | х | xx |
| | Study Vaccination 1 Not Received | х | xx | Х | XX | х | XX | х | xx | х | XX | х | XX | X | xx |
| | Study Vaccination 2 Not Received | х | XX | X | XX | х | XX | Х | XX | х | XX | х | xx | X | XX |
| | Study Vaccination 2 Out of Window | х | xx | X | xx | Х | XX | х | xx | Х | xx | Х | xx | х | xx |
| | No Baseline Results Available | х | XX | х | xx | x | XX | Х | XX | х | xx | х | xx | X | xx |
| | No Day 181 post Vac 2 Result<br>Reported by Lab | х | xx | х | xx | Х | xx | x | XX | х | xx | Х | xx | х | xx |

| Analysis Populations | Reason Subjects Excluded | 3.75+<br>20173.7<br>(D1- | up 1<br>013<br>AS03/<br>25+AS03<br>-D22)<br>=X) | 20<br>3.75+<br>20<br>3.75+ | up 2<br>13<br>AS03/<br>17<br>-AS03<br>D121)<br>=X) | 20<br>3.75+<br>201<br>(D1- | oup 3<br>013<br>AS03/<br>7 15<br>D121)<br>=X) | 3.75<br>3.75<br>(D | roup 4<br>2017<br>4+AS03/<br>2017<br>5+AS03<br>1-D22)<br>N=X) | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 5<br>017<br>-AS03/<br>017<br>-AS03<br>D121)<br>=X) | 20<br>3.75+<br>201<br>(D1- | up 6<br>17<br>AS03/<br>7 15<br>D121)<br>=X) | A<br>Subj<br>(N= | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Lost to Follow-up Before Day 181 post Vac 2 | Х | XX | Х | xx | х | xx | X | XX | X | XX | Х | XX | X | xx |
| | Receipt of Non-Study Vaccination | X | XX | X | XX | х | XX | X | XX | X | XX | X | XX | X | xx |
| | Receipt of Immunosuppressive medication | X | XX | Х | xx | х | xx | X | XX | X | XX | X | xx | X | xx |
| | Day 181 post Vac 2 Visit Out of<br>Window | Х | XX | Х | XX | х | xx | Х | XX | X | XX | X | XX | Х | xx |

Table 16: Subject Disposition by Study Group, All Enrolled Subjects

| Subject<br>Disposition | 2013<br>2017 | Group 1<br>3.75+AS03/<br>3.75+AS03<br>D1-D22)<br>(N=X) | 2013 3.<br>2017 3.<br>(D1 | oup 2<br>75+AS03/<br>75+AS03<br>-D121) | 2013 3.<br>20<br>(D1 | roup 3<br>.75+AS03/<br>.17 15<br>D121)<br>N=X) | 2017 3.7<br>2017 3.7<br>(D1- | | Gro<br>2017 3.7<br>2017 3.7<br>(D1-1<br>(N= | 5+AS03/<br>/5+AS03<br>D121) | 2017 3.7<br>201<br>(D1- | rup 6<br>75+AS03/<br>7 15<br>D121)<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | X | | X | | X | | X | | X | | X | | X | |
| Enrolled/Randomized | X | 100 | X | 100 | X | 100 | X | 100 | X | 100 | X | 100 | X | 100 |
| Received Vaccination 1 | X | xx | X | XX | X | XX | X | XX | X | XX | X | xx | X | XX |
| Received Vaccination 2 | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Received All Scheduled Vaccinations <sup>a</sup> | x | XX | X | XX | X | XX | X | XX | Х | XX | X | XX | X | XX |
| Completed Blood Draw for<br>Primary Immunogenicity<br>Analysis <sup>b</sup> | х | XX | X | XX | X | XX | х | XX | х | XX | Х | XX | Х | XX |
| Included in Per Protocol<br>Immunogenicity Analysis<br>of Primary Immunogenicity<br>Outcomes <sup>b c</sup> | Х | xx | х | XX | х | XX | х | XX | х | XX | х | XX | х | xx |
| Completed Primary Follow-up <sup>a b c</sup> | X | XX | X | XX | х | xx | X | XX | Х | XX | X | XX | Х | xx |
| Completed Final Study<br>Visit <sup>b</sup> | X | xx | X | xx | х | xx | X | XX | Х | XX | X | XX | Х | xx |

N=Number of subjects enrolled.

<sup>&</sup>lt;sup>a</sup> Refer to Listing 2 for reasons subjects discontinued from study vaccinations or terminated early.

<sup>&</sup>lt;sup>b</sup> The final blood draw for Primary Immunogenicity Analysis occurs at 21 days post final vaccination (Day 43 for Groups 1 and 4; Day 142 for Groups 2, 3, 5 and 6).

<sup>&</sup>lt;sup>c</sup> Refer to Listing 5 for reasons subjects are excluded from the Per Protocol Population.

Table 17: Dates of First Study Vaccination by Site and Study Group

| Dates of Dosing | Group 1<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | | | [Site 1] | | | | |
| Total (Entire period of enrollment) | х | X | X | X | X | х | X |
| DDMMMYYYY-DDMMMYYYY | х | X | X | X | X | X | X |
| | | | [Site 2] | | | | |
| Total (Entire period of enrollment) | х | X | X | X | X | x | х |
| DDMMMYYYY-DDMMMYYYY | х | X | X | X | X | X | X |
| | | [Repe | at for all sites] | | | | |
| N= Number of subjects in the Safety Popula | ation. | | | | | | |

Table 18: Dates of Second Study Vaccination by Site and Study Group

# 14.1.2 Demographic Data by Study Group

 Table 19:
 Summary of Categorical Demographic and Baseline Characteristics by Site, All Enrolled Subjects

| Variable | Characteristic | | te 1]<br>=X) | | te 2]<br>=X) | | te 3]<br>=X) | | te 4]<br>=X) | | e 5]<br>=X) | | te 6]<br>=X) | A<br>Subj<br>(N= | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | х | XX | х | XX | X | XX | Х | XX | Х | xx | X | XX | х | xx |
| | Female | | | | | | | | | | | | | | |
| BMI | < 30 | | | | | | | | | | | | | | |
| | ≥ 30 | | | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | X | XX | X | XX | X | xx | X | XX | Х | XX | X | XX | х | xx |
| | Hispanic or Latino | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Race | American Indian or Alaska Native | Х | XX | X | XX | X | XX | X | XX | Х | xx | X | XX | Х | xx |
| | Asian | | | | | | | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | | | | | | | |
| | Black or African American | | | | | | | | | | | | | | |
| | White | | | | | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Prior Seasonal Influenza<br>Vaccination (Prior Seasons) | 2016-2017 Received | | | | | | | | | | | | | | |
| | 2016-2017 Not Received | | | | | | | | | | | | | | |

| Variable | Characteristic | _ | te 1]<br>=X) | | te 2]<br>=X) | _ | te 3]<br>=X) | _ | e 4]<br>=X) | [Site | - | _ | te 6]<br>=X) | A<br>Subj<br>(N= | ects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | 2016-2017 Unknown | | | | | | | | | | | | | | |
| | 2017-2018 Received | | | | | | | | | | | | | | |
| | 2017-2018 Not Received | | | | | | | | | | | | | | |
| | 2017-2018 Unknown | | | | | | | | | | | | | | |
| Seasonal Influenza Vaccination (Current Season) | 2018-2019 Received | | | | | | | | | | | | | | |
| | 2018-2019 Not Received | | | | | | | | | | | | | | |
| | 2018-2019 Unknown | | | | | | | | | | | | | | |
| Prior Receipt of H5 Influenza<br>Vaccine | No Prior H5 Influenza Vaccination(s) | | | | | | | | | | | | | | |
| | Received Prior H5 Influenza<br>Vaccination(s) | | | | | | | | | | | | | | |

**Table 20:** Summary of Continuous Demographic and Baseline Characteristics by Site, All Enrolled Subjects

| Variable | Statistic | [Site 1]<br>(N=X) | [Site 2]<br>(N=X) | [Site 3]<br>(N=X) | [Site 4]<br>(N=X) | [Site 5]<br>(N=X) | [Site 6]<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|
| Age | Mean | X.X | x.x | X.X | X.X | x.x | x.x | x.x |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | x.x | x.x |
| | Minimum | X | X | X | X | X | Х | X |
| | Maximum | X | X | X | X | X | Х | X |
| BMI | Mean | X.X | X.X | X.X | X.X | X.X | x.x | x.x |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | x.x | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | x.x | X.X |
| | Minimum | X | X | X | X | X | Х | X |
| | Maximum | х | х | Х | X | x | Х | X |

N= Number of subjects enrolled.

Table 21: Summary of Categorical Demographic and Baseline Characteristics by Study Group, All Enrolled Subjects

| Variable | Characteristic | 20<br>3.75+<br>(D1- | 13<br>AS03/ | 3.75-<br>2/<br>3.75-<br>(D1- | oup 2<br>013<br>+AS03/<br>017<br>+AS03<br>-D121) | 20<br>3.75+2<br>201'<br>(D1-I<br>(N= | 13<br>AS03/<br>7 15<br>D121) | 20<br>3.75+<br>20<br>3.75+<br>(D1- | up 4<br>17<br>AS03/<br>17<br>AS03<br>-D22)<br>=X) | 3.75+<br>20<br>3.75-<br>(D1- | oup 5<br>017<br>-AS03/<br>017<br>+AS03<br>-D121) | 3.75<br>20<br>(D1 | oup 6<br>017<br>+AS03/<br>17 15<br>-D121) | Sub | All<br>ojects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | X | XX | X | XX | X | xx | X | XX | X | XX | X | XX | X | XX |
| | Female | | | | | | | | | | | | | | |
| BMI | < 30 | | | | | | | | | | | | | | |
| | ≥ 30 | | | | | | | | | | | | | | |
| Age | 19-34 | x | XX | х | XX | Х | xx | х | xx | х | XX | х | XX | х | xx |
| | 35-50 | | | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | X | XX | Х | XX | X | xx | Х | xx | Х | XX | х | XX | х | XX |
| | Hispanic or Latino | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Race | American Indian or Alaska<br>Native | Х | xx | х | xx | х | xx | х | xx | х | xx | Х | XX | X | xx |
| | Asian | | | | | | | | | | | | | | |
| | Native Hawaiian or Other<br>Pacific Islander | | | | | | | | | | | | | | |
| | Black or African American | | | | | | | | | | | | | | |
| | White | | | | | | | | | | | | | | |

| Variable | Characteristic | 3.75+<br>20<br>3.75+<br>(D1- | 013<br>AS03/<br>017 | 3.75-<br>20<br>3.75-<br>(D1- | oup 2<br>013<br>+AS03/<br>017<br>+AS03<br>-D121) | 3.75+A<br>2017<br>(D1-I<br>(N= | 13<br>AS03/<br>7 15<br>D121) | 3.75+2<br>20<br>3.75+<br>20<br>3.75+<br>(D1-<br>(N= | 17<br>AS03/<br>17<br>AS03<br>D22) | 3.75+<br>20<br>3.75-<br>(D1- | oup 5<br>017<br>-AS03/<br>017<br>+AS03<br>-D121)<br>=X) | 3.75-<br>20<br>(D1 | oup 6<br>017<br>+AS03/<br>17 15<br>-D121) | Sub | All<br>ojects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Multi-Racial | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Prior<br>Seasonal<br>Influenza<br>Vaccination<br>(Prior<br>Seasons) | 2016-2017 Received | | | | | | | | | | | | | | |
| | 2016-2017 Not Received | | | | | | | | | | | | | | |
| | 2016-2017 Unknown | | | | | | | | | | | | | | |
| | 2017-2018 Received | | | | | | | | | | | | | | |
| | 2017-2018 Not Received | | | | | | | | | | | | | | |
| | 2017-2018 Unknown | | | | | | | | | | | | | | |
| Seasonal<br>Influenza<br>Vaccination<br>(Current<br>Season) | 2018-2019 Received | | | | | | | | | | | | | | |
| | 2018-2019 Not Received | | | | | | | | | | | | | | |
| | 2018-2019 Unknown | | | | | | | | | | | | | | |

| Variable | Characteristic | Groud<br>20<br>3.75+2<br>20<br>3.75+2<br>(D1-<br>(N= | 13<br>AS03/<br>17<br>AS03<br>D22) | 20<br>3.75+<br>20<br>3.75-<br>(D1- | oup 2<br>013<br>-AS03/<br>017<br>+AS03<br>-D121)<br>=X) | Grou<br>201<br>3.75+A<br>2017<br>(D1-I<br>(N= | 13<br>AS03/<br>7 15<br>D121) | Grood<br>20<br>3.75+2<br>20<br>3.75+<br>(D1-<br>(N= | 17<br>AS03/<br>17<br>AS03<br>D22) | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 5<br>017<br>AS03/<br>017<br>-AS03<br>D121)<br>=X) | 2<br>3.75-<br>20<br>(D1 | oup 6<br>017<br>+AS03/<br>17 15<br>-D121)<br>N=X) | Sub | All<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | <b>%</b> | n | % | n | % |
| Prior Receipt<br>of H5 Influenza<br>Vaccine | No Prior H5 Influenza<br>Vaccinations | | | | | | | | | | | | | | |
| | Received Prior H5 Influenza<br>Vaccinations | | | | | | | | | | | | | | |

N= Number of subjects enrolled.

**Table 22:** Summary of Continuous Baseline Characteristics by Study Group, All Enrolled Subjects

| | 2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | 2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | All<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Mean | X.X | X.X | X.X | X.X | X.X | x.x | x.x |
| Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | x.x |
| Median | X.X | X.X | X.X | X.X | X.X | x.x | x.x |
| Minimum | x | X | X | X | х | X | Х |
| Maximum | X | X | X | X | X | X | х |
| Mean | X.X | X.X | x.x | X.X | X.X | x.x | x.x |
| Standard Deviation | X.X | X.X | X.X | X.X | X.X | x.x | x.x |
| Median | X.X | X.X | x.x | X.X | X.X | x.x | x.x |
| Minimum | X | Х | X | X | X | X | х |
| Maximum | X | X | X | X | X | X | X |
| | Standard Deviation Median Minimum Maximum Mean Standard Deviation Median Minimum | 3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) Mean x.x Standard Deviation x.x Median x.x Minimum x Mean x.x Standard Deviation x.x Standard Deviation x.x Median x.x Median x.x Minimum x Maximum x | 3.75+AS03/ 3.75+AS03/ 2017 3.75+AS03 3.75+AS03 3.75+AS03 (D1-D22) (D1-D121) (N=X) X.X Mean X.X X.X Median X.X X.X Maximum X X Mean X.X X.X Standard Deviation X.X X.X Median X.X X.X Median X.X X.X Minimum X X Maximum X X Maximum X X | 3.75+AS03/ 2017 2017 3.75+AS03/ 2017 15 (D1-D121) (N=X) (N=X | 3.75+AS03/ 2017 2017 3.75+AS03/ 2017 3.75+AS03 2017 3.75+AS03 (D1-D121) (N=X) (N=X) | 3.75+AS03/ 2017 2017 2017 3.75+AS03/ (D1-D121) (N=X) (N=X) | Mean |

N= Number of subjects enrolled.

### 14.1.3 Prior and Concurrent Medical Conditions

Table 23: Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA® System Organ Class and Study Group, Safety Population

| MedDRA® System Organ Class | Groud<br>201<br>3.75+A<br>201<br>3.75+A<br>(D1-I<br>(N=) | 3<br>AS03/<br>7<br>AS03<br>D22) | Grou<br>201<br>3.75+4<br>201<br>3.75+4<br>(D1-I<br>(N= | 13<br>AS03/<br>17<br>AS03<br>D121) | Group 3<br>2013<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | | Group 5 2017 3.75+AS03/ 2017 3.75+AS03 (D1-D121) (N=X) | | Group 6<br>2017<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | | All<br>Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| [SOC 1] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| [SOC 2] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |

N=Number of subjects in the Safety Population;

n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

### 14.2 Immunogenicity Data

# 14.2.1 Antibody Response Against 2013 and 2017 A/H7N9

Table 24: Summaries of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population\*

| Time Point | Statistic | Group 1<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 1 | n | x | x | x | x | x | X |
| (Pre-Vaccination 1) | GMT (95% CI)° | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) d | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Day 22 Post | n | х | х | х | x | x | X |
| Vaccination 1 | GMT (95% CI) <sup>c</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) <sup>d</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>c</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Seroconversion - % (95% CI) <sup>d</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Day 121 post | n | NA | x | x | NA | X | X |
| Vaccination 1 | GMT (95% CI) <sup>c</sup> | NA | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | NA | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) <sup>d</sup> | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>c</sup> | NA | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | NA | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |

| Time Point | Statistic | Group 1<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | 2013 2013 20<br>3.75+AS03/ 3.75+AS03/ 3.75+<br>2017 2017 2017 201<br>3.75+AS03 3.75+AS03 (D1-<br>(D1-D22) (D1-D121) (N | | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | Seroconversion - % (95% CI) <sup>d</sup> | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) |
| Day 22 Post | n | x | x | x | x | x | X |
| Vaccination 2 <sup>a</sup> | GMT (95% CI) <sup>c</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) <sup>d</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>c</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Seroconversion - % (95% CI) <sup>d</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Day 181 Post | n | х | х | X | x | х | х |
| Vaccination 2 <sup>b</sup> | GMT (95% CI) <sup>c</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) <sup>d</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>c</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| | Seroconversion - % (95% CI) <sup>d</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

N = number of subjects in the Modified Intent-to-Treat Population; n = number of subjects with available results; GMT = Geometric Mean Titer; GMFR = Geometric Mean Fold Rise (relative to baseline).

<sup>&</sup>lt;sup>a</sup> Day 22 post vaccination 2 varies by group (Day 43 for Groups 1 and 4; Day 142 for Groups 2, 3,5, and 6).

<sup>&</sup>lt;sup>b</sup> Day 181 post vaccination 2 varies by group (Day 202 for Groups 1 and 4; Day 301 for Groups 2, 3,5, and 6).

 $<sup>^{\</sup>rm c}$  Confidence Interval calculated based on the student's T distribution.

 $<sup>^{\</sup>rm d}$  Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 25: Summaries of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Per Protocol Population\*
- Table 26: Summaries of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population\*
- Table 27: Summaries of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Day and Study Group, Per Protocol Population\*
- Table 28: Summaries of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population\*
- Table 29: Summaries of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Per Protocol Population\*
- Table 30: Summaries of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Modified Intent-to-Treat Population\*
- Table 31: Summaries of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Day and Study Group, Per Protocol Population\*

Table 32: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population

| Statistic | Group 1<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | Age 19-34 years | | | |
| n | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | (xx, xx) xx (xx, xx) | | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | | | Age 35-50 years | | | |
| n | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | | | | | | |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

N = number of subjects in the Per Protocol Population; n = number of subjects with available results; GMT = Geometric Mean Titer; GMFR = Geometric Mean Fold Rise (relative to baseline).

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 33: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population
- Table 34: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population
- Table 35: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population
- Table 36: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population
- Table 37: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population
- Table 38: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 21 Days Post Second Vaccination, Per Protocol Population
- Table 39: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Age Group at 180 Days Post Second Vaccination, Per Protocol Population

Table 40: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population

| Statistic | Group 1<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | Female | | | |
| n | X | X | X | Х | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | | | Male | | | |
| n | X | X | X | Х | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

N = number of subjects in the Per Protocol Population; n = number of subjects with available results; GMT = Geometric Mean Titer; GMFR = Geometric Mean Fold Rise (relative to baseline).

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 41: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 180 Days Post Second Vaccination, Per Protocol Population
- Table 42: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population
- Table 43: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Sex at 180 Days Post Second Vaccination, Per Protocol Population
- Table 44: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population
- Table 45: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 180 Days Post Second Vaccination, Per Protocol Population
- Table 46: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 21 Days Post Second Vaccination, Per Protocol Population
- Table 47: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Sex at 180 Days Second Vaccination, Per Protocol Population

Table 48: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population

| Statistic | Group 1<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | BMI < 30 | | | |
| n | X | X | X | Х | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | | | <b>BMI</b> ≥ 30 | | | |
| n | X | X | X | Х | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

N = number of subjects in the Per Protocol Population; n = number of subjects with available results; GMT = Geometric Mean Titer; GMFR = Geometric Mean Fold Rise (relative to baseline).

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 49: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 180 Days Post Second Vaccination, Per Protocol Population
- Table 50: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population
- Table 51: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and BMI at 180 Days Post Second Vaccination, Per Protocol Population
- Table 52: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population
- Table 53: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 180 Days Post Second Vaccination, Per Protocol Population
- Table 54: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 21 Days Post Second Vaccination, Per Protocol Population
- Table 55: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and BMI at 180 Days Second Vaccination, Per Protocol Population

Table 56: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Seasonal Influenza Vaccination Status at 21 Days Post Second Vaccination, Per Protocol Population

| Receipt of 2018-<br>2019 Seasonal<br>Influenza Vaccine | Statistic | Group 1<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | | Did Not Receive Pr | ior 2016-2017 or 201 | 7-2018 Seasonal Infl | uenza Vaccination | | |
| Did Not Receive | n | X | X | X | X | X | Х |
| 2018-2019 Seasonal<br>Influenza Vaccine | GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| | Titer $\ge 1:40 - \%(95\%$<br>CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| | Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Received 2018-2019 | n | X | X | X | X | X | Х |
| Seasonal Influenza<br>Vaccine | GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| | Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | | Received Prior 20 | 16-2017 and/or 2017 | -2018 Seasonal Influ | enza Vaccination | | |
| Did Not Receive | n | X | X | X | X | X | Х |
| 2018-2019 Seasonal<br>Influenza Vaccine | GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |

| Receipt of 2018-<br>2019 Seasonal<br>Influenza Vaccine | Statistic | Group 1<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Received 2018-2019 | n | X | X | X | X | X | x |
| Seasonal Influenza<br>Vaccine | GMT (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| | Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| | Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

Note: Receipt of 2018-2019 vaccine is counted at any timepoint prior to receipt of the second study vaccination.

N = number of subjects in the Per Protocol Population; n = number of subjects with available results; GMT = Geometric Mean Titer; GMFR = Geometric Mean Fold Rise (relative to baseline).

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 57: Summary of Hemagglutination Inhibition Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per Protocol Population
- Table 58: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per Protocol Population
- Table 59: Summary of Neutralizing Antibody Against A/Shanghai/2/2013 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per Protocol Population
- Table 60: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per Protocol Population
- Table 61: Summary of Hemagglutination Inhibition Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per Protocol Population
- Table 62: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per Protocol Population
- Table 63: Summary of Neutralizing Antibody Against A/Hong Kong/125/2017 (A/H7N9) by Study Group and Prior Seasonal Influenza Vaccination at 180 Days Second Vaccination, Per Protocol Population

Table 64: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Per Protocol Population

[Implementation Note: Two- and three-way interaction terms will be included in the model at first. If interactions are not significant, fit final model in this table without interaction, and add footnote in table "No interaction terms were significant."]

| Model | Parameter Category | A | \/Shangh | ai/2/2013 | (A/H7N9 | <b>)</b> ) | A/Hong Kong/125/2017 (A/H7N9) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | Parameter<br>Estimate | SE | p-value | Odds<br>Ratio | 95%CI | Parameter<br>Estimate | SE | p-value | Odds<br>Ratio | 95%CI |
| Intercept | N/A | XXX.X | xxx.x | x.xxx | - | - | XXX.X | XXX.X | x.xxx | - | - |
| Prime-boost | Homologous (reference) | - | - | - | - | - | - | - | - | - | - |
| | Heterologous | xxx.x | XXX.X | x.xxx | XX.X | XX.X-XX.X | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |
| Boost Dose | 15 mcg (reference) | - | - | - | - | - | - | - | - | - | - |
| | 3.75 mcg + AS03 | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x | XXX.X | xxx.x | x.xxx | XX.X | xx.x-xx.x |
| Interval | 21 days (reference) | - | - | _ | - | - | - | - | - | - | - |
| | 120 days | XXX.X | xxx.x | X.XXX | XX.X | XX.X-XX.X | xxx.x | xxx.x | x.xxx | XX.X | XX.X-XX.X |

n= XX (number of subjects with results available at 21 days post second study vaccination in the Per Protocol Population.)

- Table 65: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Per Protocol Population
- Table 66: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Per Protocol Population
- Table 67: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Per Protocol Population

XX subjects missing covariate data were excluded from this analysis.

SE = Standard Error.

Table 68: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population (N=X)

| Model Parameter | Parameter Category | A/Sh | anghai | 2/2013 | (A/H7N | N9) | A/Hong Kong/125/2017 (A/H7N9) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Parameter<br>Estimate | SE | p-<br>value | Odds<br>Ratio | 95%CI | Parameter<br>Estimate | SE | p-<br>value | Odds<br>Ratio | 95%CI |
| Intercept | N/A | xxx.x | xxx.x | x.xxx | - | - | xxx.x | xxx.x | x.xxx | - | - |
| Prime-boost | Homologous (reference) | - | - | - | - | - | - | - | - | - | - |
| | Heterologous | xxx.x | xxx.x | x.xxx | xx.x | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | xx.x | XX.X-<br>XX.X |
| Boost Dose | 15 mcg (reference) | - | - | - | - | - | - | - | - | - | - |
| | 3.75 mcg + AS03 | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X |
| Interval | 21 days (reference) | - | - | - | - | - | - | - | - | - | - |
| | 120 days | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X |
| Age (years) | N/A | XXX.X | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X |
| Sex | Female (reference) | - | - | - | - | - | - | - | - | - | - |
| | Male | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X |
| BMI | <30 (reference) | - | - | - | - | - | - | - | - | - | - |
| | ≥30 | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X |
| Prior Receipt of Influenza Vaccine<br>(Prior Seasons) | Did Not Receive 2016-2017 or<br>2017-2018 Seasonal Influenza<br>Vaccination (reference) | - | - | - | - | - | - | - | - | - | - |
| | Received 2016-2017 and/or<br>2017-2018 Seasonal Influenza<br>Vaccination | XXX.X | xxx.x | x.xxx | xx.x | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | xx.x | XX.X-<br>XX.X |

| Model Parameter | Parameter Category | A/Shanghai/2/2013 (A/H7N9) | | | | | A/Hong Kong/125/2017 (A/H7N9) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Parameter<br>Estimate | SE | p-<br>value | Odds<br>Ratio | 95%CI | Parameter<br>Estimate | SE | p-<br>value | Odds<br>Ratio | 95%CI |
| Receipt of Influenza Vaccine<br>(Concurrent Season) | Did Not Receive 2018-2019<br>Seasonal Influenza Vaccine<br>(reference) | - | - | - | - | - | - | - | - | - | - |
| | Received 2018-2019 Seasonal<br>Influenza Vaccine (reference) | xxx.x | xxx.x | x.xxx | xx.x | XX.X-<br>XX.X | XXX.X | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X |
| Prior Receipt of H5 Influenza<br>Vaccine | No Prior H5 Influenza<br>Vaccinations | - | - | - | - | - | - | - | - | - | - |
| | Received Prior H5 Influenza<br>Vaccinations | xxx.x | xxx.x | x.xxx | XX.X | XX.X-<br>XX.X | xxx.x | xxx.x | x.xxx | xx.x | XX.X-<br>XX.X |

Note: Receipt of 2018-2019 vaccine is counted at any timepoint prior to receipt of the second study vaccination.

n= XX (number of subjects with results available at 21 days post second study vaccination in the Per Protocol Population).

XX subjects missing covariate data were excluded from this analysis.

SE = Standard Error.

#### Tables with similar format:

Table 69: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population

Table 70: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population

Table 71: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population

Table 72: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Per Protocol Population (N=X)

| Model Parameter | Parameter Category | A/Sł | anghai/2/20 | )13 (A/H7N9 | A/Hong Kong/125/2017 (A/H7N9) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Parameter<br>Estimate | SE | 95%CI | p-value | Parameter<br>Estimate | SE | 95%CI | p-value |
| Intercept | N/A | XXX.X | xxx.x | x.xxx | x.xxx | xxx.x | xxx.x | x.xxx | x.xxx |
| Prime-boost | Homologous (reference) | - | - | - | - | - | - | - | - |
| | Heterologous | XXX.X | xxx.x | x.xxx | xx.x | xxx.x | xxx.x | x.xxx | xx.x |
| Boost Dose | 15 mcg (reference) | - | - | - | - | - | - | - | - |
| | 3.75 mcg + AS03 | XXX.X | xxx.x | x.xxx | xx.x | xxx.x | xxx.x | x.xxx | xx.x |
| Interval | 21 days (reference) | - | - | - | - | - | - | - | - |
| | 120 days | XXX.X | xxx.x | x.xxx | XX.X | xxx.x | xxx.x | x.xxx | xx.x |

n = XX (number of subjects with results available at 21 days post second study vaccination in the Per Protocol Population).

- Table 73: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Per Protocol Population
- Table 74: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Per Protocol Population
- Table 75: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Per Protocol Population

XX subjects missing covariate data were excluded from this analysis.

SE = Standard Error.

Table 76: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population

| Model Parameter | Parameter Category | A/Sha | nghai/2/2 | 013 (A/H7N | [9) | A/Hong I | Kong/12 | 5/2017 (A/I | 17N9) |
|---|---|---|---|---|---|---|---|---|---|
| | | Parameter<br>Estimate | SE | 95%CI | p-<br>value | Parameter<br>Estimate | SE | 95%CI | p-<br>value |
| Intercept | N/A | xxx.x | xxx.x | - | X.XXX | XXX.X | xxx.x | - | x.xxx |
| Prime-boost | Homologous (reference) | - | - | - | - | - | - | - | - |
| | Heterologous | XXX.X | xxx.x | x.xxx | XX.X | XXX.X | xxx.x | x.xxx | XX.X |
| Boost Dose | 15 mcg (reference) | - | - | - | - | - | - | - | - |
| | 3.75 mcg + AS03 | XXX.X | xxx.x | x.xxx | XX.X | XXX.X | xxx.x | x.xxx | XX.X |
| Interval | 21 days (reference) | - | - | - | - | - | - | - | - |
| | 120 days | xxx.x | xxx.x | x.xxx | XX.X | XXX.X | xxx.x | x.xxx | XX.X |
| Age (years) | N/A | xxx.x | xxx.x | xx.x-xx.x | X.XXX | XXX.X | xxx.x | xx.x-xx.x | x.xxx |
| Sex | Female (reference) | - | - | - | - | - | - | - | - |
| | Male | xxx.x | xxx.x | xx.x-xx.x | X.XXX | XXX.X | xxx.x | xx.x-xx.x | x.xxx |
| BMI | <30 (reference) | - | - | - | - | - | - | - | - |
| | ≥30 | XXX.X | xxx.x | xx.x-xx.x | X.XXX | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| Prior Receipt of Influenza Vaccine<br>(Prior Seasons) | Did Not Receive 2016-2017 or 2017-<br>2018 Seasonal Influenza Vaccination<br>(reference) | - | - | - | - | - | - | - | - |
| | Received 2016-2017 and/or 2017-<br>2018 Seasonal Influenza Vaccination | xxx.x | XXX.X | xx.x-xx.x | X.XXX | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| Receipt of Influenza Vaccine<br>(Concurrent Season) | Did Not Receive 2018-2019 Seasonal<br>Influenza Vaccine (reference) | - | - | - | - | | - | - | - |
| | Received 2018-2019 Seasonal<br>Influenza Vaccine (reference) | xxx.x | XXX.X | xx.x-xx.x | x.xxx | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| | No Prior H5 Influenza Vaccinations | - | - | - | - | - | - | - | - |

| Model Parameter | Parameter Category | A/Sha | nghai/2/2( | 013 (A/H7N | A/Hong Kong/125/2017 (A/H7N9) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Parameter<br>Estimate | SE | 95%CI | p-<br>value | Parameter<br>Estimate | SE | 95%CI | p-<br>value |
| Prior Receipt of H5 Influenza<br>Vaccine | Received Prior H5 Influenza<br>Vaccinations | xxx.x | xxx.x | xx.x-xx.x | X.XXX | XXX.X | XXX.X | xx.x-xx.x | x.xxx |

Note: Receipt of 2018-2019 vaccine is counted at any timepoint prior to receipt of the second study vaccination.

n = XX (number of subjects with results available at 21 days post second study vaccination in the Per Protocol Population).

XX subjects missing covariate data were excluded from this analysis.

SE = Standard Error.

- Table 77: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population
- Table 78: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population
- Table 79: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer Against A/H7N9 Strains at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population

# 14.2.2 Plasmablast Response Against 2013 and 2017 A/H7N9

Table 80: Summary of A/Shanghai/2/2013 (A/H7N9)—Specific Antibody Secreting Cells by Immunoglobulin Type, Study Group, and Study Day, Per Protocol Population

| Time Point | Statistic | tic Group 1 Group 2 Group 3 2013 3.75+AS03/ 2013 3.75+AS03/ 2013 3.75+AS03/ 2017 3.75+AS03 2017 3.75+AS03 2017 15 (D1-D22) (D1-D121) (D1-D121) (N=X) (N=X) IgA Antibody Secreting Cells | | Group 4<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| | | | IgA A | antibody Secreting Cells | | | |
| Day 8 Post | n | X | X | X | X | x | X |
| Vac 1 | Mean (SD) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Median<br>[IQR] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 8 Post | n | х | X | X | X | x | х |
| Vac 2 <sup>a</sup> | Mean (SD) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Median<br>[IQR] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | | | IgG A | antibody Secreting Cells | | | |
| Day 8 Post | n | х | Х | X | x | х | х |
| Vac 1 | Mean (SD) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Median<br>[IQR] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | n | х | Х | X | х | х | Х |

| Time Point | Statistic | Group 1<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 2<br>2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 3<br>2013 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | Group 4<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Group 6<br>2017 3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 8 Post | Mean (SD) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| Vac 2 <sup>a</sup> | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | [IQR] | | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | | | IgM A | antibody Secreting Cells | | | |
| Day 8 Post | n | х | X | X | x | х | X |
| Vac 1 | Mean (SD) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Median<br>[IQR] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 8 Post | n | х | X | X | X | х | х |
| Vac 2 <sup>a</sup> | Mean (SD) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Median<br>[IQR] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] | xx [xx, xx] |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

N = Number of subjects in the Modified Intent-to-Treat Population; n = number of subjects with results reported.

Table 81: Summary of A/Hong Kong/125/2017 (A/H7N9)—Specific Antibody Secreting Cells by Immunoglobulin Type, Study Group, and Study Day, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8 post vaccination 2 varies by group (Day 29 for Groups 1 and 4; Day 128 for Groups 2, 3,5, and 6).

# 14.3 Safety Data

# 14.3.1 Displays of Adverse Events

**Table 82:** Overall Summary of Adverse Events, Safety Population\*

| AE Category | AE Subcategory | 2013<br>3.75+AS03/<br>2017<br>2017<br>2017<br>3.75+AS03<br>3.75+AS03 | | Group 3<br>2013<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | | Group 5<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | | 201<br>(D1- | Group 6<br>2017<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | | All<br>ojects<br>(=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one local solicited adverse event | - | X | x | х | X | х | х | х | X | х | х | х | х | x | X |
| At least one systemic solicited adverse event | - | Х | x | X | х | х | Х | х | х | Х | х | х | Х | х | х |
| At least one laboratory adverse | Any Grade | Х | X | x | x | х | X | X | X | x | X | х | X | X | X |
| event | Mild (Grade 1) | Х | X | X | X | х | X | х | x | x | х | х | X | х | x |
| | Moderate (Grade 2) | X | X | X | X | X | X | x | X | X | X | X | X | х | x |
| | Severe (Grade 3) | X | X | X | X | X | X | X | X | X | X | X | X | X | x |
| At least one unsolicited adverse event | - | X | X | x | X | x | X | X | X | X | X | x | X | x | X |
| At least one related unsolicited | Any Grade | Х | X | X | X | х | X | х | x | x | х | х | Х | х | x |
| adverse event | Mild (Grade 1) | Х | X | x | x | х | X | X | X | x | X | х | X | X | X |
| | Moderate (Grade 2) | Х | X | x | x | х | X | X | X | x | X | х | X | X | X |
| | Severe (Grade 3) | Х | X | X | X | x | X | X | X | X | X | X | X | х | X |
| At least one severe (Grade 3) | Any Relationship | Х | X | X | X | x | X | X | X | X | X | Х | X | Х | X |
| unsolicited adverse event | Related | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | Unrelated | X | X | X | X | X | X | x | x | X | X | X | X | X | x |

| AE Category | AE Subcategory | 2017<br>3.75+AS03 | | Group 2<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | | Group 3<br>2013<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | | 7 2017<br>3.75+AS0<br>7 2017<br>AS03 3.75+AS<br>022) (D1-D12 | | 2017<br>3.75+AS03/<br>2017 15<br>03 (D1-D121)<br>(N=X) | | Sub | All ojects =X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one serious adverse event <sup>b</sup> | - | х | X | х | x | х | х | X | X | Х | Х | х | x | х | X |
| At least one related, serious adverse event | - | х | X | х | x | х | х | X | X | Х | X | х | x | х | x |
| At least one adverse event leading to early termination <sup>c</sup> | - | х | Х | х | x | х | x | X | X | X | Х | х | х | х | Х |
| At least one medically attended adverse event | - | х | Х | х | x | х | x | X | X | X | Х | х | х | х | Х |
| At least one new onset chronic medical condition | - | Х | Х | х | х | х | х | X | X | X | Х | х | X | | |
| At least one potentially immune mediated medical condition | - | х | х | X | х | х | х | X | х | х | х | Х | х | | |

N = Number of subjects who received at least one study vaccination; n= Number of subjects in the indicated category

<sup>&</sup>lt;sup>a</sup> Subjects are counted once for each category regardless of the number of events.

<sup>&</sup>lt;sup>b</sup> A listing of Serious Adverse Events is included in ****.

<sup>&</sup>lt;sup>c</sup> As reported on the Adverse Event eCRF.
Table 83: Number of Adverse Events Occurring in 5% of Subjects in Any Study Group by MedDRA® System Organ Class and Preferred Term, and Study Group, Safety Population

[Implementation Note: this table combines all adverse events – solicited events, unsolicited events, and clinical laboratory events. Sort data by SOC then PT. If >= X SAEs are reported, repeat this table for all reported SAEs]

| MedDRA System<br>Organ Class | Preferred<br>Term | | 2(<br>3.75+<br>2(<br>3.75-<br>(D1- | oup 1<br>013<br>-AS03/<br>017<br>-AS03<br>-D22)<br>=X) | | 20<br>3.75+<br>20<br>3.75-<br>(D1- | oup 2<br>013<br>-AS03/<br>017<br>+AS03<br>D121)<br>=X) | | 20<br>3.75+<br>201<br>(D1- | oup 3<br>013<br>-AS03/<br>17 15<br>D121)<br>=X) | | 20<br>3.75+<br>20<br>3.75-<br>(D1- | oup 4<br>017<br>+AS03/<br>017<br>+AS03<br>-D22)<br>(=X) | | 20<br>3.75+<br>20<br>3.75+<br>(D1- | oup 5<br>017<br>AS03/<br>017<br>+AS03<br>D121)<br>=X) | | 201<br>(D1- | oup 6<br>017<br>-AS03/<br>-7 15<br>D121)<br>=X) | F | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| | | | | | | | Seri | ous | Adve | erse Events | S | | | | | | | | | | | |
| All | All | X | X | X | X | X | X | X | x | X | X | x | X | X | X | X | X | X | X | X | X | X |
| SOC1 | PT1 | x | X | X | X | x | X | X | x | x | X | x | X | X | X | X | X | X | x | X | X | x |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | Other (No: | n-se | rious | ) Adverse | Eve | nts | | | | | | | | | | |
| All | All | X | X | X | X | х | X | x | х | X | x | х | Х | х | X | X | | | | X | х | Х |
| SOC1 | PT1 | X | Х | X | х | х | Х | x | х | Х | X | х | Х | х | Х | X | | | | Х | х | X |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | | | | |

N = number of subjects in the Safety Population (number of subjects at risk); n= number of subjects reporting event. Events = total frequency of events reported. MedDRA Version X.X.

#### 14.3.1.1 Solicited Adverse Events

Table 84: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Study Group (Safety Population) – Post Any Study Vaccination

| Symptom | 2<br>3.75-<br>2017 3.<br>(D1 | oup 1<br>013<br>+AS03/<br>75+AS03<br>-D22)<br>(=X) | 3.75<br>2017 3<br>(D) | roup 2<br>2013<br>5+AS03/<br>3.75+AS03<br>1-D121)<br>N=X) | 3.7<br>2<br>(D | Group 3<br>2013<br>5+AS03/<br>017 15<br>1-D121)<br>(N=X) | 2<br>3.75-<br>2017 3.<br>(D1 | oup 4<br>017<br>+AS03/<br>.75+AS03<br>-D22) | 3.75<br>2017 3<br>(D1 | roup 5<br>2017<br>+AS03/<br>.75+AS03<br>-D121)<br>N=X) | 3.75<br>20<br>(D1 | roup 6<br>2017<br>5+AS03/<br>017 15<br>D121)<br>N=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95% CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) |
| Any Symptom | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| Any Systemic Symptom | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| Fever | X | xx<br>(xx-xx) | x | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Feverishness | X | xx<br>(xx-xx) | x | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | x | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Fatigue | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| Malaise | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Myalgia | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| Arthralgia | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| Headache | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |

| Symptom | 3.75-<br>2017 3.<br>(D1 | oup 1<br>013<br>+AS03/<br>75+AS03<br>-D22)<br>I=X) | 3.75<br>2017 3<br>(D) | roup 2<br>2013<br>5+AS03/<br>3.75+AS03<br>1-D121)<br>N=X) | 3.7<br>2<br>(D | 2013<br>5+AS03/<br>017 15<br>1-D121)<br>(N=X) | 2<br>3.75-<br>2017 3.<br>(D1 | oup 4<br>017<br>+AS03/<br>.75+AS03<br>-D22)<br>U=X) | 3.75<br>2017 3<br>(D1 | roup 5<br>2017<br>++AS03/<br>.75+AS03<br> -D121)<br>N=X) | 3.75<br>20<br>(D1 | roup 6<br>2017<br>3+AS03/<br>017 15<br>1-D121)<br>N=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95% CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) |
| Nausea | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | x | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Any Local Symptom | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Pain | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | x | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Tenderness | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Pruritus | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | x | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Ecchymosis | X | xx<br>(xx-xx) | x | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Ecchymosis (measurement) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Erythema | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Erythema (measurement) | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Induration/Swelling | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) |
| Induration/Swelling (measurement) | X | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |

| Symptom | 2017 3. (D1 | oup 1<br>013<br>+AS03/<br>75+AS03<br>-D22)<br>[=X) | 3.75<br>2017 3<br>(D1 | roup 2<br>2013<br>5+AS03/<br>3.75+AS03<br>1-D121)<br>N=X) | 3.7<br>2<br>(D | 2013<br>'5+AS03/<br>2017 15<br>11-D121)<br>(N=X) | 3.75-<br>2017 3.<br>(D1 | oup 4<br>017<br>+AS03/<br>75+AS03<br>-D22)<br>(=X) | 2<br>3.75-<br>2017 3.<br>(D1 | oup 5<br>017<br>+AS03/<br>.75+AS03<br>-D121) | 3.75<br>20<br>(D1 | roup 6<br>2017<br>+AS03/<br>17 15<br>-D121)<br>N=X) | | abjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95% CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) |

N = Number of subjects in the Safety Population who received any study vaccination;

Table 85: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Study Group (Safety Population) – Post Study Vaccination 1

[Footnote update] N = Number of subjects in the Safety Population who received the first study vaccination.

Table 86: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Study Group (Safety Population) – Post Study Vaccination 2

[Footnote update] N = Number of subjects in the Safety Population who received the second study vaccination.

n = Number of subjects reporting event

<sup>95%</sup> CI estimated using the Clopper-Pearson exact method

# Table 87: Logistic Regression Model to Evaluate the Relationship of Study Vaccination with Reporting Any Local Event Post Second Study Vaccination, Safety Population

[Implementation Note: If statistically significant effects (defined as p-value <0.05) are observed in the model for local events then this table should be repeated for additional models which will be fit for each individual local event. Any solicited local event grade 1 or higher reported within 7 days of study vaccination will count as a reported event.]

| Model Parameter | Parameter Category | Parameter<br>Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| Intercept | N/A | xxx.x | xxx.x | x.xxx | - | - |
| Prime-boost | Homologous (reference) | - | - | - | - | - |
| | Heterologous | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Boost Dose | 15 mcg (reference) | - | - | - | - | - |
| | 3.75 mcg + AS03 | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Interval | 21 days (reference) | - | - | - | - | - |
| | 120 days | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| N = XX (number of subjects | s in the Safety Population) | | | | | |

Table with similar format:

## Table 88: Logistic Regression Model to Evaluate the Relationship of Study Vaccination with Reporting Any Systemic Event Post Second Study Vaccination, Safety Population

[Implementation Note: If statistically significant effects defined p-value <0.05 are observed in the model for systemic events then this table should be repeated for additional models which will be fit for each individual systemic event. Any solicited systemic event grade 1 or higher reported within 7 days of study vaccination will count as a reported event.]

Table 89: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Study Group (Safety Population) – Post Any Study Vaccination

| Symptom | Severity | 3. <sup>2</sup> 2017 | Group 1<br>2013<br>75+AS03/<br>73.75+AS03<br>D1-D22)<br>(N=X) | 3<br>201 | Group 2<br>2013<br>.75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3 | Group 3 2013 75+AS03/ 2017 15 D1-D121) (N=X) | 3.<br>201 | Group 4<br>2017<br>75+AS03/<br>7 3.75+AS03<br>(D1-D22)<br>(N=X) | 3.<br>201 | Group 5<br>2017<br>75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3. | Group 6<br>2017<br>75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | A | ll Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| Any Symptom | None | X | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| Any Systemic<br>Symptom | None | X | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| Fever | None | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| Feverishness | None | X | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |

| Symptom | Severity | 3.′<br>2017 | Group 1<br>2013<br>75+AS03/<br>73.75+AS03<br>D1-D22)<br>(N=X) | 3<br>201 | Group 2<br>2013<br>.75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3 | Group 3<br>2013<br>.75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | 3.<br>201 | Group 4<br>2017<br>75+AS03/<br>7 3.75+AS03<br>(D1-D22)<br>(N=X) | 3.<br>2017 | Group 5<br>2017<br>75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3. | Group 6<br>2017<br>75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | A | ll Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| Fatigue | None | X | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Malaise | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Myalgia | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Arthralgia | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Headache | None | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |

| Symptom | Severity | 3. <sup>2</sup> 2017 | Group 1<br>2013<br>75+AS03/<br>73.75+AS03<br>D1-D22)<br>(N=X) | 3<br>201 | Group 2<br>2013<br>.75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3 | Group 3<br>2013<br>.75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | 3.<br>201 | Group 4<br>2017<br>75+AS03/<br>7 3.75+AS03<br>(D1-D22)<br>(N=X) | 3.<br>2017 | Group 5<br>2017<br>75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3. | Group 6<br>2017<br>75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | A | ll Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Nausea | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Any Local<br>Symptom | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Pain | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Tenderness | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Pruritus | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |

| Symptom | Severity | 3.′<br>2017 | Group 1<br>2013<br>75+AS03/<br>73.75+AS03<br>D1-D22)<br>(N=X) | 3<br>201 | Group 2<br>2013<br>.75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3 | Group 3<br>2013<br>.75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | 3.<br>201 | Group 4<br>2017<br>75+AS03/<br>7 3.75+AS03<br>(D1-D22)<br>(N=X) | 3.<br>2017 | Group 5<br>2017<br>75+AS03/<br>73.75+AS03<br>D1-D121)<br>(N=X) | 3. | Group 6<br>2017<br>75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | A | ll Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Ecchymosis | None | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| Ecchymosis (measurement) | None | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Erythema | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Erythema (measurement) | None | X | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |

| Symptom | Severity | 3.′<br>2017 | Group 1<br>2013<br>75+AS03/<br>23.75+AS03<br>D1-D22)<br>(N=X) | 3<br>201 | Group 2<br>2013<br>.75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3 | Group 3<br>2013<br>.75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | 3.<br>201 | Group 4<br>2017<br>75+AS03/<br>7 3.75+AS03<br>(D1-D22)<br>(N=X) | 3.<br>2017 | Group 5<br>2017<br>75+AS03/<br>7 3.75+AS03<br>D1-D121)<br>(N=X) | 3. | Group 6<br>2017<br>75+AS03/<br>2017 15<br>D1-D121)<br>(N=X) | A | ll Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Induration/Swelling | None | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| Induration/Swelling (measurement) | None | X | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | х | xx (xx-xx) | Х | xx (xx-xx) | х | xx (xx-xx) |
| | Mild | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Moderate | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Severe | X | xx (xx-xx) | X | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |

N = Number of subjects in the Safety Population who received any study vaccination; n = Number of subjects reporting event.

<sup>95%</sup> CI estimated using Clopper-Pearson exact method.

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

Table 90: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Study Group (Safety Population) – Post Study Vaccination 1

[Footnote Update] N = Number of subjects in the Safety Population who received the first study vaccination = Number of subjects reporting event.

Table 91: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Study Group (Safety Population) – Post Study Vaccination 2

[Footnote Update] N = Number of subjects in the Safety Population who received the second study vaccination; n = Number of subjects reporting event.

Table 92: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, and Study Group (Safety Population) – Post Any Study Vaccination

| Symptom | Severity | Pre-Vac Post-Vac Day 1 D n % n % n % n % n Group 1: 2013 3.75+AS03/ 2017 3.75+ | | | | | | | | Da | ıy 3 | Da | ıy 4 | Da | ıy 5 | Da | ıy 6 | Da | ıy 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | • | Grou | p 1: 2 | 013 3 | .75+A | S03/ | 2017 | 3.75+ | AS03 (I | D1-D2 | 22) (N | (=X) | • | | | | | • | | | |
| Any Symptom | None | X | XX | X | XX | X | XX | X | xx | Х | xx | X | XX | X | XX | X | xx | X | XX | X | XX |
| | Mild | х | XX | X | XX | х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | Х | XX | X | XX |
| | Moderate | X | XX | X | XX | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Severe | X | XX | X | XX | X | xx | X | XX | x | xx | X | XX | X | xx | X | XX | x | xx | X | XX |
| Any Systemic Symptom | None | Х | XX | Х | XX | х | XX | Х | xx | х | xx | Х | XX | X | XX | X | XX | Х | XX | X | XX |
| | Mild | х | XX | X | XX | х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | Х | XX | X | XX |
| | Moderate | X | XX | X | XX | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Severe | X | XX | X | XX | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Fever | None | X | XX | X | XX | x | XX | X | XX | Х | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Mild | X | XX | X | XX | х | XX | X | xx | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX |
| | Moderate | X | XX | X | XX | х | XX | X | xx | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX |
| | Severe | X | XX | X | XX | x | XX | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Feverishness | None | X | XX | X | XX | x | XX | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Mild | X | XX | X | XX | x | XX | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Moderate | X | XX | X | XX | x | XX | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Severe | X | XX | X | XX | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Fatigue | None | X | XX | X | XX | X | XX | X | xx | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX |
| | Mild | X | XX | X | XX | X | XX | X | xx | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX |
| | Moderate | X | XX | X | XX | X | XX | X | xx | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX |
| | Severe | X | XX | X | XX | x | XX | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |

| Symptom | Severity | Pre | -Vac | Pos | t-Vac | D | ay 1 | Da | ıy 2 | Da | ıy 3 | Da | y 4 | Da | ıy 5 | Da | ny 6 | Da | ıy 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Malaise | None | х | XX | х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | х | XX | Х | XX | X | XX |
| | Mild | Х | XX | Х | XX | х | XX | х | XX | X | XX | X | XX | X | XX | х | XX | X | XX | х | XX |
| | Moderate | х | XX | х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | х | XX | Х | XX | X | XX |
| | Severe | Х | XX | Х | XX | х | XX | х | XX | X | XX | X | XX | X | XX | х | XX | X | XX | х | XX |
| Myalgia | None | х | XX | Х | xx | Х | XX | х | XX | X | XX | Х | XX | X | XX | х | XX | X | XX | х | XX |
| | Mild | х | XX | Х | xx | Х | XX | х | XX | X | XX | Х | XX | X | XX | х | XX | X | XX | х | XX |
| | Moderate | х | XX | Х | xx | Х | XX | х | XX | X | XX | Х | XX | X | XX | х | XX | X | XX | х | XX |
| | Severe | х | XX | Х | xx | Х | XX | х | xx | X | XX | X | XX | X | XX | х | xx | Х | XX | Х | XX |
| Arthralgia | None | х | XX | Х | xx | Х | XX | х | XX | X | XX | Х | XX | X | XX | х | XX | X | XX | х | XX |
| | Mild | х | XX | Х | xx | Х | XX | х | XX | X | XX | Х | XX | X | XX | х | XX | X | XX | х | XX |
| | Moderate | х | XX | Х | XX | X | XX | х | XX | х | XX | X | XX | X | XX | х | XX | х | XX | Х | XX |
| | Severe | х | XX | Х | xx | Х | XX | х | xx | X | XX | X | XX | X | XX | х | xx | Х | XX | Х | XX |
| Headache | None | х | XX | Х | xx | Х | XX | х | xx | X | XX | X | XX | X | XX | х | xx | Х | XX | Х | XX |
| | Mild | х | XX | Х | XX | X | XX | х | XX | х | XX | X | XX | X | XX | х | XX | х | XX | Х | XX |
| | Moderate | х | XX | Х | XX | X | XX | х | XX | х | XX | X | XX | X | XX | х | XX | х | XX | Х | XX |
| | Severe | х | XX | Х | xx | Х | XX | х | xx | X | XX | X | XX | X | XX | х | xx | Х | XX | Х | XX |
| Nausea | None | Х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Mild | Х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Moderate | Х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Severe | х | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Any Local Symptom | None | х | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Mild | х | XX | Х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Moderate | х | XX | Х | xx | Х | XX | х | XX | X | XX | Х | XX | X | XX | х | XX | X | XX | х | XX |

| Symptom | Severity | Pre | -Vac | Pos | t-Vac | D | ay 1 | Da | y 2 | Da | ıy 3 | Da | y 4 | Da | ıy 5 | Da | ny 6 | Da | ay 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Severe | Х | XX | Х | XX | Х | XX | X | XX | х | XX | X | XX | Х | XX | х | XX | X | XX | Х | XX |
| Pain | None | Х | XX | х | XX | X | XX | Х | XX | х | XX | X | XX | Х | XX | Х | XX | X | XX | Х | XX |
| | Mild | Х | XX | х | XX | X | XX | Х | XX | х | XX | X | XX | Х | XX | Х | XX | X | XX | Х | XX |
| | Moderate | Х | XX | х | XX | X | XX | Х | XX | х | XX | X | XX | Х | XX | Х | XX | X | XX | Х | XX |
| | Severe | X | XX | Х | xx | Х | XX | X | xx | х | XX | X | XX | Х | XX | х | XX | X | XX | Х | XX |
| Tenderness | None | X | XX | Х | xx | Х | XX | X | xx | х | XX | X | XX | Х | XX | х | XX | X | XX | X | XX |
| | Mild | X | XX | Х | xx | Х | XX | X | xx | х | XX | X | XX | Х | XX | х | XX | X | XX | X | XX |
| | Moderate | X | XX | Х | xx | Х | XX | X | xx | х | XX | X | XX | Х | XX | х | XX | X | XX | X | XX |
| | Severe | X | XX | Х | xx | Х | XX | X | xx | х | XX | X | XX | Х | XX | х | XX | X | XX | X | XX |
| Pruritus | None | X | XX | Х | xx | Х | XX | X | xx | х | XX | X | XX | Х | XX | х | XX | X | XX | X | XX |
| | Mild | х | XX | Х | XX | X | XX | X | xx | х | xx | X | XX | Х | xx | х | XX | Х | XX | X | XX |
| | Moderate | х | XX | Х | XX | X | XX | X | xx | х | xx | X | XX | Х | xx | х | XX | Х | XX | Х | XX |
| | Severe | х | XX | Х | XX | X | XX | X | xx | х | xx | X | XX | Х | xx | х | XX | Х | XX | Х | XX |
| Ecchymosis | None | X | XX | Х | XX | X | XX | X | XX | х | XX | X | XX | X | XX | x | XX | X | XX | X | xx |
| | Mild | X | XX | Х | XX | X | XX | X | XX | х | XX | X | XX | X | XX | x | XX | X | XX | X | xx |
| | Moderate | X | XX | X | XX | X | XX | X | XX | х | XX | X | XX | X | XX | x | XX | X | XX | X | XX |
| | Severe | X | XX | X | XX | х | XX | X | XX | х | XX | X | XX | X | XX | x | XX | X | XX | X | XX |
| Ecchymosis (measurement) | None | X | XX | Х | XX | X | XX | X | XX | х | XX | X | XX | X | XX | x | XX | X | XX | X | xx |
| | Mild | X | XX | X | XX | х | XX | X | XX | Х | XX | X | XX | X | XX | х | XX | X | XX | X | XX |
| | Moderate | X | XX | Х | XX | X | XX | X | XX | х | XX | X | XX | X | XX | x | XX | X | XX | X | xx |
| | Severe | X | XX | Х | XX | X | XX | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | Х | XX |
| Erythema | None | X | XX | X | XX | X | XX | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | Х | XX |
| | Mild | X | XX | Х | XX | х | XX | X | XX | Х | XX | X | XX | X | XX | Х | XX | X | XX | х | XX |

| Symptom | Severity | Pre | -Vac | Pos | t-Vac | D | ay 1 | Da | y 2 | Da | ıy 3 | Da | ıy 4 | Da | ıy 5 | Da | ıy 6 | Da | ıy 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | X | XX | х | xx | Х | XX | x | xx | Х | xx | Х | XX | Х | XX | х | XX | Х | XX | X | xx |
| | Severe | X | XX | х | xx | X | XX | X | xx | X | XX | X | XX | Х | XX | Х | XX | х | XX | X | xx |
| Erythema (measurement) | None | X | XX | х | xx | X | XX | X | xx | X | XX | X | XX | Х | XX | Х | XX | х | XX | X | xx |
| | Mild | Х | XX | х | XX | Х | XX | X | xx | Х | xx | Х | XX | Х | XX | Х | XX | X | XX | Х | xx |
| | Moderate | X | XX | х | XX | х | XX | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |
| | Severe | Х | XX | х | XX | Х | XX | X | xx | Х | xx | Х | XX | Х | XX | Х | XX | X | XX | Х | xx |
| Induration/Swelling | None | X | XX | х | xx | Х | XX | x | xx | Х | xx | Х | XX | Х | XX | х | XX | Х | XX | X | xx |
| | Mild | Х | XX | х | XX | X | XX | X | xx | Х | xx | Х | XX | Х | XX | Х | XX | X | XX | Х | xx |
| | Moderate | X | XX | х | XX | Х | XX | X | xx | X | XX | Х | XX | х | XX | Х | XX | Х | XX | Х | xx |
| | Severe | X | XX | Х | XX | Х | XX | X | XX | X | XX | Х | XX | х | XX | х | XX | х | XX | Х | XX |
| Induration/Swelling (measurement) | None | X | XX | х | XX | Х | XX | X | xx | X | XX | Х | XX | х | XX | Х | XX | Х | XX | Х | xx |
| | Mild | X | XX | Х | XX | Х | XX | X | XX | X | XX | Х | XX | х | XX | х | XX | х | XX | Х | XX |
| | Moderate | X | XX | Х | xx | х | XX | Х | XX | X | XX | Х | XX | х | XX | X | XX | х | XX | Х | XX |
| | Severe | X | XX | х | XX | Х | XX | X | xx | X | XX | Х | XX | х | XX | Х | XX | х | XX | X | xx |

## [repeat for all study groups & All Subjects]

N = Number of subjects in the Safety Population who received any study vaccination; n = Number Severity is the maximum severity reported post dosing for each subject for each day.

[Implementation Note: The value considered for Day 8+ for each subject will be the maximum value reported at Day 8 or after for subjects with symptoms ongoing at Day 8.]

- Table 93: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, and Study Group (Safety Population) Post Study Vaccination 1
- Table 94: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, and Study Group (Safety Population) Post Study Vaccination 2

Table 95: Number and Percentage of Subjects Experiencing Solicited Systemic Events for Study Vaccination 1 Compared with Study Vaccination 2 by Study Group—Safety Population

| | | Subjects with No<br>Symptoms | Subjects with Mild or Greater<br>Symptoms | Total Number of Subjects<br>n (Percent)<br>[p-value*] |
|---|---|---|---|---|
| | | Study Vaccination 1 vs Stu | dy Vaccination 2 | |
| Group 1: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| 2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22) | Subjects with Mild or Greater Symptoms | x (%) | x (%) | x (%) |
| (N=X) | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 2: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| 2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121) | Subjects with Mild or Greater Symptoms | x (%) | x (%) | x (%) |
| (N=X) | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 3: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| 2013 3.75+AS03/<br>2017 15<br>(D1-D121) | Subjects with Mild or Greater Symptoms | x (%) | x (%) | x (%) |
| (N=X) | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 4: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| 2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22) | Subjects with Mild or Greater Symptoms | x (%) | x (%) | x (%) |
| (N=X) | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 5: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| | Subjects with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |

| | | Subjects with No<br>Symptoms | Subjects with Mild or Greater<br>Symptoms | Total Number of Subjects<br>n (Percent)<br>[p-value*] |
|---|---|---|---|---|
| 2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 6: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| 2017 3.75+AS03/<br>2017 15<br>(D1-D121) | Subjects with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| (N=X) | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| All Subjects | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| (N=X) | Subjects with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |

Note: Denominators for percentages are the number of subjects in the Safety Population who received both the first and second study vaccination. Subjects who did not receive both indicated vaccinations are not included in this table. [x] subjects did not receive the second study vaccination.

#### Table with similar format:

Table 96: Number and Percentage of Subjects Experiencing Solicited Local Events for Study Vaccination 1 Compared with Study Vaccination 2 by Study Group, Safety Population

<sup>\*</sup> P-value is calculated from McNemar's test for each study group.

#### 14.3.1.2 Unsolicited Adverse Events

Table 97: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Study Group, Safety Population\*

| MedDRA® System<br>Organ Class | MedDRA® Preferred<br>Term | 3.75<br>3.7<br>(D | roup 1<br>2013<br>5+AS03/<br>2017<br>5+AS03<br>1-D22)<br>N=X) | 3.7<br>(D | 2013<br>5+AS03/<br>2017<br>75+AS03<br>1-D121)<br>(N=X) | 3.7<br>2<br>(D | eroup 3<br>2013<br>5+AS03/<br>017 15<br>1-D121)<br>(N=X) | 3.7<br>(I | 75+AS03/<br>2017<br>75+AS03/<br>2017<br>75+AS03<br>201-D22)<br>(N=X) | 3.7:<br>3.7<br>(D | roup 5<br>2017<br>5+AS03/<br>2017<br>5+AS03<br>1-D121)<br>(N=X) | 3.7<br>2<br>(D | 2017<br>5+AS03/<br>017 15<br>1-D121)<br>(N=X) | | Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) |
| Any SOC | Any PT | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| [SOC 1] | Any PT | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) |
| | [PT 1] | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| | [PT 2] | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| [SOC 2] | Any PT | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| | [PT 1] | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) |
| | [PT 2] | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |

N = number of subjects in the Safety Population who received any study vaccination.

This table presents number and percentage of subjects. A subject is only counted once per PT.

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row should be omitted.]

Table 98: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship, and Study Group, Safety Population

| Study Group | MedDRA® System<br>Organ Class | MedDRA® Preferred Term | | ny<br>dence | | | Severi | ty [1] | | | | ationshi<br>Vaccina | | dy |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | N | Iild | Mode | erate | Se | vere | Not Ro | elated | Rela | ated |
| | | | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1: | Any SOC | Any PT | х | XX | Х | xx | Х | xx | х | xx | Х | XX | X | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | X | XX | X | XX | X | XX | х | XX | X | XX | X | XX |
| (D1-D22) | | [PT 1] | X | XX | Х | XX | х | XX | х | XX | X | XX | X | XX |
| (N=X) | | [PT 2] | х | XX | Х | XX | Х | XX | х | XX | Х | XX | X | XX |
| | [SOC 2] | Any PT | x | XX | Х | XX | Х | XX | x | xx | X | XX | X | XX |
| | | [PT 1] | х | XX | Х | XX | Х | XX | х | XX | Х | XX | X | XX |
| | | [PT 2] | х | xx | X | xx | х | xx | х | xx | Х | XX | х | xx |
| Group 2: | Any SOC | Any PT | х | XX | Х | XX | X | XX | х | XX | Х | XX | X | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | х | xx | X | xx | х | xx | х | xx | Х | XX | х | xx |
| (D1-D121) | | [PT 1] | х | xx | X | xx | х | xx | х | xx | Х | XX | х | xx |
| (N=X) | | [PT 2] | х | XX | Х | XX | Х | XX | х | XX | Х | XX | X | XX |
| | [SOC 2] | Any PT | х | xx | X | xx | х | xx | х | xx | Х | XX | х | xx |
| | | [PT 1] | х | xx | X | xx | х | xx | х | xx | Х | XX | х | xx |
| | | [PT 2] | х | XX | Х | XX | Х | XX | х | XX | Х | XX | X | XX |
| Group 3: | Any SOC | Any PT | х | xx | X | xx | х | XX | х | xx | Х | XX | х | xx |
| 2013 3.75+AS03/<br>2017 15 | [SOC 1] | Any PT | x | XX | х | xx | х | xx | Х | xx | х | XX | X | xx |
| (D1-D121) | | [PT 1] | x | XX | х | xx | х | xx | Х | xx | Х | XX | х | xx |
| (N=X) | | [PT 2] | х | XX | Х | xx | Х | xx | х | xx | Х | XX | X | XX |
| | [SOC 2] | Any PT | x | XX | Х | xx | Х | XX | х | xx | Х | XX | X | XX |

| | | | | 1 | | 1 | ı | | 1 | ı | I | 1 | 1 | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | [PT 1] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | | [PT 2] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Group 4: | Any SOC | Any PT | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | x | xx | X | XX | X | XX | X | XX | X | XX | X | XX |
| (D1-D22)<br>(N=X) | | [PT 1] | X | XX | X | XX | X | XX | x | XX | X | XX | X | XX |
| (N-A) | | [PT 2] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | [SOC 2] | Any PT | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | | [PT 1] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | | [PT 2] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Group 5: | Any SOC | Any PT | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | Х | XX | X | XX | X | XX | х | XX | Х | XX | Х | XX |
| (D1-D121) | | [PT 1] | Х | XX | X | XX | X | XX | х | XX | Х | XX | Х | XX |
| (N=X) | | [PT 2] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | [SOC 2] | Any PT | Х | XX | X | XX | X | XX | х | XX | Х | XX | Х | XX |
| | | [PT 1] | х | xx | Х | xx | х | xx | х | xx | Х | XX | Х | XX |
| | | [PT 2] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| Group 6: | Any SOC | Any PT | Х | xx | Х | XX | X | XX | х | xx | X | XX | X | xx |
| 2017 3.75+AS03/<br>2017 15 | [SOC 1] | Any PT | X | XX | X | XX | Х | XX | x | XX | Х | XX | X | XX |
| (D1-D121) | | [PT 1] | X | XX | X | XX | Х | XX | x | XX | Х | XX | X | XX |
| (N=X) | | [PT 2] | X | XX | X | XX | Х | XX | x | XX | Х | XX | X | XX |
| | [SOC 2] | Any PT | Х | XX | X | XX | Х | XX | х | XX | Х | XX | х | XX |
| | | [PT 1] | X | XX | X | XX | Х | XX | x | XX | Х | XX | X | XX |
| | | [PT 2] | х | XX | X | XX | X | XX | X | XX | х | XX | х | XX |
| All Subjects | Any SOC | Any PT | Х | XX | Х | XX | X | xx | х | xx | X | XX | Х | XX |
| (N=X) | [SOC 1] | Any PT | х | XX | Х | XX | X | xx | х | xx | х | XX | Х | XX |

| | [PT 1] | X | XX | X | XX | X | xx | X | xx | X | XX | X | xx |
|---------|--------|---|----|---|----|---|----|---|----|---|----|---|----|
| | [PT 2] | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |
| [SOC 2] | Any PT | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |
| | [PT 1] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | [PT 2] | X | XX | X | XX | X | XX | x | XX | X | XX | X | xx |

N = Number of subjects in the Safety Population.

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row will be omitted. Only the SOC/PT with >= 1 event reported will be shown for each group.]

Table with similar format:

Table 99: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events within 21 Days of Study Vaccination by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship, and Study Group, Safety Population

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row will be omitted. Only the SOC/PT with >= 1 event reported will be shown for each group. Events through 'Day 22' include events through the study visit planned for 21 days post the relevant vaccination. If that visit is missed, then a cutoff of exactly 21 days post vaccination will be used.]

<sup>[1]</sup> For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

<sup>[2]</sup> For relationship, a subject is only counted once per preferred term and is summarized according to their closest relationship.

Table 100 Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Study Group, Safety Population

| Study Group | MedDRA® System Organ | MedDRA® Preferred | Any In | cidence | | | Sever | ity [1] | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Class | Term | | | M | ild | Mod | erate | Sev | vere |
| | | | n | % | n | % | n | % | n | % |
| Group 1: | Any SOC | Any PT | x | xx | Х | XX | Х | XX | х | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | x | xx | Х | XX | Х | XX | х | XX |
| (D1-D22) | | [PT 1] | х | xx | Х | XX | Х | XX | Х | XX |
| (N=X) | | [PT 2] | х | xx | Х | XX | Х | XX | Х | XX |
| | [SOC 2] | Any PT | х | xx | Х | XX | Х | XX | Х | XX |
| | | [PT 1] | х | xx | Х | XX | Х | XX | Х | XX |
| | | [PT 2] | х | xx | Х | XX | Х | XX | Х | XX |
| Group 2: | Any SOC | Any PT | х | xx | Х | XX | Х | XX | Х | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | Х | xx | X | XX | X | XX | X | XX |
| (D1-D121) | | [PT 1] | Х | xx | X | XX | X | XX | X | XX |
| (N=X) | | [PT 2] | Х | xx | X | XX | X | XX | X | XX |
| | [SOC 2] | Any PT | X | xx | X | XX | X | XX | X | XX |
| | | [PT 1] | Х | xx | X | XX | X | XX | X | XX |
| | | [PT 2] | Х | xx | X | XX | X | XX | X | XX |
| Group 3: | Any SOC | Any PT | х | xx | X | XX | X | XX | X | XX |
| 2013 3.75+AS03/<br>2017 15 | [SOC 1] | Any PT | Х | xx | X | XX | X | XX | X | XX |
| (D1-D121) | | [PT 1] | х | xx | Х | XX | х | XX | Х | XX |
| (N=X) | | [PT 2] | Х | xx | Х | XX | X | XX | X | XX |
| | [SOC 2] | Any PT | х | xx | Х | XX | х | XX | Х | XX |
| | | [PT 1] | x | XX | х | XX | Х | XX | Х | XX |

| | | | | I | | | | | l | ı |
|---|---|---|---|---|---|---|---|---|---|---|
| | | [PT 2] | X | XX | X | XX | X | XX | X | XX |
| Group 4: | Any SOC | Any PT | X | XX | X | XX | X | XX | X | XX |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | x | xx | X | XX | X | XX | X | XX |
| (D1-D22)<br>(N=X) | | [PT 1] | X | xx | X | XX | X | XX | X | XX |
| (N-A) | | [PT 2] | x | XX | X | XX | X | XX | X | XX |
| | [SOC 2] | Any PT | x | XX | X | XX | X | XX | X | XX |
| | | [PT 1] | X | XX | X | XX | X | XX | X | XX |
| | | [PT 2] | x | XX | X | XX | X | XX | X | XX |
| Group 5: | Any SOC | Any PT | x | XX | X | XX | X | XX | X | XX |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | [SOC 1] | Any PT | x | XX | X | XX | X | XX | X | XX |
| (D1-D121) | | [PT 1] | x | XX | X | XX | X | XX | X | XX |
| (N=X) | | [PT 2] | x | xx | X | XX | X | XX | X | XX |
| | [SOC 2] | Any PT | x | XX | X | XX | X | XX | X | XX |
| | | [PT 1] | x | xx | X | XX | X | XX | Х | XX |
| | | [PT 2] | x | xx | X | XX | X | XX | X | XX |
| Group 6: | Any SOC | Any PT | x | xx | X | XX | X | XX | X | XX |
| 2017 3.75+AS03/<br>2017 15 | [SOC 1] | Any PT | х | xx | Х | XX | X | XX | Х | XX |
| (D1-D121) | | [PT 1] | х | xx | Х | XX | X | XX | Х | XX |
| (N=X) | | [PT 2] | x | xx | X | XX | X | XX | X | XX |
| | [SOC 2] | Any PT | х | xx | Х | XX | X | XX | Х | XX |
| | | [PT 1] | х | xx | Х | XX | X | XX | Х | XX |
| | | [PT 2] | х | xx | X | XX | X | XX | Х | XX |
| All Subjects | Any SOC | Any PT | X | xx | х | XX | X | XX | х | XX |
| (N=X) | [SOC 1] | Any PT | X | xx | Х | XX | X | XX | Х | XX |
| | | [PT 1] | х | XX | X | XX | X | XX | Х | XX |

| | [PT 2] | Х | XX | X | XX | X | XX | X | XX |
|---------|--------|---|----|---|----|---|----|---|----|
| [SOC 2] | Any PT | Х | XX | X | XX | X | XX | X | xx |
| | [PT 1] | Х | XX | X | XX | X | XX | X | XX |
| | [PT 2] | Х | XX | X | XX | X | XX | X | xx |

N = Number of subjects in the Safety Population. [1] For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row will be omitted. Only the SOC/PT with >= 1 event reported will be shown for each group.]

Table with similar format:

Table 101: Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Study Group, Safety Population

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row will be omitted. Only the SOC/PT with >= 1 event reported will be shown for each group. Events through 'Day 22' include events through the study visit planned for 21 days post the relevant vaccination. If that visit is missed, then a cutoff of exactly 21 days post vaccination will be used.]

**Table 102:** Number and Percentage of Subjects Experiencing Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA® System Organ Class and Preferred Term, Day Post Study Vaccination, and Study Group, Safety Population

| MedDRA® System Organ<br>Class | MedDRA® Preferred<br>Term | | P | ost Vac | cinatior | n 1 | | | Po | ost Vac | cination | 2 | | | t Any<br>ination |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day | y 1-8 | Day | 9-22 | Day | 1-22 | Day | y 1-8 | Day | 9-22 | Day | 1-22 | Day | y 1-22 |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Group | 1: 2013 | 3.75+A | AS03/ 20 | 17 3.75 | +AS03 | (D1-D2 | 2) (N=X | () | | | | | | |
| Any SOC | Any PT | X | XX | X | xx | х | xx | X | XX | X | XX | X | XX | x | XX |
| [SOC 1] | Any PT | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | |
| | 1 | [Repe | at for a | ll study | groups | & All S | ubjects | ] | | | | 1 | | | .1 |
| N = Number of subjects in the S | afety Population. This table pr | esents n | umber a | and perc | entage c | of subject | ets. For 6 | each tim | e period | , a subj | ect is on | ly count | ted once | per PT. | |

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row will be omitted. Only the SOC/PT with >= 1 event reported will be shown for

each group. Events through 'Day 22' include events through the study visit planned for 21 days post the relevant vaccination. If that visit is missed, then a cutoff of exactly 21 days post vaccination will be used.]

Table 103: Number and Percentage of Subjects Experiencing Non-Serious, Related Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA® System Organ Class and Preferred Term, Vaccination and Study Group, Safety Population

| MedDRA® System Organ<br>Class | MedDRA® Preferred<br>Term | | Post Vaccination 1 | | | | | | | Post Vaccination 2 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day 1-8 | | Day 9-22 | | Day 1-22 | | Day 1-8 | | Day 9-22 | | Day 1-22 | | Day 1-22 | |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Group | 1: 2013 | 3.75+A | S03/ 20 | 17 3.75 | +AS03 | (D1-D2 | 2) (N=X | () | | | | | | |
| Any SOC | Any PT | х | xx | х | XX | X | XX | х | xx | X | XX | X | XX | X | XX |
| [SOC 1] | Any PT | Х | XX | х | XX | X | xx | Х | XX | Х | xx | Х | XX | Х | XX |
| | [PT 1] | Х | XX | х | XX | X | xx | Х | XX | Х | xx | Х | XX | Х | XX |
| | [PT 2] | Х | XX | Х | XX | X | XX | Х | XX | X | XX | Х | XX | Х | XX |
| [SOC 2] | Any PT | х | XX | х | XX | Х | XX | х | xx | X | XX | Х | XX | Х | XX |
| | [PT 1] | Х | XX | Х | XX | X | XX | Х | XX | X | XX | Х | XX | Х | XX |
| | [PT 2] | Х | XX | х | XX | X | XX | Х | XX | X | XX | х | XX | х | XX |
| | | [Repe | at for al | l study | groups | & All S | ubjects | ] | • | | • | | • | ı | |

N = Number of subjects in the Safety Population. This table presents number and percentage of subjects. For each time period, a subject is only counted once per PT.

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row will be omitted. Only the SOC/PT with >= 1 event reported will be shown for each group. Events through 'Day 22' include events through the study visit planned for 21 days post the relevant vaccination. If that visit is missed, then a cutoff of exactly 21 days post vaccination will be used.]

Table 104: Number of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Day Post Study Vaccination, and Study Group, Safety Population

| MedDRA® System Organ | MedDRA® Preferred | | | ] | Number of Eve | ents | | |
|---|---|---|---|---|---|---|---|---|
| Class | Term | Po | ost Vaccination | 1 | P | ost Vaccination | 2 | Post Any<br>Vaccination |
| | | Day 1-8 | Day 1-8 Day 9-22 Day 1-22 | | Day 1-8 Day 9-22 Day 1-22 | | | Day 1-22 |
| | Group | 1: 2013 3.75+A | AS03/ 2017 3.75 | +AS03 (D1-D2 | 2) (N=X) | • | | |
| Any SOC | Any PT | X | X | X | X | X | X | X |
| [SOC 1] | Any PT | X | X | X | X | X | X | X |
| | [PT 1] | X | X | X | X | X | X | X |
| | [PT 2] | X | X | X | X | X | X | X |
| [SOC 2] | Any PT | X | х | X | X | Х | X | X |
| | [PT 1] | X | х | X | X | Х | X | X |
| | [PT 2] | X | X | X | X | X | X | X |
| | | [Repeat for al | ll study groups | & All Subjects | ] | | | |
| N = Number of subjects in the Sa | fety Population. This table pr | esents number of | of events; a subj | ect may be coun | ited multiple tin | nes. | | |

[Implementation Note: If an SOC has only one PT reported, the 'Any PT' row will be omitted. Only the SOC/PT with >= 1 event reported will be shown for each group. Events through 'Day 22' include events through the study visit planned for 21 days post the relevant vaccination. If that visit is missed, then a cutoff of exactly 21 days post vaccination will be used.]

Table with similar format:

Table 105: Number of Non-Serious, Related, Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Day Post Study Vaccination, and Study Group, Safety Population

## 14.3.2 Listing of Serious and Significant Adverse Events

**Table 106:** Listing of Serious Adverse Events – Safety Population \*

| Adverse<br>Event | Associated<br>with Vac # | # of Days Post Associated Vac (Duration) | # of Days Post Vac the Event Became Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Vaccination | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Vaccination | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA®<br>Sytem<br>Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | : , Study Grou | p: , AE Numb | er: | | | | | | • | | | |
| Comments | s: | | | | | | | | | | | |
| Subject ID | :, Study Grou | p: , AE Numbe | r: | | | | | | | | | |
| Comments | S: | ı | 1 | | • | 1 | | ı | 1 | 1 | | |

## **Table 107:** Listing of Medically Attended Adverse Events – Safety Population

[Implementation Note: If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon.]

| Adverse<br>Event | Associated with Vac # | # of Days<br>Post<br>Associated<br>Vac<br>(Duration) | SAE?<br>Severity | Relationship<br>to Study<br>Vaccination | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Vaccination | Subject<br>Discontinued<br>Due to AE | Outcome | PIMMC?<br>NOCMC? | MedDRA®<br>System<br>Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject II | ): , Study Gro | up: , AE Nun | nber: | | | | | | | | |
| | | | SAE: No<br>Mild | | | | | | | | |
| Comment | s: | | | | | | | | | | |
| Subject II | ): , Study Gro | up: , AE Nun | nber: | | | | | | | | |
| Comment | s: | | | | | | | | | | |

Tables with similar format:

**Table 108:** Listing of Potentially Immune Mediated Medical Conditions

[Implementation Note: Update column 'PIMMC? NOCMC?' to 'MAAE? NOCMC?']

**Table 109: Listing of New Onset Chronic Medical Conditions** 

[Implementation Note: Update column 'PIMMC? NOCMC?' to 'MAAE? PIMMC?']

Table 110: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

[Implementation Note: Update column 'MAAE? PIMMC? NOCMC?' to 'MAAE? PIMMC?']

## 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

### 14.3.4 Displays of Laboratory Results

## 14.3.4.1 Displays of Chemistry Results

Table 111: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – All Chemistry Parameters – Safety Population

| Study Group | Study Day | N* | N | one | | ild/<br>ide 1 | | lerate/<br>ade 2 | | vere/<br>ade 3 | M | issing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| Group 1: | Baseline | х | х | XX | X | XX | X | XX | х | xx | Х | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22)<br>(N=X) | Day 8 post Vac 1 | х | х | XX | X | XX | X | XX | X | xx | X | XX |
| | Pre-Vac 2 (Day 22) | х | X | XX | X | XX | X | XX | X | xx | X | XX |
| | Day 8 post Vac 2 | х | X | XX | X | XX | X | XX | X | xx | X | XX |
| | Max Severity Post Baseline | х | X | XX | X | XX | X | XX | X | xx | X | XX |
| Group 2: | Baseline | х | X | XX | X | XX | X | XX | X | xx | X | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | х | XX | X | XX | X | XX | х | xx | Х | xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | X | XX | X | XX | X | XX | X | xx | X | XX |
| (N=X) | Day 8 post Vac 2 | х | х | XX | X | XX | X | XX | х | xx | Х | xx |
| | Max Severity Post Baseline | х | х | XX | X | XX | X | XX | х | xx | Х | xx |
| Group 3: | Baseline | х | х | XX | Х | XX | Х | XX | х | xx | Х | XX |
| 2013 3.75+AS03/<br>2017 15 | Day 8 post Vac 1 | x | х | XX | Х | XX | X | XX | х | xx | Х | xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | x | х | XX | Х | XX | X | XX | х | xx | Х | xx |
| (N=X) | Day 8 post Vac 2 | x | х | XX | Х | XX | X | XX | х | xx | Х | xx |
| | Max Severity Post Baseline | x | х | XX | Х | XX | х | XX | х | xx | х | xx |
| Group 4: | Baseline | x | х | XX | X | XX | х | XX | х | xx | х | xx |
| 2017 3.75+AS03/ | Day 8 post Vac 1 | x | х | XX | X | XX | х | XX | х | xx | х | xx |

| Study Group | Study Day | N* | N | one | | ild/<br>ide 1 | | derate/<br>ade 2 | | vere/<br>ade 3 | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| 2017 3.75+AS03<br>(D1-D22) (N=X) | Pre-Vac 2<br>(Day 22) | X | Х | xx | х | xx | Х | xx | х | XX | х | XX |
| | Day 8 post Vac 2 | х | X | XX | X | XX | X | XX | X | xx | X | XX |
| | Max Severity Post Baseline | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| Group 5 | Baseline | х | х | XX | X | XX | х | XX | Х | xx | X | xx |
| 2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121) | Day 8 post Vac 1 | х | х | XX | X | XX | х | XX | х | xx | х | xx |
| | Pre-Vac 2 (Day 121) | х | х | XX | X | XX | х | XX | х | xx | х | xx |
| (N=X) | Day 8 post Vac 2 | х | х | XX | X | XX | х | XX | х | xx | х | xx |
| | Max Severity Post Baseline | х | х | XX | X | XX | х | XX | х | xx | х | xx |
| Group 6: | Baseline | х | X | XX | X | XX | X | XX | X | xx | X | xx |
| 2017 3.75+AS03/<br>2017 15 | Day 8 post Vac 1 | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | х | XX | X | XX | х | XX | Х | xx | X | xx |
| (N=X) | Day 8 post Vac 2 | х | х | XX | X | XX | х | XX | Х | xx | X | xx |
| | Max Severity Post Baseline | х | х | XX | X | XX | х | XX | Х | xx | X | xx |
| All Subjects | Baseline | х | х | XX | Х | XX | х | XX | х | XX | х | xx |
| (N=X) | Day 8 post Vac 1 | х | х | XX | X | XX | х | XX | X | XX | х | xx |
| | Pre-Vac 2 | х | х | XX | X | XX | Х | XX | х | XX | х | xx |
| | Day 8 post Vac 2 | x | х | XX | X | XX | Х | XX | X | XX | X | xx |
| | Max Severity Post Baseline | x | х | XX | X | XX | х | XX | х | XX | X | xx |

The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N=Number of subjects in the Safety Population; N\*=Number of subjects who completed the indicated visit.

[Implementation Note: A subject should be counted within N\* only if they completed the study visit in-person (i.e. not a phone visit).]

- Table 112: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) Alanine aminotransferase (ALT)
- Table 113: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) Total Bilirubin
- Table 114: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) Creatinine

Table 115: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Alanine Aminotransferase (ALT)

| Study Group | Study Day | N* | | Va | lue | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Mean | Standard<br>Deviation | Median | Min, Max | Mean | Standard<br>Deviation | Median | Min, Max |
| Group 1: | Baseline | х | xx.x | xx.x | xx | xx, xx | NA | NA | NA | NA |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| (D1-D22)<br>(N=X) | Pre-Vac 2 (Day 22) | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| Group 2: | Baseline | х | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |
| (D1-D121)<br>(N=X) | Pre-Vac 2 (Day 121) | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |
| | Day 8 post Vac 2 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| Group 3: | Baseline | х | xx.x | XX.X | XX | xx, xx | NA | NA | NA | NA |
| 2013 3.75+AS03/<br>2017 15 | Day 8 post Vac 1 | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | xx | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| Group 4: | Baseline | х | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| (D1-D22) | Pre-Vac 2 (Day 22) | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| Group 5 | Baseline | x | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA |
| 2017 3.75+AS03/ | Day 8 post Vac 1 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | XX | xx, xx |
| 2017 3.75+AS03<br>(D1-D121) | Pre-Vac 2 (Day 121) | x | xx.x | XX.X | xx | xx, xx | XX.X | xx.x | XX | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |

| Study Group | Study Day | N* | | Va | lue | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Mean | Standard<br>Deviation | Median | Min, Max | Mean | Standard<br>Deviation | Median | Min, Max |
| Group 6:<br>2017 3.75+AS03/<br>2017 15 | Baseline | x | XX.X | xx.x | xx | xx, xx | NA | NA | NA | NA |
| | Day 8 post Vac 1 | x | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | xx | xx, xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | x | xx.x | XX.X | xx | xx, xx | xx.x | XX.X | xx | xx, xx |
| (N=X) | Day 8 post Vac 2 | x | xx.x | XX.X | xx | xx, xx | xx.x | XX.X | xx | xx, xx |
| All Subjects | Baseline | x | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA |
| (N=X) | Day 8 post Vac 1 | X | xx.x | XX.X | xx | xx, xx | xx.x | XX.X | xx | xx, xx |
| | Pre-Vac 2 | x | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |
| | Day 8 post Vac 2 | x | XX.X | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |

Table 116: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Total Bilirubin

Table 117: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Creatinine
### 14.3.4.1 Displays of Hematology Results

Table 118: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – All Hematology Parameters

| Study Group | Study Day | N* | N | one | | ild/<br>ide 1 | | lerate/<br>ade 2 | | vere/<br>ade 3 | M | issing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| Group 1: | Baseline | х | х | XX | X | XX | X | XX | X | xx | X | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| (D1-D22) | Pre-Vac 2 (Day 22) | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| (N=X) | Day 8 post Vac 2 | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| | Max Severity Post Baseline | х | х | xx | Х | XX | Х | XX | х | xx | Х | xx |
| Group 2: | Baseline | х | Х | XX | X | XX | X | XX | Х | xx | Х | xx |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | Х | XX | X | XX | X | XX | Х | xx | Х | xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | х | xx | Х | XX | X | XX | х | xx | Х | xx |
| (N=X) | Day 8 post Vac 2 | х | х | xx | Х | XX | X | XX | х | xx | Х | xx |
| | Max Severity Post Baseline | х | х | XX | Х | XX | X | XX | х | xx | Х | xx |
| Group 3: | Baseline | х | х | xx | Х | XX | Х | XX | х | xx | Х | xx |
| 2013 3.75+AS03/<br>2017 15 | Day 8 post Vac 1 | х | х | xx | Х | XX | X | XX | х | xx | Х | xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | х | xx | Х | XX | X | XX | х | xx | Х | xx |
| (N=X) | Day 8 post Vac 2 | х | Х | XX | X | XX | X | XX | Х | xx | Х | xx |
| | Max Severity Post Baseline | х | Х | XX | X | XX | X | XX | х | xx | Х | xx |
| Group 4: | Baseline | х | х | xx | Х | XX | х | XX | х | xx | х | xx |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | х | XX | Х | XX | Х | XX | х | xx | х | xx |
| (D1-D22) (N=X) | Pre-Vac 2 (Day 22) | х | х | XX | X | XX | Х | XX | Х | xx | X | xx |
| | Day 8 post Vac 2 | х | х | XX | Х | XX | Х | XX | х | xx | х | xx |

| Study Group | Study Day | N* | N | one | | ild/<br>ide 1 | | lerate/<br>ade 2 | | vere/<br>ade 3 | Mi | issing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| | Max Severity Post Baseline | х | х | XX | Х | XX | X | XX | Х | xx | Х | XX |
| Group 5 | Baseline | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| 2017 3.75+AS03/ | Day 8 post Vac 1 | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| 2017 3.75+AS03<br>(D1-D121) | Pre-Vac 2 (Day 121) | х | х | XX | X | XX | X | XX | X | xx | X | xx |
| (N=X) | Day 8 post Vac 2 | х | х | XX | Х | XX | Х | XX | х | xx | х | xx |
| | Max Severity Post Baseline | х | х | XX | Х | XX | X | XX | х | xx | X | xx |
| Group 6: | Baseline | х | х | XX | Х | XX | X | XX | Х | xx | Х | XX |
| 2017 3.75+AS03/<br>2017 15 | Day 8 post Vac 1 | х | х | XX | Х | XX | Х | XX | х | xx | х | xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | х | XX | Х | XX | Х | XX | х | xx | X | xx |
| (N=X) | Day 8 post Vac 2 | х | х | XX | Х | XX | Х | XX | х | xx | х | xx |
| | Max Severity Post Baseline | х | х | XX | Х | XX | Х | XX | х | xx | X | xx |
| All Subjects | Baseline | х | х | XX | Х | XX | Х | XX | х | xx | X | xx |
| (N=X) | Day 8 post Vac 1 | х | х | XX | Х | XX | X | XX | х | xx | х | xx |
| | Pre-Vac 2 | x | х | xx | х | XX | х | XX | х | xx | х | xx |
| | Day 8 post Vac 2 | х | х | XX | X | XX | Х | XX | х | xx | X | xx |
| | Max Severity Post Baseline | х | х | XX | Х | XX | X | XX | х | xx | х | xx |

The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N=Number of subjects in the Safety Population; N\*=Number of subjects who completed the indicated visit.

[Implementation Note: A subject should be counted within N\* only if they completed the study visit in-person (i.e. not a phone visit).]

Table with similar format:

Table 119: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – Hemoglobin

Table 120: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – White Blood Cells

| Study Group | Study Day | N* | No | ne | | Mild / 0 | Grade 1 | | M | loderate | / Grade | e 2 | S | evere / | Grade | 3 | Missi | ng |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | L | ow | Hi | igh | Le | ow | Hi | gh | Le | ow | Н | igh | | |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1: | Baseline | Х | X | XX | Х | XX | X | XX | X | XX | х | XX | Х | XX | X | XX | х | xx |
| 2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22) | Day 8 post Vac | х | X | xx | х | xx | Х | xx | Х | xx | х | XX | Х | XX | Х | xx | X | XX |
| (N=X) | Pre-Vac 2 (Day 22) | х | X | xx | х | xx | X | xx | Х | xx | х | XX | Х | XX | Х | xx | X | XX |
| | Day 8 post Vac 2 | х | Х | XX | х | xx | Х | xx | Х | xx | Х | XX | Х | XX | Х | XX | Х | XX |
| | Max Severity<br>Post Baseline | х | х | xx | х | xx | х | xx | Х | xx | х | XX | Х | xx | Х | xx | Х | XX |
| Group 2: | Baseline | X | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121) | Day 8 post Vac | х | Х | XX | х | xx | Х | xx | Х | xx | Х | XX | Х | XX | Х | XX | Х | XX |
| (N=X) | Pre-Vac 2 (Day 121) | х | х | xx | х | xx | х | xx | Х | xx | х | XX | Х | xx | X | XX | X | XX |
| | Day 8 post Vac<br>2 | х | х | xx | х | xx | х | xx | Х | xx | х | XX | Х | xx | Х | xx | Х | XX |
| | Max Severity<br>Post Baseline | х | х | xx | х | xx | х | xx | Х | xx | х | XX | Х | xx | Х | xx | X | XX |
| Group 3: | Baseline | X | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| 2013 3.75+AS03/<br>2017 15<br>(D1-D121) | Day 8 post Vac | х | х | xx | х | xx | х | xx | Х | xx | х | XX | Х | xx | х | XX | Х | XX |
| (N=X) | Pre-Vac 2 (Day 121) | х | х | xx | Х | XX | х | xx | Х | xx | х | xx | х | xx | Х | xx | х | xx |

| Study Group | Study Day | N* | No | one | | Mild / | Grade 1 | | M | loderate | / Grad | e 2 | S | evere / | Grade | 3 | Missi | ing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | L | ow | Н | igh | L | ow | H | igh | Le | )W | Н | igh | | |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Day 8 post Vac 2 | х | Х | xx | х | xx | х | xx | Х | xx | х | xx | X | XX | X | xx | X | xx |
| | Max Severity<br>Post Baseline | х | Х | xx | х | xx | х | xx | Х | xx | х | XX | Х | xx | Х | xx | Х | XX |
| Group 4: | Baseline | X | X | XX | х | XX | X | XX | X | XX | х | XX | X | XX | х | XX | X | XX |
| 2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D22) | Day 8 post Vac | х | х | xx | х | xx | х | xx | Х | xx | х | xx | Х | XX | Х | xx | Х | XX |
| (N=X) | Pre-Vac 2 (Day 22) | х | х | xx | х | xx | X | xx | Х | xx | х | xx | Х | XX | X | xx | X | XX |
| | Day 8 post Vac 2 | х | х | xx | х | xx | X | xx | Х | xx | х | xx | Х | XX | X | xx | X | XX |
| | Max Severity<br>Post Baseline | х | X | xx | х | xx | х | xx | Х | xx | х | XX | Х | XX | X | xx | X | XX |
| Group 5 | Baseline | X | X | XX | х | XX | X | XX | X | XX | х | XX | X | XX | х | XX | X | XX |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac | х | Х | XX | х | XX | Х | XX | х | xx | Х | XX | х | xx | х | xx | Х | xx |
| (D1-D121)<br>(N=X) | Pre-Vac 2 (Day<br>121) | Х | X | xx | х | xx | Х | xx | Х | xx | Х | XX | Х | XX | Х | xx | Х | XX |
| | Day 8 post Vac 2 | х | Х | xx | х | xx | х | xx | X | xx | х | xx | X | XX | X | xx | X | XX |
| | Max Severity<br>Post Baseline | х | X | xx | х | xx | х | xx | Х | xx | х | XX | Х | XX | X | xx | X | XX |
| Group 6: | Baseline | х | X | XX | х | XX | Х | XX | X | XX | х | XX | X | XX | х | XX | х | xx |
| 2017 3.75+AS03/<br>2017 15<br>(D1-D121) | Day 8 post Vac | х | х | xx | х | xx | х | xx | х | xx | х | xx | Х | xx | Х | xx | Х | xx |
| (N=X) | Pre-Vac 2 (Day 121) | х | х | XX | х | xx | х | xx | х | xx | х | xx | х | xx | X | XX | X | xx |

| Study Group | Study Day | N* | No | ne | | Mild / C | Grade 1 | | M | oderate | / Grade | e 2 | S | evere / | Grade | 3 | Missi | ng |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Lo | OW | Hi | igh | Le | OW | Hi | gh | Le | OW | Н | igh | | |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Day 8 post Vac 2 | х | X | XX | X | XX | X | XX | Х | XX | X | XX | X | XX | X | XX | х | XX |
| | Max Severity<br>Post Baseline | Х | Х | XX | Х | XX | X | XX | Х | xx | Х | XX | Х | XX | Х | XX | X | XX |
| All Subjects | Baseline | Х | X | XX | X | xx | X | xx | X | XX | х | XX | X | XX | х | XX | х | xx |
| (N=X) | Day 8 post Vac | Х | X | XX | X | XX | X | XX | Х | XX | X | XX | X | XX | X | XX | Х | XX |
| | Pre-Vac 2 | Х | X | XX | X | xx | X | xx | X | XX | х | XX | X | XX | х | XX | х | xx |
| | Day 8 post Vac 2 | Х | Х | XX | Х | XX | Х | XX | Х | xx | Х | XX | Х | XX | Х | XX | X | XX |
| | Max Severity<br>Post Baseline | х | Х | XX | Х | XX | х | XX | Х | xx | х | xx | Х | xx | Х | XX | X | XX |

The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N = Number of subjects in the Safety Population;  $N^* = N$  the number of subjects that completed the indicated visit.

Table with similar format:

Table 121: Laboratory Results by Parameter, Maximum Severity, Study Day, and Study Group (Safety Population) – Platelets

Table 122: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Hemoglobin

| Study Group | Study Day | N* | | Va | lue | | | Change | e from Basel | ine |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Mean | Standard<br>Deviation | Median | Min, Max | Mean | Standard<br>Deviation | Median | Min, Max |
| Group 1: | Baseline | x | XX.X | XX.X | XX | xx, xx | NA | NA | NA | NA |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |
| (D1-D22) | Pre-Vac 2 (Day 22) | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| Group 2: | Baseline | х | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| Group 3: | Baseline | х | xx.x | XX.X | XX | xx, xx | NA | NA | NA | NA |
| 2013 3.75+AS03/<br>2017 15 | Day 8 post Vac 1 | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | xx | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| Group 4: | Baseline | х | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | Day 8 post Vac 1 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | xx | xx, xx |
| (D1-D22) | Pre-Vac 2 (Day 22) | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | XX | xx, xx |
| Group 5 | Baseline | х | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA |
| 2017 3.75+AS03/ | Day 8 post Vac 1 | х | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | XX | xx, xx |
| 2017 3.75+AS03<br>(D1-D121) | Pre-Vac 2 (day 121) | х | xx.x | XX.X | xx | xx, xx | XX.X | xx.x | XX | xx, xx |
| (N=X) | Day 8 post Vac 2 | х | xx.x | xx.x | xx | xx, xx | XX.X | XX.X | xx | xx, xx |

| Study Group | Study Day | N* | | Va | lue | | | Change | from Baseli | ne |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Mean | Standard<br>Deviation | Median | Min, Max | Mean | Standard<br>Deviation | Median | Min, Max |
| Group 6: | Baseline | х | XX.X | XX.X | XX | xx, xx | NA | NA | NA | NA |
| 2017 3.75+AS03/<br>2017 15 | Day 8 post Vac 1 | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | xx | xx, xx |
| (D1-D121) | Pre-Vac 2 (Day 121) | х | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | xx | xx, xx |
| (N=X) | Day 8 post Vac 2 | X | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | xx | xx, xx |
| All Subjects | Baseline | х | xx.x | XX.X | XX | xx, xx | NA | NA | NA | NA |
| (N=X) | Pre-Vac 2 | x | xx.x | XX.X | xx | xx, xx | XX.X | XX.X | XX | xx, xx |
| | Day of Vac 2 | x | xx.x | XX.X | XX | xx, xx | xx.x | XX.X | xx | xx, xx |
| | Day 8 post Vac 2 | X | xx.x | XX.X | XX | xx, xx | XX.X | XX.X | XX | xx, xx |

Tables with similar format:

Table 123: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – White Blood Cells

Table 124: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Study Group (Safety Population) – Platelets

### 14.3.4.5 Clinical Laboratory Reference Ranges

(Placeholder for the CSR)

### 14.3.5 Abnormal Laboratory Value Listings (by Subject)

**Table 125:** Listing of Abnormal Laboratory Results - Chemistry

| Subject<br>ID | Study<br>Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Study<br>Vaccination | If Not<br>Related,<br>Alternate<br>Etiology | Action Taken with Study Vaccination | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

**Table 126:** Listing of Abnormal Laboratory Results - Hematology

| Subject<br>ID | Study<br>Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Study<br>Vaccination | If Not<br>Related,<br>Alternate<br>Etiology | Action Taken with Study Vaccination | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

### 14.3.6 Displays of Vital Signs

Table 127: Vital Signs by Assessment, Maximum Severity, Study Day, Study Group (Safety Population) – Any Assessment

| Study Group | Study Day | N* | No | one | M | ild | Mod | erate | Sev | vere | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| Group 1: | Baseline | х | х | xx | х | xx | X | xx | x | xx | х | xx |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 22 post Vac 1 (Vac 2) | х | х | xx | х | xx | X | xx | x | xx | х | xx |
| (D1-D22)<br>(N=X) | Max Severity Post<br>Baseline | Х | х | xx | X | xx | х | XX | Х | xx | х | xx |
| Group 2: | Baseline | х | х | xx | х | xx | X | xx | x | xx | х | xx |
| 2013 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121) | Day 121 post Vac 1 (Vac 2) | Х | х | xx | х | xx | х | xx | Х | xx | х | xx |
| (N=X) | Max Severity Post<br>Baseline | X | х | xx | х | xx | X | XX | Х | xx | х | xx |
| Group 3: | Baseline | X | х | xx | х | xx | X | XX | х | xx | х | XX |
| 2013 3.75+AS03/<br>2017 15<br>(D1-D121) | Day 121 post Vac 1 (Vac 2) | х | х | xx | х | xx | х | XX | Х | xx | х | xx |
| (N=X) | Max Severity Post<br>Baseline | Х | х | xx | х | xx | х | xx | Х | xx | х | xx |
| Group 4: | Baseline | x | х | xx | х | xx | x | xx | x | xx | х | xx |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | Day 22 post Vac 1 (Vac 2) | х | х | xx | х | xx | X | xx | x | xx | х | xx |
| (D1-D22)<br>(N=X) | Max Severity Post<br>Baseline | Х | х | xx | х | xx | х | xx | X | xx | х | xx |
| Group 5 | Baseline | x | х | xx | х | xx | x | xx | x | xx | х | xx |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | Day 121 post Vac 1 (Vac 2) | Х | Х | xx | х | xx | х | XX | х | xx | х | xx |
| (D1-D121)<br>(N=X) | Max Severity Post<br>Baseline | X | Х | XX | х | xx | X | XX | X | xx | Х | xx |

| Study Group | Study Day | N* | No | one | М | ild | Mod | erate | Sev | ere | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| Group 6: | Baseline | X | x | xx | x | xx | X | xx | x | xx | X | xx |
| 2017 3.75+AS03/<br>2017 15<br>(D1-D121) | Day 121 post Vac 1 (Vac 2) | х | х | xx | х | xx | х | xx | х | xx | х | XX |
| (N=X) | Max Severity Post<br>Baseline | Х | х | xx | х | xx | х | xx | х | xx | х | XX |
| All Subjects | Baseline | X | x | xx | x | xx | X | xx | x | xx | X | xx |
| (N=X) | Vac 2 | X | х | xx | х | xx | X | xx | х | xx | x | xx |
| | Max Severity Post<br>Baseline | X | х | xx | X | xx | х | xx | X | xx | х | XX |

The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population; N\*= Number of subjects who completed the indicated visit

Table with similar format:

Table 128: Vital Signs by Assessment, Maximum Severity, Study Day, Study Group (Safety Population) – Oral Temperature

Table 129: Vital Signs by Assessment, Maximum Severity, Study Day, and Study Group (Safety Population) – Systolic Blood Pressure

| <b>Study Group</b> | Study Day | N* | No | one | | M | ild | | | Mod | erate | | | Sev | ere | | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | L | ow | Hi | igh | L | ow | Н | igh | L | ow | Hi | gh | | |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1: | Baseline | X | х | XX | Х | XX | х | XX | х | XX | х | XX | Х | XX | X | XX | Х | XX |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 22 post Vac<br>1 (Vac 2) | X | X | XX | X | XX | Х | XX | X | XX | Х | xx | Х | xx | X | XX | X | XX |
| (D1-D22)<br>(N=X) | Max Severity<br>Post Baseline | X | X | XX | X | XX | Х | XX | X | XX | Х | xx | Х | xx | X | XX | X | XX |
| Group 2: | Baseline | X | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |
| 2013 3.75+AS03/<br>2017 3.75+AS03 | Day 121 post<br>Vac 1 (Vac 2) | X | Х | xx | X | xx | Х | XX | х | XX | Х | XX | X | XX | X | XX | X | XX |
| (D1-D121)<br>(N=X) | Max Severity<br>Post Baseline | X | X | xx | X | xx | Х | XX | х | XX | Х | XX | X | XX | X | XX | X | XX |
| Group 3: | Baseline | х | Х | XX | Х | XX | Х | XX | х | XX | х | XX | х | XX | х | XX | X | xx |
| 2013 3.75+AS03/<br>2017 15 | Day 121 post<br>Vac 1 (Vac 2) | X | X | xx | X | xx | X | XX | х | XX | Х | xx | X | XX | X | XX | X | XX |
| (D1-D121)<br>(N=X) | Max Severity<br>Post Baseline | X | X | XX | X | xx | X | XX | Х | XX | X | xx | Х | XX | X | XX | X | XX |
| Group 4: | Baseline | X | Х | XX | Х | XX | Х | XX | Х | XX | Х | XX | X | XX | X | XX | X | xx |
| 2017 3.75+AS03/<br>2017 3.75+AS03 | Day 22 post Vac<br>1 (Vac 2) | X | X | XX | X | xx | Х | XX | Х | XX | X | xx | Х | XX | X | XX | X | XX |
| (D1-D22)<br>(N=X) | Max Severity<br>Post Baseline | X | X | XX | X | XX | X | XX | X | xx | X | xx | X | XX | X | XX | X | XX |
| | Baseline | X | х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | X | XX | X | xx |
| | Day 121 post<br>Vac 1 (Vac 2) | Х | X | xx | X | xx | х | xx | х | xx | х | xx | X | xx | х | xx | X | XX |

| Study Group | Study Day N* | | N* None | | Mild | | | Moderate | | | Severe | | | | Mis | sing | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | L | ow | Hi | gh | L | ow | Н | igh | L | ow | Hi | igh | | |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 5<br>2017 3.75+AS03/<br>2017 3.75+AS03<br>(D1-D121)<br>(N=X) | Max Severity<br>Post Baseline | х | х | xx | х | xx | х | XX | X | xx | х | xx | х | xx | х | xx | х | XX |
| Group 6: | Baseline | X | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| 2017 3.75+AS03/<br>2017 15 | Day 121 post<br>Vac 1 (Vac 2) | Х | X | XX | X | xx | X | XX | X | xx | X | XX | X | xx | X | xx | X | xx |
| (D1-D121)<br>(N=X) | Max Severity<br>Post Baseline | Х | Х | XX | Х | XX | Х | XX | X | xx | Х | XX | Х | xx | Х | XX | Х | xx |
| All Subjects | Baseline | X | х | XX | х | XX | X | XX | X | XX | х | XX | X | XX | х | XX | X | XX |
| (N=X) | Vac 2 | X | х | XX | х | XX | Х | XX | X | XX | х | XX | Х | XX | х | XX | Х | XX |
| | Max Severity<br>Post Baseline | Х | X | XX | X | xx | X | XX | X | xx | X | XX | X | xx | X | xx | X | xx |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population.

### Tables with similar format:

Table 130: Vital Signs by Assessment, Maximum Severity, Study Day, and Study Group (Safety Population) – Diastolic Blood Pressure

Table 131: Vital Signs by Assessment, Maximum Severity, Study Day, and Study Group (Safety Population) – Pulse

### 14.4 Summary of Concomitant Medications

Table 132: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Study Group

| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2, Therapeutic<br>Subgroup | Group 1<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | | Group 2<br>2013<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D121)<br>(N=X) | | Group 3 2013 3.75+AS03/ 2017 15 (D1-D121) (N=X) | | Group 4<br>2017<br>3.75+AS03/<br>2017<br>3.75+AS03<br>(D1-D22)<br>(N=X) | | Group 5 2017 3.75+AS03/ 2017 3.75+AS03 (D1-D121) (N=X) | | Group 6<br>2017<br>3.75+AS03/<br>2017 15<br>(D1-D121)<br>(N=X) | | All<br>Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |
| [ATC Level 1 – 1] | Any [ATC 1 – 1] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | [ATC 2 - 1] | Х | XX | X | XX | Х | XX | Х | XX | X | XX | х | XX | х | xx |
| | [ATC 2 - 2] | Х | xx | X | XX | Х | XX | Х | XX | X | XX | х | XX | X | XX |
| | [ATC 2 - 3] | Х | xx | X | XX | Х | XX | Х | XX | X | XX | х | XX | X | XX |
| [ATC Level 1 – 2] | [ATC 2 - 1] | Х | xx | X | XX | Х | XX | Х | XX | X | XX | х | XX | X | XX |
| | [ATC 2 - 2] | Х | xx | X | XX | х | XX | х | XX | X | XX | х | XX | X | xx |
| | [ATC 2 - 3] | X | XX | X | xx | X | xx | х | XX | X | xx | х | XX | X | XX |

N= Number of subjects in the Safety Population. n = Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

## APPENDIX 2. FIGURE MOCK-UPS

### LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram |
|---|---|
| Figure 2: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody by Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 3: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody by Study Day and Study Group, Per Protocol Population |
| Figure 4: | Reverse Cumulative Distribution of Neutralizing Antibody by Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 5: | Reverse Cumulative Distribution of Neutralizing Antibody by Study Day and Study Group, Per Protocol Population |
| Figure 6: | Geometric Mean Titers of Hemagglutination Inhibition Antibody by Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 7: | Geometric Mean Titers of Hemagglutination Inhibition Antibody by Study Day and Study Group, Per Protocol Population |
| Figure 8: | Geometric Mean Titers of Neutralizing Antibody by Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 9: | Geometric Mean Titers of Neutralizing Antibody by Study Day and Study Group, Per Protocol Population |
| Figure 10: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody by Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 11: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody by Study Day and Study Group, Per Protocol Population |
| Figure 12: | Box Plots of IgA Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 13: | Box Plots of IgA Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Per Protocol Population |
| | Box Plots of IgG Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 15: | Box Plots of IgG Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Per Protocol Population |
| Figure 16: | Box Plots of IgM Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Modified Intent-to-Treat Population |
| Figure 17: | Box Plots of IgM Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Per Protocol Population |
| Figure 18: | Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 1, Per Protocol Population170 |
| Figure 19: | Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 2, Per Protocol Population171 |

8

8

| Figure 20: | Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 1, Per Protocol Population171 |
|---|---|
| Figure 21: | Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 2, Per Protocol Population171 |
| Figure 22: | Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells at Day 8 Post Vaccination 1 with Antibody Response at Day 21 Post Vaccination 1, Per Protocol Population |
| Figure 23: | Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells at Day 8 Post Vaccination 2 with Antibody Response at Day 21 Post Vaccination 2, Per Protocol Population |
| Figure 24: | Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells at Day 8 Post Vaccination 1 with Antibody Response at Day 21 Post Vaccination 1, Per Protocol Population |
| Figure 25: | Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells at Day 8 Post Vaccination 2 with Antibody Response at Day 21 Post Vaccination 2, Per Protocol Population |
| Figure 26: | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Study Vaccination |
| Figure 27: | Maximum Severity of Solicited Local Symptoms per Subject by Day Post Study Vaccination |
| Figure 28: | Frequency of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity |
| Figure 29: | Frequency of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Severity |
| Figure 30: | Incidence of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity |
| Figure 31: | Incidence of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Severity |
| Figure 32: | Frequency of Adverse Events by MedDRA® System Organ Class and Relationship to Study Vaccination |
| Figure 33: | Frequency of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Relationship to Study Vaccination |
| Figure 34: | Incidence of Adverse Events by MedDRA® System Organ Class and Relationship to Study Vaccination |
| Figure 35: | Incidence of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Relationship to Study Vaccination |
| Figure 36: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter and Study Group – White Blood Cells |

| Figure 37: | Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Study Group – Hemoglobin177 |
|---|---|
| Figure 38: | Laboratory Summary Statistics of Change from Baseline Results by Parameter,<br>Maximum Severity, Study Day, and Study Group – Platelets |
| Figure 39: | Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Study Group – Alanine Aminotransferase (ALT)177 |
| Figure 40: | Laboratory Summary Statistics of Change from Baseline Results by Parameter,<br>Maximum Severity, Study Day, and Study Group – Total Bilirubin |
| Figure 41: | Laboratory Summary Statistics of Change from Baseline Results by Parameter,<br>Maximum Severity, Study Day, and Study Group – Creatinine |

#### 10.1 **Disposition of Subjects**

Figure 1: **CONSORT Flow Diagram** 



### 14.2.2 Immunogenicity Figures

### 14.2.2.1 Serum Antibody Figures

# Figure 2: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody by Study Day and Study Group, Modified Intent-to-Treat Population

[Implementation Note: A generic sample figure is shown below. The RCD curves should be presented in a single figure with six separate panels (4 columns for timepoints (Day 1, Day 22 post Vac 1, Day 22 post Vac 2, Day 181 Post Vac 2), and 2 rows for strains (A/Shanghai/2/2013 (A/H7N9), A/Hong Kong/125/2017 (A/H7N9))). Visit labels should be included in the panel headers. Within each panel individual curves should be used for each Study Group (six curves).]



- Figure 3: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody by Study Day and Study Group, Per Protocol Population
- Figure 4: Reverse Cumulative Distribution of Neutralizing Antibody by Study Day and Study Group, Modified Intent-to-Treat Population
- Figure 5: Reverse Cumulative Distribution of Neutralizing Antibody by Study Day and Study Group, Per Protocol Population

Figure 6: Geometric Mean Titers of Hemagglutination Inhibition Antibody by Study Day and Study Group, Modified Intent-to-Treat Population

[Implementation Note: A generic sample figure is shown below. Planned Study Day is plotted along the x-axis, with visit labels as tick labels. This figure will have two panels for the A/Shanghai/2/2013 (A/H7N9) and A/Hong Kong/125/2017 (A/H7N9) strains. Titer is plotted on the y-axis on the log-10 scale. GMT should be plotted at each visit with upper and lower error bars for the 95% CI for each study group with different marker shapes/colors for each study group. Each study group should have a separate color and marker shape]



- Figure 7: Geometric Mean Titers of Hemagglutination Inhibition Antibody by Study Day and Study Group, Per Protocol Population
- Figure 8: Geometric Mean Titers of Neutralizing Antibody by Study Day and Study Group, Modified Intent-to-Treat Population
- Figure 9: Geometric Mean Titers of Neutralizing Antibody by Study Day and Study Group, Per Protocol Population

Figure 10: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody by Study Day and Study Group, Modified Intent-to-Treat Population

[Implementation Note: A generic sample figure is shown below. The scatter plots should be presented in a seven figure files (one for each study group, and one for overall) each with 8 separate panels (4 columns for each visit (Baseline, Day 22 post vaccination 1, Day 22 post vaccination 2, and Day 181 post vaccination 2) and 2 rows for the strains (A/Shanghai/2/2013 (A/H7N9), A/Hong Kong/125/2017 (A/H7N9))). Visit labels should be included in the panel header. Within each panel distinct marker types and colors should be used to indicate the study groups, with study group labels included in a legend. Each study group should have a unique color and marker shape used within its individual figure file. The spearman correlation should be calculated over all subjects and annotated within each panel as "Spearman Correlation (r=0.xx, p=0.xx)"]



Figure 11: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody by Study Day and Study Group, Per Protocol Population

### 14.2.2.2 Antibody Secreting Cell Figures

# Figure 12: Box Plots of IgA Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Modified Intent-to-Treat Population

[Implementation Note: A generic sample figure is shown below. The box plots should be presented in a single figure with 4 separate panels (2 columns for each visit (Day 8 post vaccination 1 and Day 8 post vaccination 2) and 2 rows for the strains (A/Shanghai/2/2013 (A/H7N9), A/Hong Kong/125/2017 (A/H7N9))). Visit labels should be included in the panel header. Within each panel distinct marker types and colors should be used to indicate the study groups, with study group labels included in a legend. Each study group should have a unique color and marker shape.]



Boxes indicate the 25th and 75th percentiles with the center line indicating the median. Whiskers extend to the 2.5th and 97.5th percentiles. To better visualize the results, the y-axis is presented on a log 2 scale and percent responses =0 are replaced with 0.0001.

- Figure 13: Box Plots of IgA Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Per Protocol Population
- Figure 14: Box Plots of IgG Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Modified Intent-to-Treat Population
- Figure 15: Box Plots of IgG Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Per Protocol Population
- Figure 16: Box Plots of IgM Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Modified Intent-to-Treat Population
- Figure 17: Box Plots of IgM Antibody Secreting Cells by A/H7N9 Strain, Study Day and Study Group, Per Protocol Population

Figure 18: Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 1, Per Protocol Population

[Implementation Note: A generic sample figure is shown below. The scatter matrix should be presented in a single figure with as shown below. Within each panel distinct marker types and colors should be used to indicate the study groups, with study group labels included in a legend. Each study group should have a unique color and marker shape. The spearman correlation should be calculated over all subjects an included in the top-right diagonal as "Spearman Correlation (r=0.xx, p=0.xx)" A legend will include the axis units. The Scatterplot matrix will be repeated twice in the same figure file for HA and NA specific ASC expression.]



### Figures with similar format:

- Figure 19: Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 2, Per Protocol Population
- Figure 20: Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 1, Per Protocol Population
- Figure 21: Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells by Immunoglobulin Type at Day 8 Post Vaccination 2, Per Protocol Population
- Figure 22: Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells at Day 8
  Post Vaccination 1 with Antibody Response at Day 21 Post Vaccination 1, Per Protocol
  Population

[Implementation Note Update: The scatter matrix should be presented in a single figure with one column for each Immunoglobulin type (IgM, IgG, IgA) and one row for each antibody titer (HAI, Neut). Within each panel distinct marker types and colors should be used to indicate the study groups, with study group labels included in a legend. Each study group should have a unique color and marker shape. The spearman correlation should be calculated over all subjects an included in the top-right diagonal as "Spearman Correlation (r=0.xx, p=0.xx)" A legend will include the axis units. The Scatterplot matrix will be repeated twice in the same figure file for HA and NA specific ASC expression.]

- Figure 23: Correlation of A/Shanghai/2/2013 (A/H7N9)-Specific Antibody Secreting Cells at Day 8
  Post Vaccination 2 with Antibody Response at Day 21 Post Vaccination 2, Per Protocol
  Population
- Figure 24: Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells at Day 8 Post Vaccination 1 with Antibody Response at Day 21 Post Vaccination 1, Per Protocol Population
- Figure 25: Correlation of A/Hong Kong/125/2017 (A/H7N9)-Specific Antibody Secreting Cells at Day 8 Post Vaccination 2 with Antibody Response at Day 21 Post Vaccination 2, Per Protocol Population

#### 14.3.1.1 Solicited Adverse Events

# Figure 26: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Study Vaccination

[Implementation Note: A Generic figure is shown below. A *horizontal* bar chart should be presented in 6 image files (one per study group) with separate panels for each study vaccination (2 columns for vaccination #). Axes should be labeled as follows: x-axis label: Study Day, y-axis label: Percentage of Subjects (%). Study vaccination should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the Safety Population who received the relevant study vaccination. Subjects are counted at most once at the maximum severity across all systemic events reported for the specified time point]



Figure 27: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Study Vaccination

#### 14.3.1.2 Unsolicited Adverse Events

# Figure 28: Frequency of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in 3 image files (one per vaccination, and one for all vaccinations) with separate panels for each study groups (6 columns (study groups)). Axes should be labeled as follows: y-axis label: System Organ Class, y-axis label: Number of Events. The study groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the Safety Population. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events" first, then in decreasing order of total incidence]



Figure 29: Frequency of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Severity

### Figure 30: Incidence of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in 3 image files (one per vaccination, and one for all vaccinations) with separate panels for each study group (6 columns). Axes should be labeled as follows: y-axis label: System Organ Class, x-axis label: Percentage of Subjects (%). The study groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. Subjects are counted at most once at the maximum severity across for any events in the applicable SOC. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events" first then in decreasing order of total incidence]



Figure 31: Incidence of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Severity

Figure 32: Frequency of Adverse Events by MedDRA® System Organ Class and Relationship to Study Vaccination

[Implementation Note: A generic sample figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in 1 image file with separate panels for each study group and study dose (6 columns (study groups). Axes should be labeled as follows: y-axis label: System Organ Class, y-axis label: Number of Events. The study groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first then in decreasing order of total frequency]



Figure 33: Frequency of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Relationship to Study Vaccination

Figure 34: Incidence of Adverse Events by MedDRA® System Organ Class and Relationship to Study Vaccination

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in a 1 image file with separate panels for each study group (6 columns (study groups)). Axes should be labeled as follows: y-axis label: System Organ Class, x-axis label: Percentage of Subjects (%). The study groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. Subjects are counted at most once at the maximum relationship (related >not-related) across for any events in the applicable SOC. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first, then in decreasing order of total incidence across groups]



Figure 35: Incidence of Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Relationship to Study Vaccination

#### 14.3.5 Displays of Laboratory Results

Figure 36: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter and Study Group – White Blood Cells

[Implementation note: A generic figure is shown below. Plot should be generated with all study groups in a single image file with panels for each study group (6 columns (study groups)) with a box plot shown for each post-baseline study day that labs are drawn (Day 8 post first vaccination, Day 121 Post first vaccination (only for study groups 2,3,5, and 6), and Day 22 post first vaccination, Day 8 post second study vaccination). Y-axis should be labeled "[Parameter] Change from baseline ([units]). Repeat for all clinical laboratory parameters: WBC, Hgb, PLT, ALT, T. Bili, Cr]



- Figure 37: Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Study Group Hemoglobin
- Figure 38: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Study Group Platelets
- Figure 39: Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Study Group Alanine Aminotransferase (ALT)
- Figure 40: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Study Group Total Bilirubin
- Figure 41: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Study Group Creatinine

## APPENDIX 3. LISTINGS MOCK-UPS

## **LISTINGS**

| Listing 1: | 16.1.6 - Listing of Subjects Receiving Investigational Product | 180 |
|---|---|---|
| Listing 2: | 16.2.1 - Early Terminations or Discontinued Subjects | 181 |
| Listing 3: | 16.2.2.1 - Subject-Specific Protocol Deviations | 182 |
| Listing 4: | 16.2.2.2 - Non-Subject-Specific Protocol Deviations | 183 |
| Listing 5: | 16.2.3: Subjects Excluded from Analysis Populations | 184 |
| Listing 6: | 16.2.4.1 - Demographics Data | 185 |
| Listing 7: | 16.2.4.2 – Pre-Existing and Concurrent Medical Conditions | 186 |
| Listing 8: | 16.2.4.3 – Influenza Vaccination History | 187 |
| Listing 9: | 16.2.6.1 - Individual Immunogenicity Response Data (HAI and Neut) | 189 |
| Listing 10: | 16.2.6.2 - Individual Immunogenicity Response Data (Antibody Secreting Cells). | 189 |
| Listing 11: | 16.2.7.1 - Solicited Events – Systemic Symptoms | 190 |
| Listing 12: | 16.2.7.2 - Solicited Events – Local Symptoms | 191 |
| Listing 13: | 16.2.7.3 - Unsolicited Adverse Events | 192 |
| Listing 14: | 16.2.8.1 - Clinical Laboratory Results – Chemistry | 193 |
| Listing 15: | 16.2.8.2 - Clinical Laboratory Results – Hematology | 194 |
| Listing 16: | 16.2.9.1 - Vital Signs | 195 |
| Listing 17: | 16.2.9.2 - Physical Exam Findings | 196 |
| Listing 18: | 16.2.10 - Concomitant Medications. | 197 |
| Listing 19: | 16.2.11.1 - Pregnancy Reports – Maternal Information | 198 |
| Listing 20: | 16.2.11.2 - Pregnancy Reports – Gravida and Para | 198 |
| Listing 21: | 16.2.11.3 - Pregnancy Reports – Live Birth Outcomes | 199 |
| Listing 22: | 16.2.11.4 - Pregnancy Reports – Still Birth Outcomes | 199 |
| Listing 23: | 16.2.11.5 - Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 199 |

### 16.1.6 Listing of Subjects Receiving Investigational Product

Listing 1: 16.1.6 - Listing of Subjects Receiving Investigational Product

| Subject ID | Randomized<br>Study Group | Product Received Study<br>Vaccination 1 | Product Received Study<br>Vaccination 2 |
|---|---|---|---|
| XXXXXXXXX | Group 1 | 2013 A/H7N9 IIV + AS03 | 2017 A/H7N9 IIV + AS03 |
| XXXXXXXXX | Group 2 | 2013 A/H7N9 IIV + AS03 | 2017 A/H7N9 IIV + AS03 |
| XXXXXXXXX | Group 3 | 2013 A/H7N9 IIV + AS03 | 2017 A/H7N9 IIV |
| XXXXXXXXX | Group 4 | 2017 A/H7N9 IIV + AS03 | 2017 A/H7N9 IIV + AS03 |
| XXXXXXXXX | Group 5 | 2017 A/H7N9 IIV + AS03 | 2017 A/H7N9 IIV + AS03 |
| XXXXXXXXX | Group 6 | 2017 A/H7N9 IIV + AS03 | 2017 A/H7N9 IIV |
### 16.2 Database Listings by Subject

### 16.2.1 Discontinued Subjects

### Listing 2: 16.2.1 - Early Terminations or Discontinued Subjects

[Implementation Note: Category will be either "Early Termination" or "Treatment Discontinuation." In the "Reason" column, concatenate any "specify" fields, including AE number and DV number.]

| Subject ID | Study Group | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

### 16.2.2 Protocol Deviations

### **Listing 3:** 16.2.2.1 - Subject-Specific Protocol Deviations

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal."]

| | Subject<br>ID | Study<br>Group | DV<br>Number | Deviation | Deviation<br>Category | Study<br>Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Ī | | | | | | | | | | | | |
| Ī | | | | | | | | | | | | |

# **Listing 4:** 16.2.2.2 - Non-Subject-Specific Protocol Deviations

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal."]

| Site | Deviation | Start<br>Date | End<br>Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

### 16.2.3 Subjects Excluded from the Analysis

### Listing 5: 16.2.3: Subjects Excluded from Analysis Populations

[Implementation Note: This data in this listing should be congruent with the "Analysis Populations by Study Group" table. The reasons included here should match the SAP text that describes who will be excluded from analyses.]

| Study Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

# 16.2.4 Demographic Data

# **Listing 6:** 16.2.4.1 - Demographics Data

[Implementation Note: If a subject is multi-racial, in "Race" column, note "Multiple: (list races, separated by a comma)."]

| Subject ID | Study Group | Sex | Age at Enrollment (years) | Ethnicity | Race | BMI |
|---|---|---|---|---|---|---|

# Listing 7: 16.2.4.2 – Pre-Existing and Concurrent Medical Conditions

[Implementation Note: "Condition Start Day" and "Condition End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). If ongoing, display "Ongoing" in the "Condition End Day" column]

| Subject ID | Study<br>Group | MH<br>Number | Medical History<br>Term | Condition Start<br>Day | Condition End<br>Day | MedDRA® System Organ<br>Class | MedDRA® Preferred Term |
|---|---|---|---|---|---|---|---|

**Listing 8:** 16.2.4.3 – Influenza Vaccination History

| Subject ID | Study group | Vaccine Type | Month/Year Received | Vaccination Type / Subtype |
|---|---|---|---|---|
| | | [Inactivated/ LAIV/ Unknown] | September 2018 | Seasonal Influenza Vaccination (2017-2018) |
| | | [Inactivated/ LAIV/ Unknown] | June 2017 | Non-Seasonal Influenza A Vaccine Subtype H5N8 |
| | | [Inactivated/ LAIV/ Unknown] | June 2017 | Non-Seasonal Influenza Vaccinae Subtype M-001 |

# 16.2.5 Compliance and/or Drug Concentration Data (if available)

Not applicable for this study.

### 16.2.6 Individual Immunogenicity Response Data

Listing 9: 16.2.6.1 - Individual Immunogenicity Response Data (HAI and Neut)

| Subject ID | Study Group | Planned Time Point | Actual Study<br>Day | Assay | Strain | Titer Replicate 1 | Titer Replicate 2 |
|---|---|---|---|---|---|---|---|
| | | | | | | | · |

# Listing 10: 16.2.6.2 - Individual Immunogenicity Response Data (Antibody Secreting Cells)

| Subject ID | Study Group | Planned Time Point | Actual Study<br>Day | Strain | IgA<br>Frequency | IgG<br>Frequency | IgM<br>Frequency |
|---|---|---|---|---|---|---|---|

#### 16.2.7 Adverse Events

**Listing 11:** 16.2.7.1 - Solicited Events – Systemic Symptoms

| Subject ID | Study Group | Vaccination<br>Number | Post Dose Day | Assessment <sup>1</sup> | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>2</sup> | Alternate<br>Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

<sup>&</sup>lt;sup>1</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.).

<sup>&</sup>lt;sup>2</sup> Grade 3 events only.

**Listing 12:** 16.2.7.2 - Solicited Events – Local Symptoms

| Subject ID | Study Group | Vaccination<br>Number | Product<br>Received <sup>1</sup> | Post Vaccination<br>Day | Assessment <sup>1</sup> | Symptom | Severity |
|---|---|---|---|---|---|---|---|
| | | | | | MA | | |
| | | | | | Clinic | | |

<sup>&</sup>lt;sup>1</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.).

**Listing 13:** 16.2.7.3 - Unsolicited Adverse Events

| Adverse<br>Event | Associated with Vac # | # of Days Post Associated Vac (Duration) | Severity | SAE?<br>MAAE?<br>PIMMC? | Relationship<br>to Study<br>Vaccination | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Vaccination | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA <sup>®</sup><br>System<br>Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | :, Study Gro | up: , AE Num | ber: | | | | | | | | |
| | | | | SAE: No<br>MAAE: Yes<br>PIMMC: No | | | | | | | |
| Comments | <b>S:</b> | | | | | | | | | | |
| Subject ID | :, Study Gro | up: , AE Num | ber: | | | | | | | | |
| Comments | ) <b>:</b> | | | | | | | • | | | |
| Note: For a | dditional detai | ls about SAEs | , see Section | 14.3.3 . | | | | | | | |

### 16.2.8 Individual Laboratory Measurements

### **Listing 14:** 16.2.8.1 - Clinical Laboratory Results – Chemistry

[Implementation Note: These listings (for hematology and chemistry) include all laboratory results, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal results, e.g., 16.2 (Mild). The "extra" fields that are completed for abnormal results are not included in this listing; they are included in the listing of abnormal laboratory results that is included in the table shells.]

| Subject ID | Study Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Alanine aminotransferase (IU/L) | Total Bilirubin<br>(mg/dL) | Creatinine<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|

**Listing 15:** 16.2.8.2 - Clinical Laboratory Results – Hematology

| Subject ID | Study Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | White Blood Cell (10³/μL) | Hemoglobin<br>(g/dL) | Platelets<br>(10³/μL) |
|---|---|---|---|---|---|---|---|---|

### 16.2.9 Vital Signs and Physical Exam Findings

# **Listing 16:** 16.2.9.1 - Vital Signs

[Implementation Note: This listing includes all vital sign assessments, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal assessments, e.g., 100.7 (Mild).]

| Subject ID | Study Group | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Pulse<br>(beats/min) |
|---|---|---|---|---|---|---|---|

### Listing 17: 16.2.9.2 - Physical Exam Findings

[Implementation Note: This listing includes all physical exam findings, scheduled and unscheduled. If a subject does not have any findings upon examination, they will not be included in this listing. If reported as an AE, display "Yes" with the AE Number in parentheses, e.g., "Yes (7)".]

| Subject ID | Study Group | Planned<br>Time Point | Actual<br>Study Day | <b>Body System</b> | Abnormal Finding | Reported as an AE?<br>(AE Number) |
|---|---|---|---|---|---|---|

#### 16.2.10 Concomitant Medications

### **Listing 18:** 16.2.10 - Concomitant Medications

[Implementation Note: "Medication Start Day" and "Medication End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). For medication start dates that are > 30 days prior to enrollment, rather than use exact study days, categorize as follows:

- > 5 years prior to enrollment
- 1-5 years prior to enrollment
- 1-12 months prior to enrollment

If ongoing, display "Ongoing" in the "Medication End Day" column. If taken for an AE or MH, display "Yes" with the AE or MH Number in parentheses, e.g., "Yes (7)".]

| Subject<br>ID | Study<br>Group | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an<br>AE?<br>(AE Number) | Taken for a condition<br>on Medical History?<br>(MH Number) |
|---|---|---|---|---|---|---|---|---|

#### 16.2.11 Pregnancy Reports

[Implementation Note: Only include the "Pregnancy Number" column if a subject has more than 1 pregnancy. Date of Conception will be calculated based on estimated delivery date. BMI will be calculated based on pre-pregnancy height and weight. Mother's weight gain will be calculated based on pre-pregnancy weight and end of pregnancy weight. If a major congenital anomaly with previous pregnancy, display "Yes" and the text from the "specify" field, separated by a colon. If any substance use is reported, include a listing of substance use. If autopsy revealed an alternate etiology, display "Yes" and the text from the "specify" field, separated by a colon. If abnormality in product of conception, display "Yes" and the text from the "specify" field, separated by a colon.]

**Listing 19:** 16.2.11.1 - Pregnancy Reports – Maternal Information

| Subject<br>ID | Study<br>Group | Pregnancy<br>Number | Study Day Corresponding to Estimated Date of Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal Complications During Labor, Delivery, or Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 20: 16.2.11.2 - Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| bject<br>ID | Pregnancy<br>Number | Gravida | Extremely PB <sup>1</sup> | Very<br>Early<br>PB <sup>1</sup> | Early<br>PB <sup>1</sup> | Late<br>PB <sup>1</sup> | Early<br>TB <sup>2</sup> | Full<br>TB <sup>2</sup> | Late<br>TB <sup>2</sup> | Post<br>TB <sup>2</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly with<br>Previous<br>Pregnancy? |

<sup>&</sup>lt;sup>1</sup> Preterm Birth.

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>2</sup> Term Birth.

### **Listing 21:** 16.2.11.3 - Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score,<br>1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month<br>of Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

# **Listing 22:** 16.2.11.4 - Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for Still<br>Birth Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

# **Listing 23:** 16.2.11.5 - Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy<br>Outcome (for this<br>Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|